| This supplement contains the following items for: Douglas PS, Nanna MG, Kelsey MD, et al. |
|---|
| Comparison of an Initial Risk-Based Testing Strategy vs Usual Testing in Stable Symptomatic |
| Patients With Suspected Coronary Artery Disease: The PRECISE Randomized Trial: |

Original protocol, final protocol, and summary of amendments

### **Table of Contents**

| Original Protocol | Page 3 |
|--------------------------------|----------|
| Final Protocol | Page 53 |
| Summary of Protocol Amendments | Page 108 |

CP-907-001-A Jun-29, 2018

#### The **PRECISE** Protocol

# <u>Prospective Randomized Trial of the Optimal Evaluation of Cardiac Symptoms and Revascularization</u>

#### **Study Objective**

The primary objective of the PRECISE trial is to assess clinical outcomes, decision making regarding noninvasive testing and invasive angiography, and costs using a precision evaluation strategy as compared to a usual care strategy in participants with stable symptoms suggestive of coronary artery disease. The precision evaluation strategy will be based on a pre-test risk assessment and will incorporate cCTA with selective FFR<sub>CT</sub> and guideline-recommended care with symptom and risk factor management and no immediately planned testing.

#### **Study Design**

The study will be a prospective, pragmatic, randomized clinical trial of the comparative effectiveness of diagnostic evaluation strategies for stable CAD, to be performed in outpatient settings, including primary care and cardiology practices. Qualifying patients presenting with new symptoms suspicious for clinically significant CAD (and without known CAD), who are recommended for diagnostic testing and did not receive any cardiovascular testing within the past 12 months, will be randomized to an initial strategy of either precision care or usual care. All subsequent decisions in the usual care arm regarding additional testing, medications, and/or procedures will be at the discretion of the responsible clinical care team.

## Study Principal Investigator

Pamela S. Douglas, MD Duke University Durham, NC 27701 USA

#### **Sponsor**

HeartFlow, Inc. 1400 Seaport Blvd., Building B Redwood City, CA 94063 Campbell Rogers, MD Chief Medical Officer


Version Date: Jun 29, 2018

CP-907-001-A Jun-29, 2018

#### **Investigator Protocol Signature Page**

I have read and understand the protocol and agree that it contains all the ethical, legal, and scientific information necessary to conduct this study. I will personally conduct the study as described. I will provide copies of the protocol to all assigned physicians, nurses, and other professional personnel who will participate in the study and will be responsible for their compliance and adherence to the study protocol. I am aware that this protocol must be approved by the Institutional Review Board or Ethics Committee. I agree to adhere strictly to the attached protocol. I agree that clinical data entered on case report forms by me and my staff will be supplied to HeartFlow and may be utilized by HeartFlow in various ways, such as for submission to governmental regulatory authorities and/or in combination with clinical data gathered from other research sites, whenever applicable. I agree to allow HeartFlow monitors and auditors and their designees full access to all medical records at the research facility for participants screened or randomized in the study. I agree to provide all participants with informed consent forms and will ensure adequate informed consent is obtained, as required by government regulations and International Conference on Harmonization guidelines.

| Site Name | Site Number |
|---------------------------------------|-------------|
| Principal Investigator (print name) | Date |
| Pamela S. Douglas, MD CESFFC194FCE4S9 | 6/30/2018 |
| Pamela Douglas, MD, Trial PI | Date |
| DocuSigned by: | 7/2/2018 |
| Campbell Rogers MD HeartFlow CMO | Date |


CP-907-001-A Jun-29, 2018

## **Protocol Version and Amendment Tracking**

| Version Number/Amendment | Approval Date |
|--------------------------|---------------|
| 1.0 | Jun-29, 2018 |


**TABLE OF CONTENTS** 

| I. STUDY SYNOPSIS |
|---|
| II. INTRODUCTION |
| II.A. Primary Hypothesis |
| II.B. Signifance of the Study |
| III. BACKGROUND AND STUDY RATIONALE |
| III.A. Prior Literature and Studies |
| III.B. Rationale for the Current Study: A Precision Approach to Chest Pain Evaluation |
| IV. STUDY OVERVIEW AND OBJECTIVES |
| IV.A. Overview of PRECISE |
| IV.B. Primary Objective and Endpoints |
| IV.C. Secondary Endpoints |
| IV.D. Rationale for the Selection of Outcome Measures |
| IV.E. Rationale for the Selection of Testing in Each Arm |
| IV.F. Participant Randomization |
| IV.G. Diagnostic Evaluations and Subsequent Care |
| V. STUDY PROCEDURES |
| V.A. Participant Screening For Eligibility |
| V.B. Participant Randomization and Enrollment |
| V.C. Participant Cohort Assignment |
| V.D. Participant Follow-Up |
| V.E. Cross Over Participants |
| V.F. Participant Withdrawal |
| V.G. Schedule of Assesments |
| VI. ADDITIONAL ASSESMENTS AND SUBSTUDIES |
| VI.A. Quality of Life Assesments |
| VI.B. Economic and Resource Utilization Assesments |
| VI.C. Imaging and other Cardiac Assessments |
| VII. ENDPOINT DETERMINATION, SAFETY AND MONITORING |
| VII.A. Primary Endpoint Definitions |
| VII.B. Secondary Endpoint Definitions |
| VII.C. Testing Complications and Reporting |
| VII.D. Independent Clinical Event Adjudication Committee |
| VII.E. Data and Safety Monitoring Board |
| Design A of FC |


| VIII. STATISTICAL PLAN |
|---------------------------------------------------------|
| VIII.A. Sample Size Determination and Statistical Power |
| VIII.B. Statistical Analysis Plan |
| IX. ETHICAL CONSIDERATIONS AND RISK ANALYSIS |
| IX.A. Ethical Considerations |
| IX.B. Study Risks and Benefits |
| X. DATA HANDLING AND QUALITY ASSURANCE |
| X.A. Completing and Signing Case Report Forms |
| X.B. Clinical Data Management |
| X.C. Archiving of Data |
| XI. STUDY MONITORING, AUDITING, AND INSPECTING |
| XI.A. Study Monitoring |
| XI.B. Auditing and Inspecting |
| XII. REFERENCES |


### **TABLE OF ABBREVIATIONS**

| ACC | American College of Cardiology |
|---|---|
| AHA | American Heart Association |
| BMI | body mass index |
| BP | blood pressure |
| CAD | coronary artery disease |
| CV | cardiovascular |
| CCC | Clinical Coordinating Center |
| CI | confidence interval |
| CK-MB | creatinine kinase-myocardial band |
| CMS | Centers for Medicare & Medicaid Services |
| COCATS | Core Cardiology Training Symposium |
| cCTA | coronary computed tomographic angiography |
| DCRI | <u>Duke Clinical Research Institute</u> |
| DECISION | <u>D</u> ecisive <u>E</u> valuation of <u>C</u> ardiac <u>I</u> schemia, <u>S</u> ymptoms and Revascularizat <u>ion</u> |
| DSMB | Data and Safety Monitoring Board |
| ECG | electrocardiogram |
| Echo | echocardiogram |
| EDC | electronic data capture |
| EQ-5D-5L | A standardized instrument developed by the <i>EuroQol</i> Group as a measure of health-related quality of life. |
| eCRF | electronic case report form |
| FFR | fractional flow reserve |
| FS | Finkelstein and Schoenfeld statistical method |
| FFR <sub>CT</sub> | non-invasive technique using cCTA to determine FFR |
| g/L | grams per liter |
| HDL | high-density lipoprotein |


| ICA | invasive coronary angiography |
|---|---|
| IRB | institutional review board |
| IVUS | intravascular ultrasound |
| IXRS | interactive voice/web response system |
| LDL | low-density lipoprotein |
| LV | left ventricular |
| MACE | major adverse cardiovascular event |
| MAR | missing at random |
| MDCT | multidetector computed tomography |
| MI | myocardial infarction |
| MOP | manual of procedures |
| mSv | milliSievert |
| NICE | National Institute for Health and Care Excellence (In the United Kingdom's National Health Service) |
| NHPR | non hyperemic pressure ratio |
| PAD | peripheral arterial disease |
| PCI | percutaneous coronary intervention |
| PI | principal investigator |
| PLATFORM | Prospective LongitudinAl Trial of FFR <sub>CT</sub> : Outcome and Resource Impacts study |
| PRECISE | Prospective Randomized Trial of the Optimal Evaluation of Cardiac Symptoms and Revascularization |
| PROMISE | PROspective Multicenter Imaging Study for Evaluation of Chest Pain randomized clinical trial |
| QoL | quality of life |
| ROC | receiver operating characteristic |
| SAQ | Seattle Angina Questionnaire |
| SCOT-<br>HEART | Scottish Computed Tomography of the HEART randomized clinical trial |
| ULN | upper limit of normal |


CP-907-001-A Jun-29, 2018

### I. STUDY SYNOPSIS

| Protocol Title | PRECISE: Prospective Randomized Trial of the Optimal Evaluation of |
|---|---|
| In continuation of Otmoto and | Cardiac Symptoms and Revascularization |
| Investigational Strategy | Precision diagnostic evaluation as the initial strategy for suspected CAD in patients with stable symptoms |
| Study Principal | Pamela S Douglas, MD |
| Investigator | Duke Clinical Research Institute, Duke University, Durham NC |
| Academic Research | Duke Clinical Research Institute (DCRI), Durham, NC, USA |
| Organizations | Cardiovascular Research Foundation (CRF), New York, NY, USA |
| Clinical Research<br>Organization | Medpace Research, Inc. |
| Sponsor | HeartFlow Inc. |
| | 1400 Seaport Blvd |
| | Redwood City, CA 94063 |
| Participants and Study<br>Centers | Approximately 2100 participants randomized at approximately 100 outpatient sites in the US and outside of the US |
| Planned Study Duration | Approximately 48 months |
| Primary Study Objective | To assess clinical outcomes, decision making regarding noninvasive testing and invasive angiography, and costs using a precision evaluation strategy as compared to a usual care strategy in participants with stable symptoms suggestive of coronary artery disease. The precision evaluation strategy will be based on a pre-test risk assessment, and will incorporate cCTA with selective FFR <sub>CT</sub> and guideline-recommended care with symptom and risk factor management and no immediately planned testing. |
| Primary Hypotheses | In stable participants with a clinical recommendation for testing to evaluate suspected coronary artery disease (CAD) a precision evaluation strategy, incorporating a risk-based assignment to guideline recommended medical management without planned testing for selected low risk participants and cCTA with selective FFR <sub>CT</sub> in elevated risk participants, will result in improved clinical outcomes of death/MI and a lower rate of catheterization without obstructive CAD as compared to usual care strategy. |
| Population | Stable patients who have a clinical recommendation for testing (noninvasive or invasive) for suspected coronary artery disease |
| Study Design and Methods | Prospective, pragmatic, randomized clinical trial of diagnostic evaluation strategies for stable CAD, to be performed in outpatient settings, including primary care and cardiology practices. Qualifying patients presenting with new symptoms suspicious for clinically significant CAD (and without known CAD), who are recommended for diagnostic testing and did not receive any cardiovascular testing within the past 12 months, will be randomized to an initial strategy of either precision care or usual care of the site's choosing. All subsequent decisions in the usual care arm regarding additional testing, medications, and/or procedures will be at the discretion of the responsible clinical care team; the use of cCTA as the initial diagnostic strategy is not allowed in the usual care arm. |


| | T |
|---|---|
| | Precision evaluation: Participants randomized to a precision strategy will be assigned to either guideline-recommended care without immediately planned testing (low risk) or cCTA with selective FFR <sub>CT</sub> (elevated risk) using a risk tool based on pre-test clinical characteristics derived from the PROMISE trial and validated in SCOT-HEART trial. Participants assigned to guideline-recommended care without planned testing will be treated with preventive and antianginal medical treatment per guideline recommendations and clinical judgment and followed without testing. Participants and their providers will be provided informational resources explaining the safety and rationale of this strategy based on pre-test probabilities and the PROMISE Minimal Risk Score. Participants with documented intractable symptoms despite maximal medical management may undergo cCTA with selective FFR <sub>CT</sub> at the participant's or site clinician's discretion. |
| | <b>Usual Care:</b> For participants randomized to usual care, the participant's care team will select the specific noninvasive stress test (exercise electrocardiogram, stress nuclear imaging [including PET], stress MR, or stress echocardiogram); OR invasive test: (direct to diagnostic catheterization). The use of cCTA as the <u>initial</u> diagnostic strategy is explicitly excluded in this arm. |
| | In both arms, the participant's care team will be provided with physician and patient informational resources summarizing current recommendations for test interpretation and preventive care. Optimal medical management will be recommended but not mandated in either arm. |
| Randomization and Stratification | Participants will be randomized using a 1:1 randomization scheme via an interactive web or voice-based system (IXRS). Randomization will be stratified by intended first test if randomized to usual care, low vs. elevated pre-test risk, and site. |
| | Enrollment in the strata of intended noninvasive test first (vs. intended invasive angiography first) will be capped at 90%. |
| Primary Endpoint | Time to a composite of: MACE (all cause death, non-fatal MI) or invasive cardiac catheterization without obstructive CAD (obstructive CAD defined as diameter stenosis ≥50% according to clinical site interpretation, FFR≤0.80, or NHPR<0.90) at one year (intention to treat) |
| Secondary Effectiveness<br>Endpoints | <ul><li>Endpoints will be assessed at 45 days, 6 months, 1 year, and 2 years.</li><li>Hierarchical analysis (Finkelstein and Schoenfeld (FS) or Pocock's win ratio) of primary endpoint</li></ul> |
| | Resource use patterns (all patients) and medical costs (US patients) to 12 months |
| | 3. QoL: measured by the Seattle Angina Questionnaire (SAQ) to assess angina-specific Quality of Life and the EuroQoL 5D (EQ-5D-5L) survey to assess overall (generic) health status |
| | 4. Death: All-cause, cardiovascular, non-cardiovascular |
| | 5. Myocardial infarction: All, procedural, spontaneous MI |


| | Hospitalizations: All, cardiovascular, non-cardiovascular, and for progressive or unstable angina |
|---|---|
| | 7. Preventive medication use (ASA, statins) in participants with clinical indication for use: eg: hyperlipidemia, diabetes, documented CAD |
| | 8. Cumulative radiation exposure at 1 year |
| | 9. PRECISE primary endpoint at 24 months |
| | 10. MACE, defined as all-cause death myocardial infarction, or ischemia-driven revascularization at 24 months (DECISION co-primary end point) |
| | 11. All-cause death, MI, all follow-up unplanned revascularization procedures, cardiac catheterizations without actionable findings at 24 months (DECISION co-primary end point) |
| | 12. Proportion of invasive cardiac catheterization patients who undergo revascularization (PCI or CABG) within 6 months of enrollment |
| Pre-specified subgroup | Low risk vs. elevated risk by PROMISE score |
| analyses | 2. Intended initial test: functional stress test vs. invasive (direct to cath) |
| | 3. Clinical factors: Sex, age, diabetes |
| | Presentation: Primary symptom (chest pain vs. other), SAQ angina frequency score |
| Inclusion Criteria | Inclusion criteria (all must be present): |
| | 1. Age ≥18 years |
| | 2. Stable typical or atypical symptoms suspicious for coronary artery disease with further non-emergent testing or elective catheterization recommended to evaluate the presence of suspected coronary artery disease |
| | 3. Safe performance of cCTA: |
| | Creatinine clearance ≥45 ml/min |
| | <ul> <li>For a female participant of childbearing potential, a pregnancy test<br/>must be performed with negative results known within 7 days prior to<br/>randomization</li> </ul> |
| | 4. Willingness to comply with all aspects of the protocol, including adherence to the assigned strategy and follow-up visits |
| | 5. Ability to provide written informed consent |
| Exclusion criteria | Exclusion criteria (all must be absent): |
| | Acute chest pain |
| | 2. Unstable clinical status |
| | 3. Noninvasive or invasive CV testing for CAD within 1 year |
| | 4. Lifetime history of any obstructive CAD (no prior CABG or PCI, stenosis ≥50%), or known EF ≤40% or moderate to severe valvular or congenital cardiac disease |
| | <ol> <li>Contraindications to cCTA including but not limited to estimated<br/>creatinine clearance (GFR) &lt;45 ml/min measured within 90 days</li> </ol> |
| | 6. Exceeds local weight or size limit for cCTA or cardiac catheterization |
| | 7. Any condition leading to possible inability to comply with the protocol procedures or follow-up |
| | 8. Any condition that might interfere with the study procedures or follow-up |


CP-907-001-A Jun-29, 2018

| | <ul> <li>9. Enrolled in an investigational trial that involves a non-approved cardiac drug or device which has not reached its primary endpoint</li> <li>10. Life expectancy less than 2 years due to non-cardiovascular comorbidities</li> </ul> |
|---|---|
| Study Follow-up | Participant follow-up will be done at 45 days, 6 months, 1 year, and 2 years. |
| Sample Size<br>Considerations | Primary superiority testing hypothesis of all cause death/MI or invasive cardiac catheterization without obstructive CAD (diameter stenosis ≥50% or FFR≤0.80/ or NHPR<0.90) at one year (intention to treat, time to first event analysis): Assuming an 8% event rate at 1 year in the usual care group and 5% in the precision care group (3% absolute [37.5% relative] effect magnitude). Assumed rates are based on 30% assigned to guideline-recommended care with symptom management and no planned testing (within which 30% will cross over to cCTA with selective FFR <sub>CT</sub> ); and overall 10% will not receive assigned testing; enrolling 1050 participants per group (2100 total participants) would provide at least 90% power to demonstrate superiority accounting for 10% attrition rate. |


CP-907-001-A Jun-29, 2018

#### II. INTRODUCTION

#### **II.A. Primary Hypotheses**

The overarching goal of the Prospective Randomized Trial of the Optimal Evaluation of Cardiac Symptoms and Revascularization (PRECISE) research program is to assess clinical outcomes, decision making regarding noninvasive testing and invasive angiography, and costs using a precision evaluation strategy as compared to a usual care strategy in participants with stable symptoms suggestive of coronary artery disease. The precision evaluation strategy will be based on a pre-test risk assessment, and will incorporate cCTA with selective FFR<sub>CT</sub> and guideline-recommended care with symptom management and no planned testing.

The primary hypothesis of PRECISE is: in stable participants with a clinical recommendation for testing to evaluate suspected coronary artery disease (CAD) a precision evaluation strategy will result in improved clinical outcomes of death/MI and a lower rate of catheterization without obstructive CAD as compared to a usual care strategy.

An important secondary hypothesis is that the precision evaluation strategy will result in improved patient-reported outcomes, reflected in the SAQ angina frequency and quality of life scores. We also expect the precision strategy to result in reduced resource utilization and net cost savings compared to usual care evaluation.

The usual care arm participants will undergo either noninvasive stress testing, with the specific modality at the discretion of the participant's clinician, or invasive cardiac catheterization (ICA) as the initial test.

The precision evaluation arm starts with the use of the PROMISE Risk Tool to categorize patient risk for CAD and events. The PROMISE Risk Tool is a validated risk model that has been shown to accurately identify chest pain patients who are unlikely to benefit from non-invasive testing (i.e. have minimal or no atherosclerosis and likely to have no events within two years). The lowest risk group in the precision arm identified using this model will be assigned to guideline-recommended care focused on symptom and risk factor management without planned cardiac diagnostic testing. The remaining participants, who will be of elevated risk, will be initially evaluated with cCTA with selective  $FFR_{CT}$ .

#### I.B. Significance of the Study

The goal of PRECISE is to define the optimal evaluation and management strategy of stable, symptomatic participants with suspected CAD. If the hypotheses of PRECISE are supported by the results of the trial, PRECISE will form the core of a compelling body of evidence supporting important changes in clinical practice guidelines and clinical care that will both improve outcomes for patients and reduce the use of unnecessary (low yield) testing and associated medical costs. Chest pain is one of the most common symptoms that bring patients into the health care system and one of the most difficult for providers to address confidently. The variability of current practice and the frequent overuse of testing derive from the lack of consensus among experts and among guidelines about how best to achieve a secure diagnosis and appropriate management plan. The results of PRECISE will have major implications for all health systems where stable chest pain is a common reason for subjects to seek care.


CP-907-001-A Jun-29, 2018

#### III. BACKGROUND AND STUDY RATIONALE

#### III.A. Prior Literature and Studies

<u>Unmet need to develop novel approaches for the diagnostic evaluation in stable chest pain</u> patients

Coronary artery disease is an extremely common diagnosis worldwide and results in significant morbidity and mortality<sup>1, 2</sup>. Among the common presentations, stable symptoms of chest pain or exertional dyspnea can be diagnostically puzzling and often require diagnostic testing or angiography to be certain of the diagnosis and treatment. Current US, EU and UK guidelines recommend risk stratification using presentation characteristics and risk factors to determine which patients require noninvasive testing or should be referred directly to invasive catheterization<sup>3</sup>. However, in the current era, the results of using these recommended strategies are unsatisfactory. The population undergoing noninvasive testing has a low rate of obstructive CAD (10-20%) and very low annual event rates (~1-2%/year) <sup>4, 5</sup>, while patients undergoing invasive angiography frequently don't have actionable CAD<sup>6</sup>. These patterns of care have resulted in high costs without accompanying clinical benefit<sup>7</sup>. A new approach to the risk stratification and subsequent diagnostic evaluation and management of patients with stable symptoms suggestive of CAD is urgently needed.

<u>Uncertainty Regarding the Optimal First Test for Detection and Exclusion of Coronary Artery</u> Disease: Evidence For cCTA

While a number of functional and anatomic non-invasive tests are available for the evaluation of stable chest pain patients, the optimal evaluation strategy for patients with stable chest pain is uncertain, and recommendations in current guidelines differ markedly. In a recent attempt to address these issues systematically, two large multicenter, open-label, randomized controlled trials explored the diagnostic evaluation of patients with symptoms that may represent coronary artery disease. The SCOT-HEART (Scottish Computed Tomography of the HEART)<sup>4</sup> and PROMISE (PROspective Multicenter Imaging Study for Evaluation of chest pain)<sup>5</sup> trials sought to address evidence gaps in noninvasive testing in stable chest pain, an area in which few randomized trials had previously been conducted.

Key findings from SCOT-HEART and PROMISE: The overall results and important similarities and differences between the two trials have been recently described<sup>8</sup>. The SCOT-HEART study enrolled 4,146 patients with stable chest pain to cCTA in addition to usual care (which generally included electrocardiogram [ECG] stress testing) or to usual care alone. The trial used an upstream primary endpoint related to diagnostic thinking: managing clinician certainty of the diagnosis of angina secondary to CAD, which showed an increase in the cCTA group (RR: 1.79; 95% confidence interval [CI]: 1.62 to 1.96), as did the secondary endpoint of certainty of diagnosis of CAD (RR: 2.56; 95% CI: 2.33 to 2.79). The clinical outcomes-related secondary endpoint of the rate of cardiovascular death or nonfatal myocardial infarction (MI) appeared to be reduced in the cCTA group at 20 months (RR: 0.62, 95% CI: 0.38 to 1.01; p=0.0527), although the overall event rates were low in both arms, reflecting the inclusion of a large number of patients without


CAD. Of note, a landmark analysis excluding the 7 week delay to receiving a cCTA yielded a hazard ratio of 0.50 for CV death and MI<sup>9</sup>.

The larger PROMISE trial randomly assigned 10,003 symptomatic, stable outpatients requiring evaluation for suspected CAD to either initial cCTA or functional stress testing (exercise treadmill testing [ETT], nuclear stress testing, or stress echocardiography), with a median follow-up of 25 months. The event related composite primary endpoint (death, MI, hospitalization for unstable angina, or major cardiovascular procedural complication) occurred at similar rates in the cCTA and functional testing groups (3.3% and 3.0%), which was lower than previously established historical rates. More patients in the cCTA group underwent cardiac catheterization within 90 days after randomization (12.2% vs. 8.1%), but the secondary endpoint of the frequency of catheterization showing no obstructive CAD was significantly lower in the cCTA group (3.4% vs. 4.3%, p=0.02) as was the rate of death and MI at 12 months (HR 0.66; p=0.049). Furthermore, among patients randomized to an intended nuclear testing strategy, the mean cumulative radiation exposure was lower in the cCTA group compared with the functional testing group (12.0 - 8.4 mSv vs. 14.1 - 7.6 mSv). This encompassed all downstream radiation within 90 days, including that associated with cardiac catheterization, and is particularly intriguing because more cCTA patients received cardiac catheterization.

In addition to improving triage to the cardiac catheterization lab and potentially reducing radiation exposure, mounting evidence has demonstrated that use of cCTA, compared to functional testing, yields improved preventive medical treatment and better prognostic information<sup>4, 5, 10</sup>. Patients in the PROMISE trial who underwent cCTA experienced greater uses of indicated cardio-protective medications such as aspirin and statins<sup>10</sup>. This increase is prognostically important, as data from the CONFIRM registry (Coronary CT Angiography Evaluation for Clinical Outcomes International Multicenter) demonstrated that baseline statin therapy among patients with non-obstructive CAD<sup>11</sup> identified on cCTA was associated with a reduction in mortality compared to non-use<sup>12</sup>, while statin therapy among patients with obstructive CAD identified on cCTA was associated with a reduction in MACE<sup>13</sup>.

The identification of non-obstructive CAD with high risk plaque characteristics can only be accomplished non-invasively by cCTA and is an important prognostic indicator, with even mild abnormalities conferring nearly three times the risk of death, MI and unstable angina compared to patients with a normal study<sup>14, 15</sup>. Furthermore, cCTA leads to higher yield of positive results with actionable or obstructive CAD, among patients undergoing cardiac catheterization<sup>5</sup>. This is in line with data from the CONFIRM registry, where investigators demonstrated that cCTA could be used as an effective gatekeeper prior to invasive coronary angiography<sup>16</sup>.

Most importantly, a recent meta-analysis largely based on PROMISE and SCOT-HEART data showed a clear benefit in 'hard' cardiovascular outcomes to a cCTA first strategy, with a 29% reduction in MI<sup>17</sup>. This was potentially driven by the increase in medication utilization in the cCTA arm of the study as well as more catheterization and revascularization<sup>17</sup>.

To summarize, there are several practical and clinical implications of SCOT-HEART and PROMISE which inform the proposed design of PRECISE:

 Contemporary patients with stable chest pain are at low risk of clinical events. Therefore, a strategy to test only those with an elevated likelihood of having obstructive CAD or risk for events, while instituting optimal medical care including deferring testing in those unlikely to


benefit (i.e. using the PROMISE Risk Score), may be feasible, clinically important and efficient.

- cCTA is a reasonable first test for routine assessment of patients with stable chest pain, and when compared to functional testing, is associated with an increase in preventive medication use and a reduction in myocardial infarction.
- Future trials investigating the optimal evaluation of patients with stable chest pain should include the evaluation of clinical outcomes and other measures of testing efficiency (i.e., cardiac catheterization without obstructive CAD).

#### The Case for the Use of cCTA with selective FFR<sub>CT</sub> as the Optimal First Test

The current noninvasive diagnostic testing strategies using functional testing have relatively poor accuracy given the low disease prevalence in this population, leading to high rates of false-positive results<sup>18</sup>. Specifically, current diagnostic strategies lead to high rates (~50%) of cardiac catheterization without significant obstructive disease or need for revascularization<sup>5, 7</sup>. As described above, incorporating cCTA into testing strategies can reduce the frequency of cardiac catheterization without obstructive disease but tends to increase rates of invasive angiography <sup>4, 5</sup>.

Non-invasive computationally-derived FFR<sub>CT</sub> has been developed using resting coronary CT images without the administration of adenosine or change in underlying cCTA protocols¹8-21. The methodology has been previously described elsewhere. <sup>22</sup> In short, FFR<sub>CT</sub> uses the accurate anatomical model of the coronary arteries and myocardium obtained with conventional cCTA and applies the physical laws that govern flow, microcirculatory resistance, coronary branching, and simulated hyperemia. The Navier-Stokes equations that solve for velocity, resistance and pressure for all Newtonian fluids are applied to provide a 3-dimensional pressure map across the coronary tree. This use of computational fluid dynamics generates FFR values from 0 to 1, with ≤0.80 considered hemodynamically significant. The values are congruent with invasive FFR, as shown in several prospective validation studies¹8-20. Finally, the anatomical modeling has been improved by the use of advanced deep and machine learning techniques applied to the large data sets acquired via central analysis.

The addition of FFR<sub>CT</sub> may reduce a potential limitation of a cCTA-first approach, excess invasive angiography, by providing both functional and anatomic data. Specifically, FFR<sub>CT</sub> markedly reduces in the false positive rate of cCTA alone vs. invasive FFR adjudicated ischemia with 68% of false positive CT interpretations in the NXT Trial reclassified as true negative. A retrospective analysis from the PROMISE trial in 181 patients with cCTA, cardiac catheterization and FFR<sub>CT</sub> revealed that FFR<sub>CT</sub> was a better predictor of revascularization and events than cCTA alone. Modelling of the incorporation of FFR<sub>CT</sub> into catheterization decision making suggested a reduction in catheterization rate with cCTA from 12.2% to 7.8% while reducing the rate of catheterization without obstructive CAD from 27% to 15% and increasing the yield of catheterization leading to revascularization from 49% to 61%<sup>23</sup>. Given that PCI of lesions with negative FFR is associated with worse outcomes<sup>24, 25</sup>, while treatment of FFR positive lesions with PCI vs. optimal medical therapy results in improved clinical outcomes, the potential clinical value of adding FFR<sub>CT</sub> to a cCTA based diagnostic strategy is evident.


CP-907-001-A Jun-29, 2018

The safety and utility of a CT/ FFR<sub>CT</sub> strategy were further tested in the PLATFORM Study (Prospective LongitudinAl Trial of FFR<sub>CT</sub>: Outcome and Resource Impacts) which evaluated rates of invasive catheterization without obstructive CAD in patients undergoing invasive evaluation. Patients in 2 sequential non-overlapping cohorts of patients referred for ICA were assigned to either undergo ICA or cCTA/ FFR<sub>CT</sub> with ICA use based on the results of the cCTA and FFR<sub>CT</sub>. The cCTA/FFR<sub>CT</sub> strategy resulted in a significant reduction in the rate of cath lab finding of no obstructive disease, from 73 to  $12\%^7$ . Furthermore, ICA was deferred in 61% of cCTA/FFR<sub>CT</sub> strategy patients. A follow-up at one year demonstrated that cCTA with selective FFR<sub>CT</sub> strategy yielded similar clinical outcomes and quality of life, at a substantially reduced cost.

While much of the early focus has been on a reduction in referral for ICA in the absence of actionable CAD, more recently there has been growing interest in using FFR<sub>CT</sub> to enhance catheterization lab efficiency by increasing the proportion of catheterizations that include revascularization (ICA/PCI ratio) and providing guidance regarding revascularization strategies before the invasive angiogram. Importantly, in this case FFR<sub>CT</sub> is not being used only in a binary fashion but rather to provide a richer understanding of the pattern and degree of pressure loss across the epicardial coronary system and its connection to the extent of ischemia present. The value of cCTA and FFR<sub>CT</sub> has been recognized by The National Institute for Health and Care Excellence (NICE) in their advisory for stable chest pain (Clinical Guidance 95) and technical evaluation of FFR<sub>CT</sub>, as well as by establishment of reimbursement standards by the Centers for Medicare and Medicaid Services (CMS) <sup>26, 27</sup>. The 2016 NICE guidance recognized the difficulties with risk stratification in an era of reduced obstructive CAD prevalence in the population undergoing evaluation and the importance of anatomical assessment of CAD<sup>26, 27</sup>. In response, it recommends coronary cCTA as the first-line investigation for patients presenting with new-onset chest pain felt to be due to CAD based on its superior clinical diagnostic utility and costeffectiveness<sup>26, 27</sup>. Further, based on the results of the PLATFORM trial, the NHS recommends addition of FFR<sub>CT</sub> to cCTA as a cost savings measure<sup>26</sup>. In the United States, CMS approved a New Technology Ambulatory Payment Classification (APC) for HeartFlow FFR<sub>CT</sub> analysis on January 1, 2018<sup>28</sup>. The acknowledgement of FFR<sub>CT</sub> by CMS is a critical step toward increasing the availability of the technology to patients who may benefit. However, other organizations' standards documents have not yet been revised to incorporate the emerging evidence base supporting CCTA and FFR<sub>CT</sub>, indicating that there is still a need for additional evidence to support the routine use of FFR<sub>CT</sub> in clinical practice.

## Rationale and Evidence for Incorporation of a Strategy of Guideline-recommended Care without Planned Testing in Low Risk patients

Given the low prevalence of obstructive CAD (10-20%) and very low annual event rates (~1-2%/year) among stable chest pain patients undergoing non-invasive testing, combined with the high cost of testing<sup>4, 5</sup>, prospective evaluation of the safety and efficacy of an approach of guideline-recommended care without planned testing has become a necessity. Although there are no data regarding outcomes and costs of a guideline-recommended care without planned testing in symptomatic patients, it is possible to define in principle a cohort in whom deferred testing might be the optimal strategy. The argument for testing this is further strengthened by the equivalence of medical and invasive strategies in preventing cardiovascular events in stable CAD, as several trials have shown no benefit of revascularization over optimal medical treatment <sup>29, 30</sup>. It is reasonable to hypothesize that this may be especially true for those at lowest risk, in whom noninvasive testing is even less likely to lead to outcomes-improving revascularization, thereby removing the need for testing as a gateway to the catheterization laboratory.


CP-907-001-A Jun-29, 2018

The COURAGE trial (Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation) demonstrated no significant difference in a composite of death, myocardial infarction, and stroke between patients with objective evidence of myocardial ischemia and significant CAD on medical therapy vs. those undergoing PCI (19.5% vs. 20.0%, p=0.62)<sup>29</sup>. The more recent ORBITA trial (Percutaneous coronary intervention instable angina) randomized 200 patients with stable angina and a single-vessel stenosis to optimal medical therapy + PCI vs. optimal medical therapy plus a sham procedure, with a primary endpoint of difference in exercise time during a 6-week follow-up period<sup>30</sup>. The authors found no significant difference in improvement in exercise time (+28.4 seconds in PCI group vs. +11.8 seconds in sham group, p=0.2), nor any significant change in the secondary outcome of Seattle Angina Questionnaire (SAQ)-angina frequency from baseline (14.0 in PCI group vs. 9.6 in sham group, p=0.26)<sup>30</sup>. The ongoing improvements in medical management of CAD risk, angina and established coronary artery disease further emphasize the need for diagnostic strategies that minimize unnecessary invasive angiography and revascularization by emphasizing guideline-recommended care in patients at very low risk for obstructive disease.

These studies support the development of a patient-centric strategy to identify those who may derive minimal benefit from testing, a strategy which carries several desirable implications for patients, clinicians, and clinical practice in general. For patients, this process can mean a reduction in use of testing from which they would not benefit, thereby saving time, anxiety, and cost, as well as potential reductions in radiation exposure and false-positive test results that could lead to more invasive, unnecessary procedures. For clinicians, a tool identifying the lowest risk patients has the potential to help optimize office-based decision making. From a practice and societal perspective, in an era in which practitioners are increasingly held accountable for costs and quality, the ability to confidently identify patients highly unlikely to benefit from potentially expensive testing and who may therefore be managed conservatively has many potential economic and process-of-care advantages.

The PROMISE Risk Tool was expressly developed to identify low-risk patients with stable chest pain who are unlikely to benefit from non-invasive testing, and for whom guideline-recommended medical management alone may be safe. Current guidelines recommend using a version of the Diamond and Forrester risk score for pretest likelihood of obstructive CAD, but multiple investigators have found that this tool grossly over estimates actual presence of disease<sup>5, 31, 32</sup>. The consequence is an imprecise evaluation strategy for millions of patients, resulting in unhelpful testing of lower risk individuals. For a significant portion of these, a false positive functional testing leads them to have invasive cardiac catheterizations to rule out the disease they do not have. The Risk Tool developed using the PROMISE cohort employs 10 readily available clinical variables and has been validated in the SCOT-HEART population<sup>33, 34</sup>. This risk tool identifies patients with stable chest pain who have no coronary plaque or calcification by cCTA and no cardiac events over 2 years, and who therefore would be predicted to derive minimal or no value from noninvasive testing<sup>33, 34</sup>. Testing whether this risk tool can be employed prospectively to safely and effectively risk stratify low risk patients into a strategy of guideline-recommended care with symptom and risk factor management and without diagnostic testing is one of the core secondary objectives of the PRECISE research program.

#### III.B. Rationale for the Current Study: A Precision Approach to Chest Pain Evaluation


CP-907-001-A Jun-29, 2018

Despite the high-burden of stable chest pain in the U.S., and the enormous research literature reporting on the comparative effectiveness of different options, no single diagnostic strategy has emerged with a broad consensus of support. Each testing community continues to favor its own technology and the clinicians who must select the testing approach to use for their patients are caught in the middle, unable to resolve the controversies that have characterized this area of cardiovascular medicine for decades. The situation is complicated by the heterogeneity of the current population's burden of disease. More than a quarter (27%) of the PROMISE cohort had no coronary plaque whatsoever, while high-risk CAD, defined as left main stenosis (≥50% stenosis) or either (a) ≥50% stenosis '[50]' or (b) ≥70% stenosis '[70]' of 3 vessels or 2-vessel CAD involving the proximal left anterior descending artery was identified in 6.6% [50] and 2.4% [70] of patients. Thus, the first goal of any optimal management strategy for stable symptoms in patients with suspected CAD is determination of an individual patient's risk. Using the PROMISE Risk Tool to accurately assess patient risk<sup>33, 34</sup>, we will prospectively test the hypothesis that low risk patients can be correctly identified with only baseline clinical data and that emphasizing guideline-recommended care while deferring testing in these patients improves chest pain decision making by reducing unnecessary invasive angiography without leading to an increase in MACE, and by reducing cost.

Among patients in whom contemporary risk evaluation suggests an elevated risk for obstructive CAD, the observational data suggest that cCTA with selective FFR<sub>CT</sub> may improve appropriate triage to invasive angiography<sup>5, 23</sup>, while reducing cost<sup>9</sup>.

Thus, the case for an adequately powered randomized clinical trial with a pragmatic design, comparing clinical outcomes following testing strategies regularly used in current clinical practice to a precision evaluation strategy is compelling. PRECISE is designed to be that trial

If the findings of PRECISE are positive as hypothesized, it is expected that the trial will lead to updates in appropriate use criteria, clinical practice guidelines, and payer policies such that cCTA with selective FFR<sub>CT</sub> receives a class IA recommendation for stable chest pain patients to improve outcomes and reduce costs. PRECISE will identify those chest pain patients for whom non-invasive testing may be safely deferred and simultaneously improve the efficiency of testing for elevated risk patients. The results of this study will shift the paradigm of clinical thinking in this area from the current approach of identifying a single best test for all, to incorporating a patient-centric risk-based evaluation and management strategy for stable chest pain patients.

#### IV. STUDY OVERVIEW AND OBJECTIVES

#### IV.A. Overview of PRECISE

PRECISE is a multicenter, randomized, trial that will enroll approximately 2100 participants in a comparison of a risk-based precision evaluation strategy of guideline-recommended medical management without planned testing (in minimal risk participants) and cCTA with selective FFR<sub>CT</sub> (in elevated risk participants) with usual care in stable symptomatic patients with suspected CAD.

#### Location

Participants will be enrolled at approximately 100 outpatient sites in the US and outside of the US. No center may enroll more than 315 (15%) participants in the trial.


CP-907-001-A Jun-29, 2018

#### Participant Population and Selection

Participants will be symptomatic patients with suspected CAD and a stable clinical course who are recommended by their managing clinician to have a non-invasive diagnostic test or ICA. Subjects will be excluded if they have any history of documented CAD (including revascularization, myocardial infarction or any degree of CAD proven by imaging) or have had diagnostic cardiovascular testing for suspected CAD within the last year. Subjects will also be excluded if their symptoms are not clearly stable or if their managing clinician feels testing is needed on an urgent or emergent basis.

Diagnostic testing for the assessment of CAD symptoms is ordered by physicians and other clinicians from many specialties and is performed in multiple settings, including physician offices, hospital outpatient departments, and diagnostic testing facilities. A trial, such as PRECISE, that seeks to improve the management of non-acute chest pain must incorporate this diversity in order to be broadly relevant to the target population under study. PRECISE site selection will seek to encompass this diversity.

#### Study duration

The anticipated total duration of the PRECISE study will be approximately 48 months for start-up, enrollment, follow up, and close out. Participants will be followed for 24 months after enrollment.

#### Study design

The figure below represents a diagrammatic representation of the trial design.


PRECISE Protocol CP-907-001-A



#### IV.B. Primary Objective and Endpoints

The primary objective of the PRECISE study is to assess clinical outcomes, patient-reported outcomes, decision making regarding noninvasive testing and invasive angiography, and costs using a precision evaluation strategy as compared to a usual care strategy in participants with stable symptoms suggestive of coronary artery disease. The precision evaluation strategy will be based on a pre-test risk assessment and will incorporate cCTA with selective FFR<sub>CT</sub> and guideline-recommended care with symptom and risk factor management and no immediately planned testing. We hypothesize that in stable patients with a clinical recommendation for testing to evaluate suspected CAD the proposed precision evaluation strategy will improve outcomes and reduce costs compared to usual care evaluation.

The primary endpoint is a composite of: MACE (all cause death and non-fatal MI) or invasive cardiac catheterization without CAD (no coronary stenosis ≥50%, or with FFR≤0.80, or non-hyperemic pressure ratio (NHPR) <0.90). The primary study hypothesis will be tested at one year using an intention to treat analysis.


#### IV.C. Secondary Endpoints

Endpoints will be assessed at 45 days, 6 months, 1 year, and 2 years. Secondary endpoints include:

- 1. Hierarchical analysis (Finkelstein and Schoenfeld (FS) or Pocock's win ratio) of primary endpoint (gives priority to clinical importance of the components of the composite outcome rather than time to event)
- 2. Resource use patterns (all participants) and medical costs (US participants): resources to be assessed include index testing, follow up testing, diagnostic and other cardiac procedures and hospitalizations. Primary comparisons will be made at 12 months.
- 3. QoL: the Seattle Angina Questionnaire (SAQ) will be used to assess angina-specific Quality of Life; the EuroQoL 5D (EQ-5D-5L) survey will be used for a brief assessment of overall (generic) health status; patient satisfaction with diagnostic process will be assessed once at 45 days using a 4-item instrument created for this trial.
- 4. Death: All-cause, cardiovascular, non-cardiovascular
- 5. Myocardial infarction: All, procedural, spontaneous MI
- 6. Hospitalizations: All, cardiovascular, non-cardiovascular, and for progressive or unstable angina
- 7. Rates of preventive medication use (ASA, statins) in participants with clinical indication for use: hyperlipidemia, diabetes, documented CAD
- 8. Cumulative radiation exposure at 1 year
- 9. PRECISE primary endpoint at 24 months
- 10. MACE, defined as all-cause death myocardial infarction, or ischemia-driven revascularization at 24 months (DECISION co-primary end point)
- 11. All-cause death, MI, all follow-up unplanned revascularization procedures, cardiac catheterizations without actionable findings at 24 months (DECISION co-primary end point)
- 12. Proportion of invasive cardiac catheterization patients who undergo revascularization (PCI or CABG) within 6 months of enrollment (catheterization efficiency)

#### IV.D. Rationale for the Selection of Outcome Measures

#### Rationale for Clinical Assessments

Major adverse cardiovascular events (MACE) are a primary concern for clinicians and patients presenting with stable chest pain. The primary composite endpoint of MACE at 12 months (all cause death, non-fatal MI), invasive cardiac catheterization without obstructive CAD (diameter stenosis ≥50%, FFR≤0.80 or NHPR<0.90)) is clinically relevant and, the components taken together, represent a sound measure of an effective diagnostic chest pain evaluation<sup>4, 5, 35, 36</sup>. The selection of 12 months is based on the rationale that the longer the duration between the evaluation strategy and an eventual outcome, the less likely it is that the evaluation strategy is directly related to the outcome of interest. In PROMISE, there was a significant reduction in death and MI in the cCTA arm compared to the usual care arm at 12 months, which was no longer significant after a median 25 months of follow-up<sup>5</sup>. The use of this composite clinical endpoint will be critical to assessing the PRECISE hypothesis that a precision evaluation strategy with cCTA and selective FFR<sub>CT</sub> and guideline-recommended medical management without planned testing will yield superior outcomes at lower cost compared with a usual care testing strategy.


CP-907-001-A Jun-29, 2018

#### Rationale for Economic and Quality of Life (QoL) Assessments in PRECISE

Non-invasive diagnostic testing for the evaluation of stable chest pain represents a significant cost to the U.S. and other healthcare systems. In the past when payers in the US have attempted to control costs by reducing the reimbursements provided for diagnostic testing, clinicians responded by increasing the number of tests obtained. An emphasis on generating evidence for cost-savings via a safer and more efficient approach is critical in enhancing value while reducing the financial burden on patients, providers, and the system alike. In addition, this precision-based approach to diagnostic evaluations in CAD participants may result in improvements in the quality of care of our participants. Further, since there has been no prospective trial of guideline-recommended care without planned testing, the ability of such an approach to provide equivalent symptom relief compared with usual care is of great importance and critical to the evaluation of this approach. For these reasons, the potential impact of a precision-based approach on resource use and QoL must be evaluated in PRECISE.

#### IV.E. Rationale for Selection of Testing in Each Arm

#### **Usual Care Arm**

Functional stress testing with stress nuclear, stress echocardiography, and exercise ECG for the diagnosis of CAD is well-established in clinical practice (ACC/AHA 2012 Stable Ischemic Heart Disease guidelines, class I, Level of Evidence (LOE) B)<sup>37</sup>. While stress CMR is less commonly used, it also receives a class IIa, LOE B recommendation in patients who are unable to exercise<sup>37</sup> and is used in some centers. In contrast, it is common for patients to be referred direct to diagnostic angiography without undergoing a functional test. This group represents up to 50% of elective catheterization populations and is thus an important usual care approach to suspected CAD<sup>35, 38, 39</sup>. In order to accurately capture the wide variety of testing strategies available to and used by community clinicians and real-world practice patterns, a usual care strategy arm with site clinician decision-making should include all of the above options. This will improve the generalizability of the trial while accurately capturing the potential impact of the implementation of a precision approach. Use of cCTA as the initial diagnostic strategy is specifically excluded in the usual care strategy arm.

#### Precision Evaluation Arm

PRECISE will evaluate whether a precision evaluation strategy that combines contemporary risk stratification using the PROMISE Risk Tool with functional and anatomic non-invasive evaluation with cCTA with selective FFR<sub>CT</sub> can improve outcomes over usual care in stable chest pain patients while safely deferring further testing in low-risk patients and reducing cost overall. While current guidelines recommend the non-invasive and invasive initial testing approaches for patients with stable chest pain<sup>37</sup>, current practice is known to lead to high rates of ICA without obstructive CAD<sup>6, 40</sup>. Further, although guidelines also recommend no testing in the lowest risk groups (pre-test probability of obstructive CAD <10 or 15%), currently available risk tools result in many clinicians appearing to ignore this recommendation: current patterns of care using available risk stratification tools results in testing populations with a prevalence of obstructive CAD of only 10-20%, and a prevalence of no coronary plaque of >25%<sup>4, 5</sup>. The intervention in PRECISE will triage patients into two risk groups who will be assigned to receive either guideline-recommended medical management without planned testing or cCTA with selective FFR<sub>CT</sub>. The PROMISE Risk


CP-907-001-A Jun-29, 2018

Tool can identify low-risk patients with stable chest pain that would be expected to derive minimal value from noninvasive testing and is superior to either Framingham Risk Score or Diamond and Forrester assessments<sup>33, 34</sup>. cCTA with selective  $FFR_{CT}$  represents a combined functional and anatomic testing modality that can lower the frequency of finding no obstructive CAD at catheterization and thus reduce  $costs^{7,41}$ .

#### IV.F. Randomization Method

Participants who meet all inclusion criteria and none of the exclusion criteria will be randomized in a ratio of 1:1 within a clinical center to either a precision evaluation strategy or usual care using an interactive web or voice-based system (IXRS). Randomization will be stratified by intended first test if randomized to usual care and by classification as minimal vs. elevated risk by the minimal risk model. The randomization scheme within a clinical center will be carried out by the method of random permuted block design with variable block size.

Enrollment in the randomization strata of intended first test being noninvasive (vs. direct to catheterization) will be capped at 90% of the sample size.

Risk will be classified by a risk tool using pre-test clinical characteristics derived in the PROMISE trial and validated in SCOT-HEART. Participants randomized to follow a precision strategy group will be assigned to either guideline-recommended care with symptom and risk factor management and no immediately planned testing (low risk group) or cCTA with selective FFR<sub>CT</sub> (elevated risk of obstructive coronary disease and/or events). Participants randomized to precision evaluation and risk stratified into the low risk group and their providers will be provided informational materials explaining the rationale for this decision and the safety of this strategy based on outcomes of similar participants in the PROMISE trial.

Participants randomized to usual care will undergo either noninvasive stress testing or invasive testing (direct to diagnostic catheterization), as recommended by their managing clinician and agreed to by the participant. Acceptable noninvasive testing options will include exercise electrocardiogram, stress nuclear imaging (including PET), stress MR or stress echocardiogram. The use of cCTA is explicitly excluded as the initial diagnostic strategy in this arm.

In both arms, all subsequent decisions regarding additional testing, medications, and/or procedures will be at the discretion of the responsible clinical care team. Each care team will be provided with informational materials summarizing current standards for test interpretation and preventive care. However, specific medical treatment will not be mandated by the study.

#### IV.G. Diagnostic Evaluations and Subsequent Care

#### <u>Description of Evaluations to be performed</u>

Participants will be assessed per the individual clinicians' routine approach to patients presenting with stable chest pain. Initial evaluation will include an appropriate medical history, physical examination, resting 12-lead ECG, and other routine blood work. A pregnancy test will be required for female participants of childbearing potential, and a creatinine blood test will be required for participants without a recent normal value (within previous 90 days).


CP-907-001-A Jun-29, 2018

At the time of randomization, the site clinician will specify the preferred first diagnostic strategy (noninvasive stress test vs. direct to catheterization) if randomized to the usual care arm and this choice will be used to stratify randomization. Also part of the randomization process, every participant will undergo risk stratification with the PROMISE risk calculator although sites will be blinded to results. Participants randomized to the precision evaluation arm, will be assigned to either no planned testing vs cCTA/FFR<sub>CT</sub> based on results.

Sites will be provided with informational materials outlining standards of care for all noninvasive test interpretation and guideline recommendations for care and symptom and risk factor management. Participant-friendly versions of these material will also be provided to sites, and may be used as handouts.

Symptoms and Quality of Life (QoL) will be assessed by the EuroQoL 5D (EQ-5D-5L) survey to assess overall (generic) health status and the Seattle Angina Questionnaire (SAQ) to assess angina-specific Quality of Life.

#### Equipment, Protocols & Interpretation

All participating sites will use standard equipment and procedures for usual care testing, including diagnostic angiography, stress echocardiography, stress nuclear perfusion imaging, stress CMR, and exercise ECG as defined by current practice guidelines<sup>42-49</sup>. Sites must also use at least 64-slice temulti-detector computed tomography (MDCT) for coronary cCTA<sup>49, 50</sup>. All testing protocols will be in accordance with current best-practice standards<sup>42-48, 50</sup>.

#### Interpretation

The interpretation of all diagnostic tests will be performed in a timely fashion and will capture the presence and extent of findings including diagnosing or excluding CAD (diagnostic angiography), fixed or inducible LV perfusion and wall motion abnormalities (stress echo, cMR and stress nuclear), and functional capacity (in the case of exercise ECG, exercise echo and exercise nuclear). The site interpretation and clinical report of all diagnostic tests, including noninvasive stress testing, cCTA and invasive angiography, will be uploaded through the EDC.

cCTA study interpretation will be carried out by physicians with at least ACC COCATS (Core Cardiology Training Symposium) level 2 training, Society of Cardiovascular Computed Tomography level 2, recognized by the Certification Board of Computed Cardiovascular Tomography, or equivalent<sup>50</sup>. Certification by the Certification Board of Nuclear Cardiology or Board Certification in nuclear medicine or radiology will be considered satisfactory for interpretation of stress nuclear imaging studies. Stress echo and cMR readers also be at least COCATS level 2 trained or equivalent. Prior to being opened to participant enrollment, sites will be certified to ensure that quality cCTA images can be obtained.

#### Referral of precision evaluation cCTA participants for FFR<sub>CT</sub> determinations

Participants randomized to the precision evaluation arm who are determined to be at elevated risk will undergo cCTA as the initial diagnostic strategy according to current best practice standards. Image sets showing at least one 30-90% stenosis in epicardial vessels of 2mm diameter or greater will be promptly sent to HeartFlow for analysis of FFR<sub>CT</sub>. Results will be returned to sites in < 24 hours to enable rapid incorporation into clinical decision making,


#### Subsequent Care

Subsequent care will be provided by the individual site clinicians at their own discretion, with encouragement to follow guideline-based approaches. Information will be provided to the individual sites on diagnostic test interpretation and subsequent management approaches for the various imaging modalities, including relevant guideline recommendations for primary and secondary prevention.

#### Need for testing in low risk participants randomized to the precision care arm

Participants randomized to the precision evaluation arm and determined to be at low risk will be treated for symptoms and risk factor management according to current guideline recommendations. While it is expected that this will resolve symptoms in nearly all cases it is recognized that chest pain will persist in some despite medical treatment. In some cases, additional non-cardiac diagnostic testing may be pursued. In other cases, the site clinician may decide that further cardiac testing is warranted, in which case a cCTA followed by selective FFR<sub>CT</sub> should be performed. Details regarding such decision making will be captured in the case report form.

#### V. STUDY PROCEDURES

#### V.A. Patient Screening for Eligibility

Patients will be screened by site personnel for eligibility and provided information about the study. Patients not meeting inclusion and or having exclusion criteria will be documented as being excluded. Patients meeting inclusion and not meeting any exclusion criteria will be provided an informed consent form to review and sign prior to being randomized into the study.

#### Screening visit (in-person)

At the screening visit, patients will undergo the following:

- Review consent form and have all questions appropriately answered.
- Provide consent by signing the Informed Consent Form
- Review of medical history
- Review of concomitant medications
- Pregnancy test (for females of child-bearing potential)
- Creatinine test (if not done in last 90 days)
- Resting 12-lead ECG (optional, clinical care only)

#### Inclusion Criteria

- 1. Age ≥18 years
- 2. Stable typical or atypical symptoms suggesting possible coronary artery disease (CAD) with further non-emergent testing or elective catheterization recommended to evaluate the presence of suspected CAD
- 3. Safe performance of cCTA:
  - a. Creatinine clearance ≥45 ml/min
  - b. For a female participant of childbearing potential, a pregnancy test must be performed with negative results known within 7 days prior to randomization


CP-907-001-A Jun-29, 2018

- 4. Willingness to comply with all aspects of the protocol, including adherence to the assigned strategy and follow-up visits
- 5. Ability to provide written informed consent

#### **Exclusion Criteria**

- 1. Acute chest pain
- 2. Unstable clinical status
- 3. Noninvasive CV testing within 1 year (for suspected CAD)
- 4. History of known obstructive CAD (prior myocardial infarction, CABG or PCI, stenosis ≥50%), known EF≤40% or other moderate to severe valvular or congenital disease
- 5. Contraindications to cCTA including but not limited to estimated creatinine clearance (GFR) <45 ml/min
- 6. Any condition leading to possible inability to comply with the protocol
- 7. Exceeds the weight or size limit for cCTA or cardiac catheterization at the site
- 8. Life expectancy less than 2 years due to non-cardiovascular comorbidities
- 9. Enrolled in an investigational trial that involves a non-approved cardiac drug or device which has not reached its primary endpoint
- 10. Any condition that might interfere with the study procedures or follow-up

Assessment of CAD risk will be performed during screening to ensure eligibility. It will include:

- General medical history
- Cardiovascular risk factors and comorbidities as well as prior testing or events
- Physical exam
- Laboratory testing

The following major cardiac risk factors will be assessed:

- Age
- Sex
- BP/hypertension
- Diabetes
- Cholesterol (including low-density lipoprotein [LDL], high-density lipoprotein [HDL]), if available
- Smoking status
- Family history
- Sedentary life style
- Obesity (BMI, waist hip ratio)
- Cerebrovascular and peripheral arterial disease (PAD)
- Ankle brachial index (ABI)

#### V.B. Randomization and Enrollment

Once a participant has consented to participate in the trial, participant information will be entered into the database. If a patient is a screen failure, the data that has been collected up until this point for the patient for screening purposes will be entered into the case report forms (CRF) in the electronic data capture (EDC) system. No additional information will be collected after this point for such a patient.


For eligible participants, medical history data will be captured in the EDC. In addition, sites will need to specify the intended first test which would be performed if the participant is randomized to the usual care arm. The participant will then be randomized to either the usual care arm or the precision evaluation arm. Once randomization occurs, the participant is considered enrolled in the study. If randomized to the precision evaluation arm, participants will be further assigned to guideline-recommended without planned testing or cCTA with selective FFR<sub>CT</sub>.

#### V.C. Participant Cohort Assignment

Participant will be randomized to either the usual care arm or the precision evaluation arm within 14 days of screening.

#### **Usual Care Arm**

Participants randomized to the usual care arm will undergo either noninvasive stress testing (exercise electrocardiogram, stress nuclear imaging including PET, stress MR, or stress echocardiogram), with the specific modality at the discretion of the participant's clinician, or invasive catheterization. Performance of cCTA as the initial test is excluded in this arm.

#### **Precision Evaluation Arm**

Participants randomized to the precision evaluation arm will be assigned a management approach based on their PROMISE Risk Score, a risk model based on pre-test clinical characteristics derived from the PROMISE trial and validated in SCOT-HEART<sup>34</sup>. Participants will be assigned to either guideline-recommended medical management without planned testing (low risk) or cCTA with selective FFR<sub>CT</sub> (elevated risk). Participants assigned to the strategy of guideline-recommended medical management without planned testing will be treated with risk-appropriate preventive care and symptom control (including therapeutic trials of anti-anginal medications). Participants and their providers will be provided informational materials demonstrating the safety of this strategy based on pre-test probabilities and the PROMISE Risk Score. Participants with intractable symptoms despite maximal medical management whose clinicians opt for further testing (crossovers) will undergo cCTA with selective FFR<sub>CT</sub>.

Participants undergoing cCTA as the initial test (both assigned or crossover) should have FFR<sub>CT</sub> analysis ordered if cCTA shows at least one 30-90% stenosis in epicardial vessels of 2mm diameter or greater. Image sets will be sent promptly to HeartFlow for analysis and results will be returned to sites in < 24 hours to enable rapid incorporation into clinical decision making.

#### V.D. Participant Follow-Up

Participants will be followed up at 45 (+/-14) days and at 6, 12, and 24 months (+/- 30 days) after enrollment. For North American participants, follow-up after the 45 day visit will be done by phone interviews conducted by the DCRI Outcomes Call Center. For participants outside North America, follow-up will be conducted by the site coordinators.

Activities to be conducted at each follow up contact are described below and in the Schedule of Events.


#### 45(+/-14) day follow-up visit (in-person)

At the 45-day follow-up visit, participants will be asked the following:

- Assessment if any MACE has occurred since enrollment
- CV Update: Review and documentation of any cardiovascular diagnostic test, cardiovascular procedure, or hospitalizations/clinic visits due to cardiovascular symptoms and complications since enrollment
- Review and documentation of concomitant medication changes since enrollment
- Complete the following 3 questionnaires:
  - Seattle Angina Questionnaire
  - EQ-5D-5L Questionnaire
  - Participant Satisfaction Questionnaire
- Collection of
  - Any cardiovascular test both written report and test output
  - Any cardiovascular imaging both written report and image file

#### 6 months (+/-30 days) follow-up contact

At the 6-month follow-up contact, participants will be asked the following:

- Assessment if any MACE has occurred since the 45-day visit
- CV Update: Review and documentation of any cardiovascular diagnostic test, cardiovascular procedure, or hospitalizations/clinic visits due to cardiovascular symptoms and complications since last visit
- Review and documentation of concomitant medication changes since enrollment
- Complete the following 2 questionnaires:
  - Seattle Angina Questionnaire
  - o EQ-5D-5L Questionnaire
- Collection of (may also be done centrally)
  - o Any cardiovascular test both written report and test output
  - Any cardiovascular imaging both written report and image file

#### 12 months (+/-30 days) follow-up contact

At the 12-month follow-up visit, participants will be asked the following:

- Assessment if any MACE has occurred since the 6-month visit/phone call
- CV Update: Review and documentation of any cardiovascular diagnostic test, cardiovascular procedure, or hospitalizations/clinic visits due to cardiovascular symptoms and complications since last visit
- Review and documentation of concomitant medication changes since enrollment
- Complete the following 2 questionnaires:
  - o Seattle Angina Questionnaire
  - o EQ-5D-5L Questionnaire
- Collection of (may also be done centrally)
  - Any cardiovascular test both written report and test output
  - o Any cardiovascular imaging both written report and image file

#### 24 months (+/-30 days) follow-up contact

At the 24-month follow-up visit, participants will be asked to report the following:


- Assessment if any MACE has occurred since the last visit/phone call
- CV Update: Review and documentation of any cardiovascular diagnostic test, cardiovascular procedure, or hospitalizations/clinic visits due to cardiovascular symptoms and complications since last visit
- Review and documentation of concomitant medication changes since enrollment
- Complete the following 2 questionnaires:
  - o Seattle Angina Questionnaire
  - EQ-5D-5L Questionnaire

#### V.E. Cross-over in precision evaluation arm participants

While precision evaluation participants determined to be at very low risk and assigned to the strategy of guideline-recommended medical management with no immediately planned testing are highly unlikely (by definition) to have significant obstructive CAD, their managing clinicians will be encouraged to treat them with guideline recommended preventive care and other medical therapy as deemed appropriate to their clinical circumstances. This is expected to control or eliminate symptoms in most participants. However, additional testing may be warranted for those with intractable or accelerating symptoms despite reasonable medical treatment or other compelling reasons for testing. The reasons for this will be carefully documented in the eCRF. Unless there are urgent or emergent indications to proceed with invasive testing, all such participants who require testing will have a cCTA followed by selective FFR<sub>CT</sub> rather than either stress testing or elective invasive catheterization.

#### V.F. Participant Withdrawal

In accordance with the Declaration of Helsinki, each participant is free to withdraw from the study at any time. Investigator(s) also have the right to withdraw participants from the study in the event of illness or other reasons concerning the health or wellbeing of the participant, or in the case of lack of cooperation. Should a participant decide to withdraw or should the investigator(s) decide to withdraw the participant, all efforts will be made to complete and report the observations up to the time of withdrawal as thoroughly as possible. If possible, a complete final evaluation at the time of the participant's withdrawal should be made. The reason for withdrawal must be noted in the eCRFs.


DocuSign Envelope ID: C68B333A-7FC7-483F-BE3F-204B8CC0896B

PRECISE Protocol

CP-907-001-A Jun-29, 2018

#### V.G. Schedule of Assessments

| | Screening | Randomization<br>Day 1 | Day 45<br>( <u>+/-14 d)</u> | <b>6-mo</b> .<br>( <u>+/- 30d)</u> | <b>12-mo</b> .<br>(+/- 30d <b>)</b> | <b>24-mo</b> . (+/- 30d) |
|---|---|---|---|---|---|---|
| Informed consent | Х | | | | , , | , |
| Medical history | Х | | | | | |
| Cardiovascular update 1 | | | Χ | Χ | Х | Х |
| Concomitant medications | Х | | Χ | Χ | Х | Х |
| Cardiovascular Risk factors (including PROMISE risk tool data entry for randomization) | Х | | | | | |
| Pregnancy test <sup>2</sup> | Х | | | | | |
| Creatinine <sup>3</sup> | Х | | | | | |
| Resting 12-lead ECG <sup>4</sup> | Х | | | | | |
| QoL evaluation: SAQ, EQ5D-5L | Х | | Х | Х | Х | |
| Participant Satisfaction Questionnaire | | | Х | | | |
| Randomization | | X | | | | |
| Initial diagnostic invasive or noninvasive test performed (if assigned) | | Prior to 45 day<br>visit | | | | |
| Cardiac imaging/testing clinical report and image collection | | | Х | Х | Х | |
| Interval assessment for CV events and testing | | | Х | Χ | Х | Х |
| Endpoint assessments | | | Х | Χ | Х | Х |

During cardiovascular update, if participants have received an additional diagnostic test, a cardiovascular procedure or have been hospitalized since the last visit, additional data will be collected


For a female participant of childbearing potential, a pregnancy test must be performed with negative results known within 7 days prior to randomization 2.

<sup>3.</sup> 4.

Creatinine blood draw required only for participants without a recent normal value (within previous 90 days)
Resting 12-lead ECG preferred in last 30 days (optional, clinical care only)
Use of specific medications such as beta blockers, ACE inhibitors/ARBs, statins, aspirin, and antiplatelet agent 5.

CP-907-001-A Jun-29, 2018

#### VI.ADDITIONAL ASSESSMENTS AND SUBSTUDIES

#### VI.A. Quality of Life Assessments

A short battery of instruments will be used to provide a relevant assessment of health-related quality of life that will capture the most likely health benefits to be associated with the precision strategy while not being burdensome to study participants. Quality of life (QoL) assessments will be conducted at baseline, 45 days, 6 months, and 12 months. Chest pain specific QOL will be assessed with the Seattle Angina Questionnaire (SAQ). While the full instrument has 19 items covering 5 dimensions of the impact of chest pain on QoL, we will use the scales for physical limitations, angina frequency, and disease perception/quality of life (14 items total) <sup>1</sup>. These three scales will also allow calculation of the recently described 7-item short SAQ<sup>2</sup>. The SAQ has been used as the primary disease-specific QoL outcome measure in a number of major clinical trials (including COURAGE, PROMISE, and ISCHEMIA) and is useful for this trial because it assesses chest pain and its impact on functioning and well-being regardless of whether the symptoms are due to coronary disease or are non-coronary. Since many participants in this study will be found not to have significant coronary disease and will be provided with that reassuring finding, the SAQ will allow us to assess the extent to which such information is associated with changes in the 3 dimensions noted above.

Overall health status will be assessed briefly using the EQ-5D-5L, a standardized generic measure that can also be used to link specific health states to general population-based utilities<sup>5</sup>. The EQ-5D-5L consists of two parts: (1) a descriptive assessment of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each of which can take one of five responses corresponding to the level of severity within each dimension, and (2) a self-rating 0-100 "thermometer" of current health-related quality of life.

#### VI.B. Economic and Resource Utilization Assessments

The primary economic analyses in PRECISE will be performed from the perspective of the US health care system. Detailed information regarding the quantity and cost of health care services received by participants in each treatment group will be collected prospectively as part of the trial. Relevant health care resource consumption during initial testing through 2-year follow-up will be collected on the clinical trial electronic case report form (eCRF). (The cost of acute and non-acute hospital care will be derived from billing data collected from patients enrolled at US sites.) Physician and other outpatient care reported in the eCRF will be valued using secondary sources. Primary resource use and cost comparisons will be based on participants enrolled in the US. Secondary analyses will examine the consistency of treatment related differences in resource use in the US with the sites outside the US.

#### VI.C. Imaging and other Cardiac Assessments

For all participants in either arm in whom an invasive coronary angiogram is performed within the first 12 months, procedural reports and angiographic images will be uploaded via the electronic data capture (EDC) system to create an angiographic image repository. In addition the report, as well as imaging and / or graphic data from any procedures performed to assess stenosis significance or severity such as, FFR, NHPR, IVUS, OCT should be uploaded. Similarly, for all participants receiving cCTA imaging within the first 12 months, the cCTA images and reports will CONFIDENTIAL

be uploaded via the EDC system to create an image repository. A core lab may be added to analyze these images. Data collection for these elements will be coordinated by the DCRI Outcomes Group for North American patients followed by the call center and by site coordinators for all other sites.

#### VII. ENDPOINT DETERMINATION, SAFETY, AND MONITORING

#### VII.A. Primary Endpoint Definitions

#### Major Adverse Cardiovascular Events (all cause death, non-fatal myocardial infarction)

#### All cause death

All cause death is defined as death resulting from any cause. In addition, the cause of death will be adjudicated, including cardiovascular death defined as death due to myocardial infarction, sudden cardiac death, heart failure, stroke, cardiovascular procedures, cardiovascular hemorrhage, or death due to other cardiovascular causes <sup>51</sup>.

#### Myocardial infarction

Acute myocardial infarction (MI) is defined as having evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia<sup>51</sup>. Specifically, MI is defined as having:

1) Typical rise and/or gradual fall in cardiac biomarker level (cardiac troponin preferred) with values exceeding the 99<sup>th</sup> percentile of the institutional upper limit of normal (ULN) (generally 2x the ULN)

#### AND either:

2) Clinical presentation defined as typical cardiac ischemic type pain/discomfort or dyspnea felt to be due to ischemia and consistent with the diagnosis of myocardial ischemia and infarction

Or

3) ECG manifestations of acute myocardial ischemia (in absence of left ventricular hypertrophy and left bundle branch block) including evolving ST elevation, ST depression, T-wave changes, new pathological Q-waves (R waves in V1-2) in at least two consecutive leads or new left bundle branch block.

A complete definition of the criteria for MI can be found in the 2017 Cardiovascular and Stroke Endpoint Definitions for Clinical Trials<sup>51</sup>. Peri-procedural infarctions are defined as greater than 3x ULN for serum CK-MB for PCI and greater than 5x ULN for CABG.

## <u>Cardiac catheterization without obstructive coronary artery disease (diameter stenosis <50%,</u> any FFR >0.80 or NHPR ≥0.90)

Cardiac catheterization without obstructive coronary artery disease will be defined as the absence of any  $\geq 50\%$  stenosis or hemodynamic indication of significance in any major epicardial vessel including side branches  $\geq 2$  mm in diameter, as determined by the clinical site interpretation.


#### VII.B. Secondary Endpoint Definitions

#### Hierarchical analysis

Finkelstein and Schoenfeld (FS) or Pocock's win ratio analysis of primary endpoint is defined in section VII B Statistical Analysis Plan.

#### Resource use

Resource use is defined as counts and types of baseline testing, follow up testing, diagnostic and therapeutic procedures, and both inpatient and outpatient care at 12 months. Costs from the US perspective will be estimated.

#### Quality of Life Metrics

Quality of Life assessments to be completed by the participants are the Seattle Angina Questionnaire and the EQ-5D-5L.

#### Death

Death will be categorized as all-cause, cardiovascular, non-cardiovascular.

#### Myocardial infarction

Myocardial infarction will be characterized according to Universal MI definition subtypes as Type 1, 2, 3, 4a, 4b, 4c and 5.

#### Hospitalizations

All, cardiovascular, non-cardiovascular, and for progressive or unstable angina. Urgent and unscheduled hospitalizations for other cardiovascular causes that do not meet the criteria for the specific events listed above will be classified as hospitalization for other cardiovascular causes (e.g., hospitalization for cardiac chest pain that does not meet the criteria for MI, hospitalization for arrhythmias, hospitalization for pulmonary embolism). Non-cardiovascular hospitalization are defined as any hospitalization whose primary cause is not thought to be CV in nature.

#### Preventive medication use

Information on preventive medication use will be acquired at study entry and 45 days. Participants with a clear clinical indication for use of ASA/antiplatelet agents and or, statins eg: hyperlipidemia, diabetes, documented CAD, will be characterized according to use/nonuse for each medication class.

#### DECISION co-primary end point

MACE, defined as all-cause death myocardial infarction, or ischemia-driven revascularization at 24 months as defined by the DECISION trial.

#### **DECISION** co-primary end point

All-cause death, MI, all follow-up unplanned revascularization procedures, cardiac catheterizations without actionable findings at 24 months as defined by the DECISION trial.


#### PRECISE primary endpoint at 24 months

The PRECISE primary endpoint will be determined at 24 months.

#### Radiation safety endpoint – cumulative dose at 1 year

The cumulative radiation exposure over the 12 months following enrollment will be calculated based on the participant's exposure to radiation for cardiovascular care from one or more of the following modalities. For cCTA, the administered radiation dose (computed tomography dose index volume and dose length product for cCTA) will be recorded by the individual sites. For stress nuclear imaging, the radiotracer dose(s) will be collected and converted to equivalent radiation doses for comparison to cCTA. For ICA, the radiation dose from fluoroscopy administered will be recorded by sites and converted using standardized approaches to allow for comparison to radiation from cCTA. In instances in which the information required to assess actual dose is not available, a standard dose based on accepted average exposures will be imputed for that form of testing. Cumulative radiation exposure from additional cardiac testing and procedures during the entire follow-up period will also be collected.

#### Catheterization efficiency

The proportion of invasive cardiac catheterization patients who undergo revascularization (PCI or CABG) within 6 months of enrollment will be determined.

#### VII.C Testing Complications and Reporting

The study intervention is the implementation of a precision evaluation strategy compared to usual care evaluation in non-acute chest pain participants with no history of CAD or recent testing whose clinicians recommend non-emergent non-invasive testing or ICA. Since all trial procedures represent standard of care for the eligible study population, there are no specific safety events associated with investigative procedures in this trial. However, there are known complications from these clinically recommended tests and procedures which are outlined below. These complications will be reported by site personnel.

#### For Precision Evaluation Strategy

#### For Guideline-recommended Medical Management

While participants assigned to the guideline-recommended care with no planned testing arm will have exceedingly low risk of events and are predicted to derive minimal or no value from noninvasive testing<sup>33, 34</sup>, there is a very small risk of missing left main or 3-vessel disease for which revascularization may be life-prolonging.

#### For cCTA with selective FFR<sub>CT</sub>:

Mild contrast reaction such as rash and hives.

- 1. Severe contrast reactions including anaphylaxis or death occurring within 24 hours of contrast administration.
- 2. Extravasation of contrast into the surrounding tissue of the extremity where contrast was administered intravenously.
- 3. Symptomatic bradycardia or hypotension in relation to beta blockade or nitrates administered for cCTA.


4. Acute bronchospasm following beta blockade administered for cCTA.

#### For Usual Care (noninvasive or invasive testing)

For exercise testing including during stress echo or stress nuclear (including PET):

- Hypotension defined as systolic BP less than 80 mmHg or fall in systolic BP >20 mmHg
- 2. Stress-induced symptoms or ECG changes that do not resolve within 20 minutes
- 3. Rapid atrial fibrillation that does not slow or convert with standard interventions
- 4. Ventricular tachycardia
- 5. Hospital admission not otherwise captured by pre-specified study endpoints, due to one of the above

#### For stress nuclear (including PET):

1. Any adverse reactions potentially related to the use of vasodilators such as adenosine, regadenoson, or dipyridamole

#### For stress echo:

- 1. Any stress-induced wall motion abnormality that does not resolve within 20 minutes
- 2. Any adverse reaction to echo contrast
- 3. Any adverse reaction to dobutamine, including sustained ventricular tachycardia or other tachyarrhythmias

#### For stress cardiac MRI:

- 1. Any adverse reactions potentially related to the use of vasodilators such as adenosine, regadenoson, or dipyridamole
- 2. Any adverse reaction to MRI contrast agents, including gadolinium-based agents

#### For cardiac catheterization:

- 1. Any adverse reactions potentially related to the use of sedatives, local anesthetics, contrast agent or other medication's
- 2. Any adverse reactions potentially related to arterial puncture and wire/catheter introduction
- 3. Any adverse reaction to coronary catheterization including dissection, embolization, stroke, malignant arrhythmias and asystole, and death

#### VII.D. Independent Clinical Event Adjudication Committee

An independent clinical event committee (CEC) will be responsible for the blinded review and adjudication of the primary endpoint. The CEC will settle any disputes with committee review and discussion. Any uncertainty regarding the finding of cardiac catheterization without obstructive disease will prompt review of the original cardiac catheterization images for further independent adjudication. Collection of medical records and other documentation required for CEC reviews will be coordinated by the DCRI call center for North American participants and by site coordinators for participants in all other regions.


CP-907-001-A Jun-29, 2018

#### VII.E. Data and Safety Monitoring Board

An independent Data and Safety Monitoring Board (DSMB) will be appointed to monitor participant safety and to review study performance. The DSMB will periodically review the study data and assess participant safety and adherence to the study protocol. The DSMB will define the operating guidelines and processes for study evaluation, interim analyses, event triggers for unscheduled review; these will be agreed upon at the initial meeting of the DSMB. Periodic reports will be prepared by HeartFlow (or its designee) for the DSMB on based on the operational plan outlined by the DSMB charter. The DSMB will make its recommendations to the study Steering Committee and the sponsor following their meeting. Details on statistical stopping rules guidelines will be provided in the DSMB charter.

#### **VIII. Statistical Methods**

Separate, complete Statistical Analysis Plan (SAP) documents will be prepared for the clinical outcome analyses and the economics and quality of life (EQOL) outcomes.

#### VIII.A. Sample Size Determination and Statistical Power

Sample size and power calculations for this study are based on the hypothesis that the precision evaluation arm is superior to the usual care arm on the time-to-first event of the composite MACE endpoint (defined as: all-cause death, non-fatal MI) or invasive cardiac catheterization without obstructive CAD (obstructive CAD defined as diameter -stenosis ≥50%, FFR≤0.80 or NHPR <0.90). Time to event analysis will use the date of the event, including the date of catheterization which is used to determine the absence of obstructive CAD. Assuming 10% of usual care participants will receive angiography as a first test results in an 8% primary endpoint event rate at 1 year in the usual care group and 5% (absolute) event rate in the precision care group (i.e., 37.5% relative effect size) with 30% assigned to guideline-recommended care with symptom management and no planned testing. Assumptions used in the primary endpoint event rate calculations (i.e. 8% vs. 5%) were: an overall 10% will not receive randomized testing and within the precision evaluation arm, 30% of those assigned to guideline-recommended care will cross over to cCTA with selective FFR<sub>CT</sub>.

Enrolling 1050 patients per group (2100 total participants) would provide at least 90% power to detect a relative risk reduction of 37.5% in the precision evaluation arm. Sample size calculations are based on the log-rank test <sup>52</sup> with 12-month accrual period, a minimum 12-month follow-up (i.e., last participant will be followed for at least 12-months), 10% attrition rate (i.e., lost to follow-up, dropouts) and a two-sided type I error rate of 0.05.

| 1-yr event rate in precision evaluation arm | Power | Total<br>number of<br>participants<br>needed | Total number of MACE events needed |
|---|---|---|---|
| 5% | 85% | 1792 | 173 |
| (37.5% effect size) | 90% | 2096 | 202 |
| (67.670 611661 6126) | 95% | 2592 | 250 |

**Table** shows total number of participants needed for 85%, 90% and 95% power. Although, this is not an event-driven study, the table below also provides total number of MACE needed.


Power curves (Figure: Long-Rank for Two Survival Curves) provide total sample size needed for several relative effect size (i.e., 1-hazard ratio) scenarios.



Figure: Long-Rank for Two Survival Curves

#### VIII.B. Statistical Analysis Plan

#### Analysis of the Primary Endpoint

The primary endpoint of this study is based on time-to-first occurrence of any of the MACE components, which is defined as a composite of all-cause death, non-fatal MI or invasive cardiac catheterization without obstructive CAD (obstructive CAD defied as diameter stenosis ≥50%, FFR≤0.80, or NHPR<0.90). The time from randomization to the first event among the components of the MACE endpoint will be measured (in days) for those who experienced an event and calculated as the date of the first event minus the date of randomization. For participants who do not experience any of the MACE component events or who withdraw consent or drop out of the study before experiencing an event, time from randomization to the date of last contact will be used in the analysis, and those participants will be considered as censored observations in the time-to-event analysis.

The primary and secondary endpoint comparisons between the randomized groups in this study will be performed according to the principle of "intention-to-treat" (ITT); that is, participants will be analyzed according to the treatment arm to which they were randomized, regardless of subsequent crossover or post-randomization strategy.

The log-rank test<sup>53</sup> will be the primary analytic tool for statistically assessing outcome differences between the two randomized treatment strategies with respect to the primary composite endpoint. Cox proportional hazards model<sup>54</sup> will be used to estimate the hazard ratio (HR) and 95% confidence interval (CI) summarizing the difference in outcome between the two randomized arms, using treatment as the only predictor in the model. Proportionality assumption in the Cox model (i.e., constant hazard over time) will be checked and tested.

Cumulative event rates will be calculated according to the method of Kaplan and Meier<sup>55</sup> for each randomized arm as a function of time from randomization, and the estimated event probabilities


will be displayed graphically. Adjusted HR and its 95% CI will be estimated using Cox proportional hazards model by including pre-specified baseline risk factors as covariates in the model.

A sensitivity analysis for the primary composite MACE endpoint will be conducted using the method of "win-ratio"<sup>56</sup>. The win-ratio method of Pocock et al is an extension of Finkelstein and Schoenfeld rank-test method<sup>57</sup> which order-rank composite endpoints based on their clinical importance. More details on primary, secondary and sensitivity analyses will be provided in the complete Statistical Analysis Plan (SAP).

#### Subgroup analyses

If there is an overall difference in MACE outcome between treatment strategies, subgroup analyses will be performed to assess whether the intervention effect is consistent across all participants, or whether it varies according to specific participant characteristics. In particular, these analyses will focus on whether the relative intervention effect compared to usual care differs according to the following baseline variables:

- Low risk vs. elevated risk by PROMISE Risk score
- Intended first test: functional vs. invasive
- Sex (male vs. female)
- Age (<65, 65 to 74, and >75 years)
- History of diabetes
- Presentation: primary symptom (chest pain vs. other), SAQ angina score (daily/weekly angina at baseline versus less frequent)
- Geographic region (US, Canada, Europe, Other Regions)

These analyses will utilize the Cox model and will be accomplished by testing for interactions between the randomized treatment strategy and the specific baseline variables listed above. In addition to the formal assessment of treatment by covariate interactions, the effect of the treatment strategy characterized by a hazard ratio and 95% confidence interval will be calculated and displayed using a forest plot for the subgroups of participants defined by the variables listed above. These descriptive hazard ratios will be carefully interpreted in conjunction with the formal interaction tests.

The effect of the treatment strategy may also be examined in other subgroups of clinical interest in addition to those listed above.

#### Analysis of the Secondary Endpoints

The secondary endpoints listed in section III.C. Secondary Endpoints that are measured as time-to-event will be analyzed using the same statistical methods used for the primary efficacy endpoint (Section VI.A. Primary Endpoint Definitions). Specifically, the log-rank test will be the primary analytic tool for statistically assessing mortality differences between the two randomized treatment strategies. A hazard ratio and 95% confidence interval summarizing the difference in outcome between the two randomized arms will be computed using the Cox model.

Participant deaths will be classified by the Clinical Events Committee (CEC) as to whether the mode of death was due to a cardiovascular (CV) cause. If insufficient source documents are obtained to allow CEC adjudication of the cause of death, and the CEC classifies the cause of death as "unknown," then the site-reported cause of death (if available) will be used. If neither the site nor the CEC can provide a classification of the cause of death, the death will not be


considered as a cardiovascular death. As supplemental analyses, however, this endpoint will also be examined using (a) only the deaths classified by the CEC as cardiovascular, and (b) using deaths classified by the CEC as cardiovascular, but also including any deaths in the cardiovascular category that are classified as unknown by the CEC.

Competing risks methodology of Fine and Gray<sup>58</sup>, where death due to a non-cardiovascular cause is considered as a competing risk. This methodology, rather than treating non-cardiovascular death as a censoring event, makes incidence use of the cumulative function, and is performed within the proportional hazards framework using the marginal failure sub-distribution associated with the event of interest (cardiovascular death). Similar analyses will be conducted for time-to-event endpoints in which death is not part of the endpoint of interest.

#### Analysis of Resource Use Endpoints

For the Economics outcomes, we will compare resource use at 12 months between treatment arms by intention-to-treat. All-cause hospitalizations, cardiovascular hospitalizations, ER visits not resulting in hospitalization, and major outpatient procedures will be enumerated. In addition, we will examine length of stay by intensity of care, numbers of CTAs, noninvasive stress tests (stress perfusion imaging, stress echocardiography, exercise electrocardiography, stress cardiac magnetic resonance imaging), invasive tests (invasive coronary angiography, invasive fractional flow reserve or equivalent, optical coherence tomography, intravascular ultrasound), coronary revascularization procedures (coronary artery bypass graft surgery (CABG), percutaneous coronary intervention (PCI), number of coronary stents), and cardiac medications (beta blockers, aspirin, statins, antiplatelet medications).

Confidence intervals for differences will be estimated using the bootstrap approach. Differences in resource use will be interpreted in the context of the trial clinical results, looking for both consistency and plausibility. Descriptive comparisons of intensity of care/resource consumption according to clinical variables defining subgroups of interest will be performed. The primary economic analyses will focus on the US enrollment and in secondary analyses, resource use patterns for all patients enrolled in the trial will be compared by intention-to-treat to develop an understanding of the degree to which treatment related differences in the trial are region dependent.

#### Analyses of Medical Costs (US participants)

To compare medical costs between treatment arms, we must: 1) assign costs to all medical resources consumed during the study period; 2) compute mean costs by treatment group (defined by the principle of intention-to-treat); and 3) calculate the difference in mean costs between treatment arms and generate confidence intervals.

#### A) Derivation of Cost Estimates.

The cost of US hospital-based care will be estimated by applying hospital-specific, revenue center level cost-to-charge ratios to empirical billing data collected during the study. This approach, which has been used successfully in numerous previous clinical trials including the PROMISE trial takes advantage of the objective, detailed account in hospital bills of services provided to patients, and recalibrates hospital charges to more closely reflect costs. Based on experience in similar studies, we anticipate having complete billing data for 95% of patients treated in hospitals that generate bills. For the small percentage of patients without billing data, we will impute costs using a generalized linear model developed using study data. In this model, the dependent variable will be defined as total cost, and independent variables will include resource use elements available in the case report form, such as number of hospitalized nights

CONFIDENTIAL


by intensity of care and number of relevant high cost procedures. Coefficients for model parameters will be estimated using study data of patients with complete costs and then used to predict costs for patients without billing information.

The cost of stays at non-acute care facilities will be estimated by multiplying the length of stay by the corresponding per-diem/reimbursement rate.

Costs for physician services will be estimated by mapping major inpatient and outpatient procedures and services recorded on the case report form to appropriate CPT codes in the Medicare Fee Schedule. We will also assign rounding fees for inpatient stays based on type of unit.

Costs for diagnostic testing procedures done in an outpatient or standalone facility will be derived from secondary sources available to the DCRI Outcomes Group at the time of study analysis.

The cost of medications of interest/relevance will be estimated on the basis of medication use recorded in the eCRF and unit costs by medication type and class, based on current estimates of acquisition cost.

#### B) Cost Comparisons

Primary statistical comparisons of costs between the two treatment groups will be performed using the intention-to-treat principle in the US cohort. A nonparametric partitioned estimator will be used to estimate diagnostic strategy-specific, 2-year medical costs with 8 partitions corresponding to 3-month intervals following randomization. Comparisons between the two testing strategies will be made using a normal approximation with standard errors estimated using the bootstrap approach. Bootstrapping will be performed using 10,000 repetitions, with percentile-based confidence intervals reported. The primary cost comparison will be made for cumulative costs at 12 months. The primary effect size will be the mean cost difference between the two arms with 95% confidence intervals. P values will be calculated for selective comparisons, with a "significant" p value equivalent to a 95% confidence interval that excludes 0. No adjustment in significance levels for multiple comparisons will be used.

Differences in cost will be interpreted in the context of the trial clinical results, looking for both consistency and plausibility. Costs will be presented both overall and by category (e.g., inpatient hospitalization, outpatient procedures, concomitant medications, non-acute institutional care). Hospitalizations will be classified as cardiovascular or non-cardiovascular by the Clinical Events Committee. For illustrative purposes, we will use bootstrap methods to plot the probability of a difference in total costs greater than arbitrary thresholds of interest (such as \$500, \$750, or \$1000).

#### C) Cost Sensitivity Analyses

In secondary sensitivity analyses, we will apply US unit costs to all resource use of all patients and compare costs between treatment groups across all patients enrolled in the trial. While US unit costs may not reflect the absolute or relative costs of health care services internationally, their application to all patients will permit a weighted aggregation and comparison of resource use in the total trial population. In this manner, the effect of overall patterns of resource use in the US cohort versus ex-US on cost differences by treatment group can be assessed. We will also perform a per protocol analysis of costs.

#### Analyses of Quality of Life Outcomes

For each of the QOL measures examined in this study, we will provide simple descriptive and


comparative analyses by intention-to-treat. To address the multiple comparisons problem arising from testing each individual scale and time point separately, we propose two complementary approaches. First, we will pre-specify the angina frequency scale from the SAQ as the primary QOL comparison of interest and assign all other comparisons to a secondary (supportive) status. Second, we will use a repeated-measures mixed model with the baseline score as a covariate, Day 45, Month 6, Month 12, Month 18, and Month 24 responses included as outcome variables, and time as a fixed variable. Restricted maximum likelihood estimation will be used to model all available data from each subject without imputing missing values. An unstructured covariance matrix will be used.

Point estimates for each diagnostic strategy arm and strategy arm mean differences (precision strategy – usual care) with 95% confidence intervals (CIs) will be generated for each time point. The primary assessment will be based on the strategy arm difference at Month 12. Additional analyses will examine the intervention effect at the other contact time points. Additionally, the intervention effect will be averaged across all the follow-up time points. The estimated intervention difference and 95% CIs will be obtained using the ESTIMATE Statement in SAS PROC MIXED.

We expect to have analyzable data on ≥95% of survivors at each follow-up interview, and, with 90%+ data collection (945+ patients per treatment group), consistent with our past performance in trials of this size and complexity and using similar methods, even accounting for loss of data due to death or incapacity, we should have 90% or greater statistical power to detect clinically significant differences in our major QOL measures.

Major QOL subgroups to be examined will be those prespecified for the clinical analysis of this trial. In addition, we will use baseline angina frequency from the SAQ to create a subgroup of subjects with daily or weekly chest pain versus those with less frequent symptoms.

#### IX. ETHICAL CONSIDERATIONS AND RISK ANALYSIS

#### IX.A. Ethical Considerations

PRECISE will be conducted in accordance with the recommendations for human research from the 18<sup>th</sup> World Medical Assembly, Helsinki 1964. All potential sites will obtain Institutional Review Board (IRB) or Ethics Committee (EC) approval of the protocol, the associated consent form and any participant facing recruitment tools. Written informed consent will be obtained from each patient before any study procedures are performed. Patients will have the option to consent for the study after receiving a full explanation of the risks, benefits, and available diagnostic options, with the right to refuse participation. Clinicians will have the option to pursue alternative diagnostic pathways if they deem it to be in the best interest of the patient, with the reason for study protocol deviation documented. Participants can withdraw from the study at any time.

#### IX.B. Study Risks and Benefits

#### Potential Risks


Participation in PRECISE does not present any extra risks other than the risks associated with the clinically indicated care recommended by the participant's treating physicians to evaluate and treat symptoms suggestive of CAD. As all approaches included in the trial are recognized as standard of care, the risk associated with the trial can be described in detail by the treating physician.

Noninvasive diagnostic imaging is generally considered a safe and effective diagnostic approach. FFR<sub>CT</sub> does not pose any additional risk to participants beyond the performance of cCTA itself. It does offer the potential benefit to participants of the recognition of hemodynamically significant lesions (FFR  $\leq$ 0.80 or NHPR <0.90) that may not demonstrate anatomic significance (<50% diameter stenosis) and avoidance of unnecessary revascularization of  $\geq$ 50% lesions that are not hemodynamically significant (FFR>0.80).

The risks of guideline-recommended care without planned testing in the lowest risk participants has not been extensively studied prospectively. However, validation of the PROMISE Risk Tool in SCOT-HEART indicate that participants in this risk category have a CV death/MI event rate <1%/year, similar to the event rate observed in an age and sex matched US population. While the risk of guideline-recommended care without planned testing in the precision evaluation arm has not been quantified prospectively it is not expected to differ from the excellent outcomes noted above in such patients who do undergo testing. Further, participants with continued symptoms not controlled by medications will be permitted to cross over to the precision strategy arm and receive, cCTA with selective FFR<sub>CT</sub>.

#### Potential Loss of Confidentiality

In any clinical trial, there is a possible risk of loss of confidentiality. To prevent this from occurring, HeartFlow has strict procedures in place to ensure that all study data are confidential and anonymized except as required for centralized follow-up data collection for North America, which will be performed by the DCRI Outcomes Call Center. For all data transferred from enrolling sites or from the Call Center, participants will be identified only by unique patient identifiers. Data transmitted will not contain any protected health information and participants will be identified only by unique patient identifiers. Data transmitted will not contain any protected health information. All applicable study data will be transferred in a secure manner and in accordance with applicable regulations.

#### Potential Benefits

The PRECISE results should improve the care of future patients recommended for additional evaluation for suspected CAD. In addition, the trial will deliver high-quality data on radiation exposure, incidental findings, and other clinically important "side effects" of the evaluation and management strategies that will be examined in a large real-world experience. All participants may benefit from increased contact with health care providers due to study-required visits.

### X. DATA HANDLING AND QUALITY ASSURANCE

#### X.A. Completing and Signing Case Report Forms

Electronic CRFs will be employed. Trained site personnel or the trained DCRI Outcomes Group will enter data into the eCRFs. Data changes and corrections should be done within the electronic system. The audit trail will record all changes made, the date and time of the CONFIDENTIAL


correction, the person making the change and a reason for the change. The appropriate electronic signature will be provided by the investigator as indicated.

#### X.B. Clinical Data Management

The sponsor or its designees will be responsible for the handling, processing, and quality control of the data in compliance with all applicable regulatory guidelines.

The training of clinical site personnel and the DCRI Outcomes Group on eCRF completion will be the responsibility of the sponsor or its designees. To ensure uniform data collection, a Case Report Form Guide will be created to assist with eCRF completion. All clinical site research coordinators will undergo site initiation training to become thoroughly familiar with the protocol, case report forms, and with methods of data verification.

#### X.C. Archiving of Data

All study documentation at the investigator site and sponsor site will be archived in accordance with ICH GCP. It is HeartFlow's policy to retain the data collected in this clinical study for a minimum of 5 years after termination of the study. Clinical sites will be asked to retain the data for at least 2 years following completion of the study or longer as required by local laws.

#### XI. STUDY MONITORING, AUDITING, AND INSPECTING

HeartFlow or its designees will monitor this clinical study to check the adequacy of clinical site staff and facilities, and to ensure adherence to the protocol, study procedures, and applicable regulations. In accordance with ICH E6 GCP guidelines, the clinical site monitor will also assess proper eCRF completion and source document retention. The investigator and clinical site staff are expected to provide adequate space for monitoring visits and to allocate sufficient time to permit adequate review of the study's progress. The investigator will permit study-related monitoring, audits, IRB review, and regulatory inspection(s), providing direct access to source data/documents and study-related facilities (e.g., pharmacy, diagnostic testing and laboratories).

#### XI.A. Study Monitoring

Study monitoring will be performed in accordance with ICH E6GCP, this protocol, and applicable local regulations. A Clinical Monitoring Plan will be written at the outset of the study to provide project-specific operational guidelines for the clinical monitoring process and procedures, define responsibilities of the Site Management/Monitoring Team, which will in turn ensure the quality and integrity of data collected.

#### XI.B. Auditing and Inspecting

HeartFlow quality assurance personnel and/or their designee(s) may conduct audits at the study site(s). Audits may include, but not be limited to: audit trail of data handling and processes, SOPs, presence of required documents, the informed consent process, and comparison of case report forms/database with source documents. The investigator agrees to accommodate and participate in audits conducted at a reasonable time in a reasonable manner, as needed.


CP-907-001-A Jun-29, 2018

#### XII. References

- 1. Benjamin EJ, Virani SS, Callaway CW, Chamberlain AM, Chang AR, Cheng S, Chiuve SE, Cushman M, Delling FN, Deo R, de Ferranti SD, Ferguson JF, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Lutsey PL, Mackey JS, Matchar DB, Matsushita K, Mussolino ME, Nasir K, O'Flaherty M, Palaniappan LP, Pandey A, Pandey DK, Reeves MJ, Ritchey MD, Rodriguez CJ, Roth GA, Rosamond WD, Sampson UKA, Satou GM, Shah SH, Spartano NL, Tirschwell DL, Tsao CW, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS and Muntner P. Heart Disease and Stroke Statistics-2018 Update: A Report From the American Heart Association. Circulation. 2018;137:e67-e492.
- 2. World Health Organization. Cardiovascular diseases (CVDs).(Fact-sheet) 2017.
- 3. Fordyce CB and Douglas PS. Optimal non-invasive imaging test selection for the diagnosis of ischaemic heart disease. *Heart (British Cardiac Society)*. 2016;102:555-64.
- 4. Newby D, et al. CT coronary angiography in patients with suspected angina due to coronary heart disease (SCOT-HEART): an open-label, parallel-group, multicentre trial. *Lancet (London, England)*. 2015;385:2383-91.
- 5. Douglas PS, Hoffmann U, Patel MR, Mark DB, Al-Khalidi HR, Cavanaugh B, Cole J, Dolor RJ, Fordyce CB, Huang M, Khan MA, Kosinski AS, Krucoff MW, Malhotra V, Picard MH, Udelson JE, Velazquez EJ, Yow E, Cooper LS and Lee KL. Outcomes of anatomical versus functional testing for coronary artery disease. *N Engl J Med*. 2015;372:1291-300.
- 6. Patel MR, Peterson ED, Dai D, Brennan JM, Redberg RF, Anderson HV, Brindis RG and Douglas PS. Low diagnostic yield of elective coronary angiography. *N Engl J Med*. 2010;362:886-95.
- 7. Douglas PS, De Bruyne B, Pontone G, Patel MR, Norgaard BL, Byrne RA, Curzen N, Purcell I, Gutberlet M, Rioufol G, Hink U, Schuchlenz HW, Feuchtner G, Gilard M, Andreini D, Jensen JM, Hadamitzky M, Chiswell K, Cyr D, Wilk A, Wang F, Rogers C and Hlatky MA. 1-Year Outcomes of FFRCT-Guided Care in Patients With Suspected Coronary Disease: The PLATFORM Study. *Journal of the American College of Cardiology*. 2016;68:435-445.
- 8. Fordyce CB, Newby DE and Douglas PS. Diagnostic Strategies for the Evaluation of Chest Pain: Clinical Implications From SCOT-HEART and PROMISE. *Journal of the American College of Cardiology*. 2016;67:843-52.
- 9. Williams MC, Moss A, Nicol E and Newby DE. Cardiac CT Improves Outcomes in Stable Coronary Heart Disease: Results of Recent Clinical Trials. *Curr Cardiovasc Imaging Rep.* 2017;10:14.
- 10. Ladapo JA, Hoffmann U, Lee KL, Coles A, Huang M, Mark DB, Dolor RJ, Pelberg RA, Budoff M, Sigurdsson G, Severance HW and Douglas PS. Changes in Medical Therapy and Lifestyle After Anatomical or Functional Testing for Coronary Artery Disease. *Journal of the American Heart Association*. 2016;5.


CP-907-001-A Jun-29, 2018

- 11. Schulman-Marcus J, Lin FY, Gransar H, Berman D, Callister T, DeLago A, Hadamitzky M, Hausleiter J, Al-Mallah M, Budoff M, Kaufmann P, Achenbach S, Raff G, Chinnaiyan K, Cademartiri F, Maffei E, Villines T, Kim Y-J, Leipsic J, Feuchtner G, Rubinshtein R, Pontone G, Andreini D, Marques H, Chang H-J, Chow BJW, Cury RC, Dunning A, Shaw L and Min JK. Coronary revascularization vs. medical therapy following coronary-computed tomographic angiography in patients with low-, intermediate- and high-risk coronary artery disease: results from the CONFIRM long-term registry. *European heart journal cardiovascular Imaging*. 2017;18:841-848.
- 12. Chow BJ, Small G, Yam Y, Chen L, McPherson R, Achenbach S, Al-Mallah M, Berman DS, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Cheng VY, Chinnaiyan K, Cury R, Delago A, Dunning A, Feuchtner G, Hadamitzky M, Hausleiter J, Karlsberg RP, Kaufmann PA, Kim YJ, Leipsic J, LaBounty T, Lin F, Maffei E, Raff GL, Shaw LJ, Villines TC and Min JK. Prognostic and therapeutic implications of statin and aspirin therapy in individuals with nonobstructive coronary artery disease: results from the CONFIRM (COronary CT Angiography Evaluation For Clinical Outcomes: An InteRnational Multicenter registry) registry. Arteriosclerosis, thrombosis, and vascular biology. 2015;35:981-9.
- 13. Schulman-Marcus J, Hartaigh BO, Giambrone AE, Gransar H, Valenti V, Berman DS, Budoff MJ, Achenbach S, Al-Mallah M, Andreini D, Cademartiri F, Callister TQ, Chang HJ, Chinnaiyan K, Chow BJ, Cury R, Delago A, Hadamitzky M, Hausleiter J, Feuchtner G, Kim YJ, Kaufmann PA, Leipsic J, Lin FY, Maffei E, Pontone G, Raff G, Shaw LJ, Villines TC, Dunning A and Min JK. Effects of cardiac medications for patients with obstructive coronary artery disease by coronary computed tomographic angiography: results from the multicenter CONFIRM registry. *Atherosclerosis*. 2015;238:119-25.
- 14. Hoffmann U, Ferencik M, Udelson JE, Picard MH, Truong QA, Patel MR, Huang M, Pencina M, Mark DB, Heitner JF, Fordyce CB, Pellikka PA, Tardif JC, Budoff M, Nahhas G, Chow B, Kosinski AS, Lee KL and Douglas PS. Prognostic Value of Noninvasive Cardiovascular Testing in Patients With Stable Chest Pain: Insights From the PROMISE Trial (Prospective Multicenter Imaging Study for Evaluation of Chest Pain). Circulation. 2017;135:2320-2332.
- 15. Ferencik M, Mayrhofer T, Bittner DO, Emami H, Puchner SB, Lu MT, Meyersohn NM, Ivanov AV, Adami EC, Patel MR, Mark DB, Udelson JE, Lee KL, Douglas PS and Hoffmann U. Use of High-Risk Coronary Atherosclerotic Plaque Detection for Risk Stratification of Patients With Stable Chest Pain: A Secondary Analysis of the PROMISE Randomized Clinical Trial. *JAMA Cardiol.* 2018;3:144-152.
- 16. Shaw LJ, Hausleiter J, Achenbach S, Al-Mallah M, Berman DS, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Kim YJ, Cheng VY, Chow BJ, Cury RC, Delago AJ, Dunning AL, Feuchtner GM, Hadamitzky M, Karlsberg RP, Kaufmann PA, Leipsic J, Lin FY, Chinnaiyan KM, Maffei E, Raff GL, Villines TC, Labounty T, Gomez MJ and Min JK. Coronary computed tomographic angiography as a gatekeeper to invasive diagnostic and surgical procedures: results from the multicenter CONFIRM (Coronary CT Angiography Evaluation for Clinical Outcomes: an International Multicenter) registry. Journal of the American College of Cardiology. 2012;60:2103-14.
- 17. Foy AJ, Dhruva SS, Peterson B, Mandrola JM, Morgan DJ and Redberg RF. Coronary Computed Tomography Angiography vs Functional Stress Testing for Patients With Suspected Coronary Artery Disease: A Systematic Review and Meta-analysis. *JAMA internal medicine*. 2017;177:1623-1631.


CP-907-001-A Jun-29, 2018

- 18. Norgaard BL, Leipsic J, Gaur S, Seneviratne S, Ko BS, Ito H, Jensen JM, Mauri L, De Bruyne B, Bezerra H, Osawa K, Marwan M, Naber C, Erglis A, Park SJ, Christiansen EH, Kaltoft A, Lassen JF, Botker HE and Achenbach S. Diagnostic performance of noninvasive fractional flow reserve derived from coronary computed tomography angiography in suspected coronary artery disease: the NXT trial (Analysis of Coronary Blood Flow Using CT Angiography: Next Steps). *Journal of the American College of Cardiology*. 2014;63:1145-1155.
- 19. Koo BK, Erglis A, Doh JH, Daniels DV, Jegere S, Kim HS, Dunning A, DeFrance T, Lansky A, Leipsic J and Min JK. Diagnosis of ischemia-causing coronary stenoses by noninvasive fractional flow reserve computed from coronary computed tomographic angiograms. Results from the prospective multicenter DISCOVER-FLOW (Diagnosis of Ischemia-Causing Stenoses Obtained Via Noninvasive Fractional Flow Reserve) study. *Journal of the American College of Cardiology*. 2011;58:1989-97.
- 20. Min JK, Leipsic J, Pencina MJ, Berman DS, Koo BK, van Mieghem C, Erglis A, Lin FY, Dunning AM, Apruzzese P, Budoff MJ, Cole JH, Jaffer FA, Leon MB, Malpeso J, Mancini GB, Park SJ, Schwartz RS, Shaw LJ and Mauri L. Diagnostic accuracy of fractional flow reserve from anatomic CT angiography. *JAMA*: the journal of the American Medical Association. 2012;308:1237-45.
- 21. Min JK, Taylor CA, Achenbach S, Koo BK, Leipsic J, Norgaard BL, Pijls NJ and De Bruyne B. Noninvasive Fractional Flow Reserve Derived From Coronary CT Angiography: Clinical Data and Scientific Principles. *JACC Cardiovascular imaging*. 2015;8:1209-22.
- 22. Taylor CA, Fonte TA and Min JK. Computational fluid dynamics applied to cardiac computed tomography for noninvasive quantification of fractional flow reserve: scientific basis. *Journal of the American College of Cardiology*. 2013;61:2233-41.
- 23. Lu MT, Ferencik M, Roberts RS, Lee KL, Ivanov A, Adami E, Mark DB, Jaffer FA, Leipsic JA, Douglas PS and Hoffmann U. Noninvasive FFR Derived From Coronary CT Angiography: Management and Outcomes in the PROMISE Trial. *JACC Cardiovascular imaging*. 2017;10:1350-1358.
- 24. De Bruyne B, Fearon WF, Pijls NH, Barbato E, Tonino P, Piroth Z, Jagic N, Mobius-Winckler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd K, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Limacher A, Nuesch E and Juni P. Fractional flow reserve-guided PCI for stable coronary artery disease. *N Engl J Med*. 2014;371:1208-17.
- 25. De Bruyne B, Pijls NH, Kalesan B, Barbato E, Tonino PA, Piroth Z, Jagic N, Mobius-Winkler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd KG, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Juni P and Fearon WF. Fractional flow reserve-guided PCI versus medical therapy in stable coronary disease. *N Engl J Med*. 2012;367:991-1001.
- 26. National Clinical Guideline Centre for A and Chronic C. Chest Pain of Recent Onset: Assessment and Diagnosis of Recent Onset Chest Pain or Discomfort of Suspected Cardiac Origin: NICE (National Institute for Health and Care Excellence); 2010.


CP-907-001-A Jun-29, 2018

- 27. Moss AJ, Williams MC, Newby DE and Nicol ED. The Updated NICE Guidelines: Cardiac CT as the First-Line Test for Coronary Artery Disease. *Curr Cardiovasc Imaging Rep.* 2017;10:15.
- 28. Services DoHaH. Medicare program: Hospital Outpatient Prospective Payment and Ambulatory Surgical Center Payment Systems and Quality Reporting Programs. *42 CFR Parts 414, 416 and 419*. December 14, 2017;82:282.
- 29. Boden WE, O'Rourke RA, Teo KK, Hartigan PM, Maron DJ, Kostuk WJ, Knudtson M, Dada M, Casperson P, Harris CL, Chaitman BR, Shaw L, Gosselin G, Nawaz S, Title LM, Gau G, Blaustein AS, Booth DC, Bates ER, Spertus JA, Berman DS, Mancini GB and Weintraub WS. Optimal medical therapy with or without PCI for stable coronary disease. *N Engl J Med*. 2007;356:1503-16.
- 30. Al-Lamee R, Thompson D, Dehbi HM, Sen S, Tang K, Davies J, Keeble T, Mielewczik M, Kaprielian R, Malik IS, Nijjer SS, Petraco R, Cook C, Ahmad Y, Howard J, Baker C, Sharp A, Gerber R, Talwar S, Assomull R, Mayet J, Wensel R, Collier D, Shun-Shin M, Thom SA, Davies JE and Francis DP. Percutaneous coronary intervention in stable angina (ORBITA): a double-blind, randomised controlled trial. *Lancet (London, England)*. 2018;391:31-40.
- 31. Genders TS, Steyerberg EW, Alkadhi H, Leschka S, Desbiolles L, Nieman K, Galema TW, Meijboom WB, Mollet NR, de Feyter PJ, Cademartiri F, Maffei E, Dewey M, Zimmermann E, Laule M, Pugliese F, Barbagallo R, Sinitsyn V, Bogaert J, Goetschalckx K, Schoepf UJ, Rowe GW, Schuijf JD, Bax JJ, de Graaf FR, Knuuti J, Kajander S, van Mieghem CA, Meijs MF, Cramer MJ, Gopalan D, Feuchtner G, Friedrich G, Krestin GP and Hunink MG. A clinical prediction rule for the diagnosis of coronary artery disease: validation, updating, and extension. Eur Heart J. 2011;32:1316-30.
- 32. Hadamitzky M, Achenbach S, Al-Mallah M, Berman D, Budoff M, Cademartiri F, Callister T, Chang HJ, Cheng V, Chinnaiyan K, Chow BJ, Cury R, Delago A, Dunning A, Feuchtner G, Gomez M, Kaufmann P, Kim YJ, Leipsic J, Lin FY, Maffei E, Min JK, Raff G, Shaw LJ, Villines TC and Hausleiter J. Optimized prognostic score for coronary computed tomographic angiography: results from the CONFIRM registry (COronary CT Angiography Evaluation For Clinical Outcomes: An InteRnational Multicenter Registry). *Journal of the American College of Cardiology*. 2013;62:468-76.
- 33. Adamson PD, Fordyce CB, McAllister DA, Udelson JE, Douglas PS and Newby DE. Identification of patients with stable chest pain deriving minimal value from coronary computed tomography angiography: An external validation of the PROMISE minimal-risk tool. *International journal of cardiology*. 2018;252:31-34.
- 34. Fordyce CB, Douglas PS, Roberts RS, Hoffmann U, Al-Khalidi HR, Patel MR, Granger CB, Kostis J, Mark DB, Lee KL and Udelson JE. Identification of Patients With Stable Chest Pain Deriving Minimal Value From Noninvasive Testing: The PROMISE Minimal-Risk Tool, A Secondary Analysis of a Randomized Clinical Trial. *JAMA Cardiol*. 2017;2:400-408.
- 35. Douglas PS, Pontone G, Hlatky MA, Patel MR, Norgaard BL, Byrne RA, Curzen N, Purcell I, Gutberlet M, Rioufol G, Hink U, Schuchlenz HW, Feuchtner G, Gilard M, Andreini D, Jensen JM, Hadamitzky M, Chiswell K, Cyr D, Wilk A, Wang F, Rogers C and De Bruyne B. Clinical outcomes of fractional flow reserve by computed tomographic angiography-guided diagnostic strategies vs. usual care in patients with suspected coronary artery disease: the


CP-907-001-A Jun-29, 2018

- prospective longitudinal trial of FFR(CT): outcome and resource impacts study. *Eur Heart J.* 2015;36:3359-67.
- 36. Fordyce CB and Douglas PS. Outcomes-Based CV Imaging Research Endpoints and Trial Design: From Pixels to Patient Satisfaction. *JACC Cardiovascular imaging*. 2017;10:253-263.
- 37. Fihn SD, Gardin JM, Abrams J, Berra K, Blankenship JC, Dallas AP, Douglas PS, Foody JM, Gerber TC, Hinderliter AL, King SB, 3rd, Kligfield PD, Krumholz HM, Kwong RY, Lim MJ, Linderbaum JA, Mack MJ, Munger MA, Prager RL, Sabik JF, Shaw LJ, Sikkema JD, Smith CR. Smith SC. Spertus JA and Williams Jr., Jr., ACCF/AHA/ACP/AATS/PCNA/SCAI/STS Guideline for the diagnosis and management of patients with stable ischemic heart disease: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines, and the American College of Physicians, American Association for Thoracic Surgery, Preventive Cardiovascular Nurses Association, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. Journal of the American College of Cardiology. 2012;60:e44-e164.
- 38. Bradley SM, Spertus JA, Kennedy KF, Nallamothu BK, Chan PS, Patel MR, Bryson CL, Malenka DJ and Rumsfeld JS. Patient selection for diagnostic coronary angiography and hospital-level percutaneous coronary intervention appropriateness: insights from the National Cardiovascular Data Registry. *JAMA internal medicine*. 2014;174:1630-9.
- 39. Lin GA, Dudley RA, Lucas FL, Malenka DJ, Vittinghoff E and Redberg RF. Frequency of stress testing to document ischemia prior to elective percutaneous coronary intervention. *JAMA : the journal of the American Medical Association*. 2008;300:1765-73.
- 40. Patel MR, Dai D, Hernandez AF, Douglas PS, Messenger J, Garratt KN, Maddox TM, Peterson ED and Roe MT. Prevalence and predictors of nonobstructive coronary artery disease identified with coronary angiography in contemporary clinical practice. *American heart journal*. 2014;167:846-52.e2.
- 41. Colleran R, Douglas PS, Hadamitzky M, Gutberlet M, Lehmkuhl L, Foldyna B, Woinke M, Hink U, Nadjiri J, Wilk A, Wang F, Pontone G, Hlatky MA, Rogers C and Byrne RA. An FFRCT diagnostic strategy versus usual care in patients with suspected coronary artery disease planned for invasive coronary angiography at German sites: one-year results of a subgroup analysis of the PLATFORM (Prospective Longitudinal Trial of FFRCT: Outcome and Resource Impacts) study. *Open heart*. 2017;4:e000526.
- 42. Gibbons RJ, Balady GJ, Bricker JT, Chaitman BR, Fletcher GF, Froelicher VF, Mark DB, McCallister BD, Mooss AN, O'Reilly MG, Winters WL, Gibbons RJ, Antman EM, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Hiratzka LF, Jacobs AK, Russell RO and Smith SC. ACC/AHA 2002 guideline update for exercise testing: summary article. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Update the 1997 Exercise Testing Guidelines). *Journal of the American College of Cardiology*. 2002;40:1531-40.
- 43. Pellikka PA, Nagueh SF, Elhendy AA, Kuehl CA and Sawada SG. American Society of Echocardiography Recommendations for Performance, Interpretation, and Application of


CP-907-001-A Jun-29, 2018

- Stress Echocardiography. *Journal of the American Society of Echocardiography*. 2007;20:1021-1041.
- 44. Tilkemeier PL, Bourque J, Doukky R, Sanghani R and Weinberg RL. ASNC imaging guidelines for nuclear cardiology procedures. *Journal of Nuclear Cardiology*. 2017;24:2064-2128.
- 45. Henzlova MJ, Duvall WL, Einstein AJ, Travin MI and Verberne HJ. ASNC imaging guidelines for SPECT nuclear cardiology procedures: Stress, protocols, and tracers. *Journal of nuclear cardiology : official publication of the American Society of Nuclear Cardiology*. 2016;23:606-39
- 46. Henzlova MJ, Duvall WL, Einstein AJ, Travin MI and Verberne HJ. Erratum to: ASNC imaging guidelines for SPECT nuclear cardiology procedures: Stress, protocols, and tracers. *Journal of nuclear cardiology: official publication of the American Society of Nuclear Cardiology*. 2016;23:640-642.
- 47. Dilsizian V, Bacharach SL, Beanlands RS, Bergmann SR, Delbeke D, Dorbala S, Gropler RJ, Knuuti J, Schelbert HR and Travin MI. ASNC imaging guidelines/SNMMI procedure standard for positron emission tomography (PET) nuclear cardiology procedures. *Journal of nuclear cardiology:* official publication of the American Society of Nuclear Cardiology. 2016;23:1187-1226.
- 48. Hundley WG, Bluemke DA, Finn JP, Flamm SD, Fogel MA, Friedrich MG, Ho VB, Jerosch-Herold M, Kramer CM, Manning WJ, Patel M, Pohost GM, Stillman AE, White RD and Woodard PK. ACCF/ACR/AHA/NASCI/SCMR 2010 expert consensus document on cardiovascular magnetic resonance: a report of the American College of Cardiology Foundation Task Force on Expert Consensus Documents. *Circulation*. 2010;121:2462-508.
- 49. Leipsic J, Abbara S, Achenbach S, Cury R, Earls JP, Mancini GJ, Nieman K, Pontone G and Raff GL. SCCT guidelines for the interpretation and reporting of coronary CT angiography: a report of the Society of Cardiovascular Computed Tomography Guidelines Committee. *Journal of cardiovascular computed tomography*. 2014;8:342-58.
- 50. Abbara S, Blanke P, Maroules CD, Cheezum M, Choi AD, Han BK, Marwan M, Naoum C, Norgaard BL, Rubinshtein R, Schoenhagen P, Villines T and Leipsic J. SCCT guidelines for the performance and acquisition of coronary computed tomographic angiography: A report of the society of Cardiovascular Computed Tomography Guidelines Committee: Endorsed by the North American Society for Cardiovascular Imaging (NASCI). *Journal of cardiovascular computed tomography*. 2016;10:435-449.
- 51. Hicks KA, Mahaffey KW, Mehran R, Nissen SE, Wiviott SD, Dunn B, Solomon SD, Marler JR, Teerlink JR, Farb A, Morrow DA, Targum SL, Sila CA, Thanh Hai MT, Jaff MR, Joffe HV, Cutlip DE, Desai AS, Lewis EF, Gibson CM, Landray MJ, Lincoff AM, White CJ, Brooks SS, Rosenfield K, Domanski MJ, Lansky AJ, McMurray JJV, Tcheng JE, Steinhubl SR, Burton P, Mauri L, O'Connor CM, Pfeffer MA, Hung HMJ, Stockbridge NL, Chaitman BR and Temple RJ. 2017 Cardiovascular and Stroke Endpoint Definitions for Clinical Trials. *Journal of the American College of Cardiology*. 2018;71:1021-1034.
- 52. Collet D. Modeling survival data in medical research (2nd edition). London: Chapman & Hall; 2003.


- 53. Kalbfleisch JD, Prentice RL. The Statistical Analysis of Failure Time Data. 2nd edition. 2002, John Wiley & Sons, Inc. Hoboken, New Jersey.
- 54. Cox DR. Regression Models and Life-Tables. *Journal of the Royal Statistical Society Series B (Methodological)*. 1972;34:187-220.
- 55. Kaplan EL and Meier P. Nonparametric Estimation from Incomplete Observations. *Journal of the American Statistical Association*. 1958;53:457-481.
- 56. Pocock SJ, Ariti CA, Collier TJ and Wang D. The win ratio: a new approach to the analysis of composite endpoints in clinical trials based on clinical priorities. *Eur Heart J.* 2012;33:176-82.
- 57. Finkelstein DM and Schoenfeld, DA. Combining mortality and longitudinal measures in clinical trials. *Statistics in Medicine*. 1999;18:1341-1354.
- 58. Fine JP and Gray RJ. A Proportional Hazards Model for the Subdistribution of a Competing Risk. *Journal of the American Statistical Association*. 1999;94:496-509.


#### The **PRECISE** Protocol

# <u>Prospective Randomized Trial of the Optimal Evaluation of Cardiac Symptoms and Revascularization</u>

#### **Study Objective**

The primary objective of the PRECISE trial is to assess clinical outcomes, decision making regarding noninvasive testing and invasive angiography, and costs using a precision evaluation strategy as compared to a usual care strategy in participants with stable symptoms suggestive of significant coronary artery disease. The precision evaluation strategy will be based on a pre-test risk assessment and will incorporate cCTA with selective FFR<sub>CT</sub> and guideline-recommended care with symptom and risk factor management and no immediately planned testing.

#### Study Design

The study will be a prospective, pragmatic, randomized clinical trial of the comparative effectiveness of diagnostic evaluation strategies for stable suspected CAD, to be performed in outpatient settings, including primary care and cardiology practices. Qualifying patients presenting with new symptoms suspicious for clinically significant CAD (and without known CAD), who are recommended for diagnostic testing and did not receive any cardiovascular testing within the past 12 months, will be randomized to an initial strategy of either precision care or usual care. All subsequent decisions in the usual care arm regarding additional testing, medications, and/or procedures will be at the discretion of the responsible clinical care team.

## Study Principal Investigator

Pamela S. Douglas, MD Duke University Durham, NC 27701 USA

#### **Sponsor**

HeartFlow, Inc. 1400 Seaport Blvd., Building B Redwood City, CA 94063 Campbell Rogers, MD Chief Medical Officer Version Date: Oct 15, 2019

#### **Investigator Protocol Signature Page**

I have read and understand the protocol and agree that it contains all the ethical, legal, and scientific information necessary to conduct this study. I will personally conduct the study as described. I will provide copies of the protocol to all assigned physicians, nurses, and other professional personnel who will participate in the study and will be responsible for their compliance and adherence to the study protocol. I am aware that this protocol must be approved by the Institutional Review Board or Ethics Committee. I agree to adhere strictly to the attached protocol. I agree that clinical data entered on case report forms by me and my staff will be supplied to HeartFlow and may be utilized by HeartFlow in various ways, such as for submission to governmental regulatory authorities and/or in combination with clinical data gathered from other research sites, whenever applicable. I agree to allow HeartFlow monitors and auditors and their designees full access to all medical records at the research facility for participants screened or randomized in the study. I agree to provide all participants with informed consent forms and will ensure adequate informed consent is obtained, as required by government regulations and International Conference on Harmonization guidelines.

| · | |
|---|---|
| Site Name | Site Number |
| Principal Investigator (print name) | |
| Principal Investigator (Signature) | Date |
| — DocuSigned by:<br>Manush Patch | 10/15/2019 |
| —a₃₄Fa8aA40884c4 Manesh Patel, MD, Trial Co-Principal Investigate | or Date |
| DocuSigned by: | 10/15/2019 |
| Campbell Rogers, MD, HeartFlow CMO | Date |

## **Protocol Version and Amendment Tracking**

| Version Number/Amendment | Approval Date |
|--------------------------|---------------|
| 1.0 | Jun 29, 2018 |
| 1.1 | Jul 31, 2018 |
| 1.2 | Sept 10, 2018 |
| 1.3 | Nov 21, 2018 |
| 1.4 | Feb 1, 2019 |
| 1.5 | Oct 15, 2019 |

## Amendment from version 1.4 dated February 1. 2019 to version 1.5 dated October 15. 2019

| Section | Version 1.4 | Version 1.5 |
|---|---|---|
| Investigator Protocol<br>Signature Page | NA | Included separate line for PI signature |
| Table of Abbreviations | NA | AG: Agatston units |
| Table of Abbreviations | DECISION: <u>Decisive Evaluation of</u> <u>Cardiac Ischemia</u> , <u>Symptoms and</u> <u>Revascularization</u> | Removed |
| Table of Abbreviations | HU: Hounsfield units | Removed |
| IV. Study Overview and<br>Objectives - Study<br>duration | The anticipated total duration of the PRECISE study will be approximately 48 months for start-up, enrollment, follow up, and close out. Participants will be followed for 24 months after enrollment. | Overall study duration reduced to 36 month and patient follow up to 12 month after enrollment. "The anticipated total duration of the PRECISE study will be approximately 36 months for start-up, enrollment, follow up, and close out. Participants will be followed for 12 months after enrollment." |
| IV.A. Overview of PRECISE – figure of the trial design | Precision evaluation Strategy assigned by PROMISE risk strata Guideline rec medical management wo planned testing CCTA +/- FFRct | Figure updated to remove 24 month and co-primary endpoints of DECISION. Arrows leading to GRMT or cCTA annotated "low risk" and "elevated risk" respectively. Patients with known nonobstructive coronary plaque or extensive coronary calcium randomized to the precision arm are mandated to undergo cCTA +/- FFR <sub>CT</sub> , independent from PROMISE risk score strata. |
| IV.B. Primary Objective and Endpoints | Per the exclusion criteria, any previous noninvasive or invasive CV diagnostic testing for suspected CAD must have been >1 year prior to enrollment. Patients with known obstructive CAD (prior myocardial infarction, CABG or PCI, any stenosis ≥50%) are ineligible for PRECISE. | Replaced with: "Patients with known nonobstructive coronary plaque or extensive coronary calcium randomized to the precision arm are mandated to undergo cCTA +/- FFR <sub>CT</sub> , independent from their PROMISE risk score strata." |
| IV.C. Secondary<br>Endpoints | Endpoints will be assessed at 45 days, 6 months, 1 year and 2 years. | Removed secondary endpoint assessment at 2 years: "Endpoints will be assessed at 45 days, 6 months and 1 year." |
| IV.C. Secondary<br>Endpoints | 9. PRECISE primary endpoint at 24 month | Removed PRECISE primary endpoint at 24 month |

|---|---|---|
| IV.C. Secondary<br>Endpoints | 10. MACE, defined as all-cause death myocardial infarction, or ischemia-driven revascularization at 24 months (DECISION co-primary end point) | Removed DECISION co-primary endpoint |
| IV.C. Secondary<br>Endpoints | 11. All-cause death, MI, all follow-up unplanned revascularization procedures, invasive coronary angiograms without actionable findings at 24 months (DECISION co-primary end point) | Removed DECISION co-primary endpoint |
| V.A. Patient Screening<br>for Eligibility – Inclusion<br>Criteria | NA | "3. If prior CV testing has occurred, it must have been performed greater than one year prior to randomization, and the following must be met: a) cCTA or invasive coronary angiography (ICA) with stenosis < 50% b) Quantified coronary artery calcium (CAC) < 100 AG |
| V.A. Patient Screening<br>for Eligibility –<br>Exclusion Criteria | 3. Noninvasive or invasive CV testing within 1 year (for suspected CAD). CV testing for CAD refers to any stress tests, ICA, and cCTA (including calcium scoring) only. Resting ECG and resting echocardiogram are not exclusionary. | Including resting CMR (MRI) as not exclusionary: "3. Noninvasive or invasive CV testing for CAD within 1 year. CV testing for CAD refers to any stress tests, invasive coronary angiography (ICA), and cCTA (including calcium scoring) only. a) Resting ECG, resting echocardiogram and resting CMR (MRI) are not exclusionary regardless of when they were performed. |

|---|---|---|
| V.D. Participant Follow-<br>Up | 24 months (+/-30 days) follow-up contact At the 24-month follow-up visit, participants will be asked to report the following: Assessment if any MACE has occurred since the last visit/phone call | Removed participant follow-up requirement at 24 month |
| | CV Update: Review and documentation of<br>any cardiovascular diagnostic test,<br>cardiovascular procedure, or<br>hospitalizations/clinic visits due to<br>cardiovascularsymptoms and complications<br>since last visit | |
| | Review and documentation of concomitant<br>cardiovascular medication changes since<br>enrollment | |
| | <ul><li>Complete the following 2 questionnaires:</li><li>Seattle Angina Questionnaire</li></ul> | |
| | ○ EQ-5D-5L Questionnaire | |
| | Collection of the following: | |
| | ○ Any cardiovascular test – both written | |
| | report and test output | |
| | <ul> <li>Any cardiovascular imaging – both written<br/>report and image file</li> </ul> | |
| VII.A. Primary Endpoint | The exception will be for peri procedural | Reference 60 (Moussa ID, Klein LW, et al) |
| Definitions – | myocardial infarctions, which are defined | removed and updated with reference 51 |
| Myocardial infarction | as biomarker elevation ≥10 times the | (Thygesen K, Alpert JS, et al) |
| | upper reference limit (URL) for creatine kinase MB (CKMB) and/or ≥70 URL for troponin as outlined in the most recent SCAI definition <sup>60</sup> . | "This definition will be followed for spontaneous as well as periprocedural MIs, for which the elevation in cTn must be at least cTn values >5 times the 99th percentile URL for PCI and >10 times for CABG related infarctions <sup>51</sup> " |
| VIII.B. Statistical Analysis Plan – Analysis of the Primary Endpoint | A sensitivity analysis for the primary composite MACE endpoint will be conducted using the method of "winratio" <sup>56</sup> . The win-ratio method of Pocock et al is an extension of Finkelstein and Schoenfeld rank-test method <sup>57</sup> which order-rank composite endpoints based on their clinical importance. | A sensitivity analysis for the primary composite MACE (all cause death and non-fatal MI) or invasive cardiac catheterization without CAD (no coronary stenosis ≥50% according to QCA by core-lab adjudication or site interpretation if QCA is not available, or with FFR≤0.80, or instantaneous wave free ratio (iFR) ≤0.89) endpoint will be conducted using the method of "win-ratio" and Finkelstein and Schoenfeld rank-test method <sup>57</sup> . |

## **TABLE OF CONTENTS**

| I. STUDY SYNOPSIS | 12 |
|---|---|
| II. INTRODUCTION | 16 |
| II.A. Primary Hypothesis | |
| II.B. Significance of the Study | |
| III. BACKGROUND AND STUDY RATIONALE | 17 |
| III.A. Prior Literature and Studies | |
| III.B. Rationale for the Current Study: A Precision Approach to Chest Pain Evaluation | |
| IV. STUDY OVERVIEW AND OBJECTIVES | 22 |
| IV.A. Overview of PRECISE | |
| IV.B. Primary Objective and Endpoints | |
| IV.C. Secondary Endpoints | |
| IV.D. Rationale for the Selection of Outcome Measures | |
| IV.E. Rationale for the Selection of Testing in Each Arm | |
| IV.F. Participant Randomization | |
| IV.G. Diagnostic Evaluations and Subsequent Care | |
| V. STUDY PROCEDURES | 30 |
| V.A. Participant Screening for Eligibility | |
| V.B. Participant Randomization and Enrollment | |
| V.C. Participant Cohort Assignment | |
| V.D. Participant Follow-Up | |
| V.E. Testing in precision evaluation arm for participants assigned to no immediate testing | |
| V.F. Participant Withdrawal | |
| V.G. Schedule of Assessments | |
| VI. ADDITIONAL ASSESMENTS AND SUBSTUDIES | 36 |
| VI.A. Quality of Life Assessments | |
| VI.B. Economic and Resource Utilization Assessments | |
| VI.C. Imaging and other Cardiac Assessments | |
| VII. ENDPOINT DETERMINATION, SAFETY AND MONITORING | 37 |
| VII.A. Primary Endpoint Definitions | |
| VII.B. Secondary Endpoint Definitions | |
| VII.C. Testing Complications and Reporting | |
| VII.D. Independent Clinical Event Adjudication Committee | |

| VII.E. Data and Safety Monitoring Board | |
|---------------------------------------------------------|----|
| VIII. STATISTICAL METHODS | 41 |
| VIII.A. Sample Size Determination and Statistical Power | |
| VIII.B. Statistical Analysis Plan | |
| IX. ETHICAL CONSIDERATIONS AND RISK ANALYSIS | 46 |
| IX.A. Ethical Considerations | |
| IX.B. Study Risks and Benefits | |
| X. DATA HANDLING AND QUALITY ASSURANCE | 47 |
| X.A. Completing and Signing Case Report Forms | |
| X.B. Clinical Data Management | |
| X.C. Archiving of Data | |
| XI. STUDY MONITORING, AUDITING, AND INSPECTING | 48 |
| XI.A. Study Monitoring | |
| XI.B. Auditing and Inspecting | |
| XII. REFERENCES | 49 |

## **TABLE OF ABBREVIATIONS**

| ACC | American College of Cardiology |
|---|---|
| ACS | acute coronary syndrome |
| АНА | American Heart Association |
| AG | Agatston units |
| ВМІ | body mass index |
| BP | blood pressure |
| CAC | Coronary Artery Calcium |
| CAD | coronary artery disease |
| CV | Cardiovascular |
| CI | confidence interval |
| CK-MB | creatine kinase-myocardial band |
| CMS | Centers for Medicare & Medicaid Services |
| COCATS | Core Cardiology Training Symposium |
| cCTA | coronary computed tomographic angiography |
| СР | chest pain |
| cTn | cardiac troponin |
| DCRI | Duke Clinical Research Institute |
| DSMB | Data and Safety Monitoring Board |
| ECG | Electrocardiogram |
| Echo | Echocardiogram |
| EDC | electronic data capture |
| EQ-5D-5L | a standardized instrument developed by the <i>EuroQol</i> Group as a measure of health-related quality of life. |
| eCRF | electronic case report form |
| FFR | fractional flow reserve |
| FS | Finkelstein and Schoenfeld statistical method |
| FFR <sub>CT</sub> | non-invasive technique using cCTA to determine FFR |

| g/L | grams per liter |
|---|---|
| HDL | high-density lipoprotein |
| ICA | invasive coronary angiography |
| iFR | instantaneous wave free ratio |
| IRB | institutional review board |
| IVUS | intravascular ultrasound |
| IXRS | interactive voice/web response system |
| LDL | low-density lipoprotein |
| LV | left ventricular |
| MACE | major adverse cardiovascular event |
| MAR | missing at random |
| MDCT | multidetector computed tomography |
| MI | myocardial infarction |
| MOP | manual of procedures |
| MPI | myocardial perfusion imaging |
| mSv | milliSievert |
| NI | non-invasive |
| NICE | National Institute for Health and Care Excellence (In the United Kingdom's National Health Service) |
| NHPR | non-hyperemic pressure ratio |
| OCT | optical coherence tomography |
| PAD | peripheral arterial disease |
| PCI | percutaneous coronary intervention |
| PI | principal investigator |
| PLATFORM | Prospective LongitudinAl Trial of FFR <sub>CT</sub> : Outcome and Resource Impacts study |
| PRECISE | Prospective Randomized Trial of the Optimal Evaluation of Cardiac Symptoms and Revascularization |
| PROMISE | PROspective Multicenter Imaging Study for Evaluation of Chest Pain randomized clinical trial |

| QCA | quantitative coronary angiography |
|---|---|
| QoL | quality of life |
| ROC | receiver operating characteristic |
| SAQ | Seattle Angina Questionnaire |
| SCAI | Society for Cardiovascular Angiography and Interventions |
| SCOT-<br>HEART | Scottish Computed Tomography of the HEART randomized clinical trial |
| ULN | upper limit of normal |
| URL | upper reference limit |

## **I.STUDY SYNOPSIS**

| Protocol Title | PRECISE: Prospective Randomized Trial of the Optimal Evaluation of Cardiac Symptoms and Revascularization |
|---|---|
| Investigational Strategy | Precision diagnostic evaluation as the initial strategy for suspected significant CAD in patients with stable symptoms |
| Study Principal | Pamela S Douglas, MD |
| Investigator | Duke Clinical Research Institute, Duke University, Durham NC |
| Academic Research | Duke Clinical Research Institute (DCRI), Durham, NC, USA |
| Organizations | Cardiovascular Research Foundation (CRF), New York, NY, USA |
| Clinical Research<br>Organization | Medpace Research, Inc. |
| Sponsor | HeartFlow, Inc.<br>1400 Seaport Blvd<br>Redwood City, CA 94063 |
| Participants and Study<br>Centers | Approximately 2100 participants randomized at approximately 100 sites in the US and outside of the US |
| Planned Study Duration | Approximately 36 months |
| Primary Study Objective | To assess clinical outcomes, decision making regarding noninvasive testing and invasive angiography, and costs using a precision evaluation strategy as compared to a usual care strategy in participants with stable symptoms suggestive of significant coronary artery disease. The precision evaluation strategy will be based on a pre-test risk assessment and will incorporate cCTA with selective FFR <sub>CT</sub> and guideline-recommended care with symptom and risk factor management and no additional immediately planned testing. |
| Primary Hypotheses | In stable participants with a clinical recommendation for testing to evaluate suspected significant CAD a precision evaluation strategy, incorporating a risk-based assignment to guideline recommended medical management without planned testing for selected low risk participants or cCTA with selective FFR <sub>CT</sub> in elevated risk participants, will result in improved clinical outcomes of death/MI and a lower rate of catheterization without obstructive CAD as compared to usual care strategy. |
| Population | Stable patients who have a clinical recommendation for testing (noninvasive or invasive) for suspected significant CAD |
| Study Design and Methods | Prospective, pragmatic, randomized clinical trial of diagnostic evaluation strategies for stable suspected significant CAD, to be performed in outpatient settings, including primary care and cardiology practices. Qualifying patients presenting with new symptoms suspicious for clinically significant CAD (and without known obstructive CAD), who are recommended for diagnostic testing and did not receive any cardiovascular testing within the past 12 months, will be randomized to an initial strategy of either precision care or usual care of the site's choosing. All subsequent decisions in the usual care arm regarding additional testing, medications, and/or procedures will be at the discretion of the responsible clinical care team; the use of cCTA as the |

initial diagnostic strategy is not allowed in the usual care arm and is prohibited as a subsequent test for the first 45 days after randomization. **Precision evaluation:** Participants randomized to a precision strategy will then be assigned to either guideline-recommended care without immediately planned testing (low risk) or cCTA with selective FFR<sub>CT</sub> (for those with elevated risk or known non-obstructive atherosclerosis) using a risk tool based on pre-test clinical characteristics derived from the PROMISE trial and validated in SCOT-HEART trial. As is recommended for all participants, those assigned to guidelinerecommended care without planned testing will be treated with preventive and antianginal medical treatment per guideline recommendations and clinical judgment and followed without testing. Participants and their providers will be provided informational resources explaining the safety and rationale of this strategy based on pre-test probabilities and the PROMISE Minimal Risk Score. Participants with documented intractable symptoms despite maximal medical management may undergo cCTA with selective FFR<sub>CT</sub> at the participant's or site clinician's discretion. **Usual Care:** For participants randomized to usual care, the participant's care team will select the specific noninvasive stress test (exercise electrocardiogram, stress nuclear imaging [including PET], stress MR, or stress echocardiogram); OR invasive test: (direct to diagnostic catheterization). The use of cCTA as the initial diagnostic strategy is explicitly excluded in this arm and prohibited as a subsequent test for the first 45 days after randomization. In both arms, the participant's care team will be provided with physician and patient informational resources summarizing current recommendations for test interpretation and preventive care. Optimal medical management will be recommended but not mandated in either arm. Randomization Participants will be randomized using a 1:1 randomization scheme via an interactive web or voice-based system (IXRS). Randomization will and Stratification be stratified by intended first test if randomized to usual care, low vs. elevated pre-test risk, and site. Enrollment in the strata of intended noninvasive test first (vs. intended invasive angiography first) will be capped at 90%. **Primary Endpoint** Time to a composite of: MACE (all cause death, non-fatal MI) or invasive cardiac catheterization without obstructive CAD (obstructive CAD defined as diameter stenosis ≥50% according to core-lab adjudicated quantitative coronary angiography (QCA), FFR≤0.80, or iFR≤0.89) at one year (intention to treat) Endpoints will be assessed at 45 days, 6 months, and 1 year. Secondary Effectiveness 1. Hierarchical analysis (Finkelstein and Schoenfeld (FS) and Pocock's win ratio) of primary endpoint **Endpoints** 2. Resource use patterns and medical costs 3. QoL: measured by the Seattle Angina Questionnaire (SAQ) to assess angina-specific Quality of Life and the EuroQoL 5D (EQ-5D-5L) survey to assess overall (generic) health status

| | 4. Death: All-cause, cardiovascular, non-cardiovascular |
|---|---|
| | 5. Myocardial infarction: All, procedural, spontaneous MI |
| | Hospitalizations: All, cardiovascular, non-cardiovascular, and for progressive or unstable angina |
| | 7. Preventive medication use (ASA, statins) in participants with clinical indication for use: e.g.: hyperlipidemia, diabetes, documented CAD |
| | 8. Cumulative radiation exposure at 1 year |
| | Proportion of invasive coronary angiogram patients who undergo revascularization (PCI or CABG) within 6 months of enrollment |
| Pre-specified subgroup | Low risk vs. elevated risk by PROMISE score or pre-existing non-<br>obstructive CAD |
| analyses | 2. Intended initial test: functional stress test vs. invasive (direct to cath) |
| | 3. Clinical factors: sex, age, diabetes |
| | Presentation: primary symptom (chest pain vs. other), SAQ angina frequency score |
| Inclusion Criteria | Inclusion criteria (all must be present): |
| | 1. Age ≥18 years |
| | <ul> <li>2. Stable typical or atypical symptoms suggesting possible significant coronary artery disease (CAD) with further non-emergent testing or elective catheterization recommended to evaluate the presence of suspected significant CAD. Stable chest pain (or equivalent) includes those who have fully been ruled out for Acute Coronary Syndrome (ACS) and for whom elective testing is recommended, regardless of the venue in which they are seen.</li> <li>3. If prior CV testing has occurred, it must have been performed greater than one year prior to randomization, and the following must be met: <ul> <li>a. cCTA or invasive coronary angiography (ICA) with stenosis &lt; 50%</li> <li>b. Quantified coronary artery calcium (CAC) &lt; 100 AG</li> </ul> </li> <li>4. Safe performance of cCTA: <ul> <li>a. Creatinine clearance ≥45 ml/min per most recent measurement within 90 days</li> <li>b. For a female participant of childbearing potential (those who have not been surgically sterilized or are not</li> </ul> </li> </ul> |
| | postmenopausal), a pregnancy test must be performed with negative results known within 7 days prior to randomization |
| | 5. Willingness to comply with all aspects of the protocol, including adherence to the assigned strategy and follow-up visits |
| | 6. Ability to provide written informed consent |
| Exclusion criteria | Exclusion criteria (all must be absent): 1. Acute chest pain (in patients who have not been ruled out for ACS) 2. Unstable clinical status |
| | 2. Onotable diffical status |

| | 3. Noninvasive or invasive CV testing for CAD within 1 year. CV testing for CAD refers to any stress tests, invasive coronary angiography (ICA) and cCTA (including calcium scoring) only. |
|---|---|
| | Resting ECG, resting echocardiogram and resting CMR (MRI) are not exclusionary regardless of when were performed |
| | 4. Lifetime history of known obstructive CAD (prior myocardial infarction, CABG or PCI, stenosis ≥50%), known EF ≤40% or other moderate to severe valvular or congenital cardiac disease |
| | 5. Contraindications to cCTA including but not limited to creatinine clearance (GFR) <45 ml/min as per most recent measurement taken within 90 days |
| | Exceeds the site's weight or size limit for cCTA or cardiac catheterization |
| | 7. Any condition leading to possible inability to comply with the protocol procedures or follow-up |
| | Any condition that might interfere with the study procedures or follow-up |
| | Enrolled in an investigational trial that involves a non-approved cardiac drug or device which has not reached its primary endpoint |
| | Life expectancy less than 2 years due to non-cardiovascular comorbidities |
| Study Follow-up | Participant follow-up will be done at 45 days, 6 months, and 1 year. |
| Sample Size<br>Considerations | Primary superiority testing hypothesis of all cause death/MI or invasive cardiac catheterization without obstructive CAD (diameter stenosis ≥50% or FFR≤0.80/ or iFR≤0.89) at one year (intention to treat, time to first event analysis): Assuming an 8% event rate at 1 year in the usual care group and 5% in the precision care group (3% absolute [37.5% relative] effect magnitude). Assumed rates are based on estimated ~20% assigned to guideline- recommended care with symptom management and no planned testing (within which 30% will cross over to cCTA with selective FFR <sub>CT</sub> ); and overall 10% will not receive assigned testing; enrolling 1050 participants per group (2100 total participants) would provide at least 90% power to demonstrate superiority accounting for 10% attrition rate. |

#### II. INTRODUCTION

#### **II.A.** Primary Hypotheses

The primary goal of the Prospective Randomized Trial of the Optimal Evaluation of Cardiac Symptoms and Revascularization (PRECISE) research program is to assess clinical outcomes, decision making regarding noninvasive testing and invasive angiography, and costs using a precision evaluation strategy as compared to a usual care strategy in participants with stable symptoms suggestive of significant coronary artery disease. The precision evaluation strategy will be based on a pre-test risk assessment and the presence or absence of known non-obstructive atherosclerosis; participants in this arm will undergo either cCTA with selective FFR<sub>CT</sub> or no immediately planned testing. All participants are encouraged to have guideline- recommended care with symptom management.

The primary hypothesis of PRECISE is: in stable participants with a clinical recommendation for testing to evaluate suspected significant coronary artery disease (CAD), a precision evaluation strategy will result in improved clinical outcomes of death/MI and a lower rate of catheterization without obstructive CAD as compared to a usual care strategy.

An important secondary hypothesis is that the precision evaluation strategy will result in improved patient-reported outcomes, reflected in the SAQ angina frequency and quality of life scores. We also expect the precision strategy to result in reduced resource utilization and net cost savings compared to usual care evaluation.

The usual care arm participants will undergo either noninvasive stress testing, with the specific modality at the discretion of the participant's clinician, or invasive coronary angiography (ICA) as the initial test.

The precision evaluation arm starts with the use of the PROMISE Risk Tool to categorize patient risk for CAD and events. The PROMISE Risk Tool is a validated risk model that has been shown to accurately identify chest pain patients who are unlikely to benefit from non-invasive testing (i.e. have minimal or no atherosclerosis and likely to have no events within two years). The lowest risk group in the precision arm identified using this model will be assigned to guideline-recommended care focused on symptom and risk factor management without planned cardiac diagnostic testing. Those participants who are identified to be of elevated risk or those with known non-obstructive coronary atherosclerosis (regardless of risk score results) will be initially evaluated with cCTA with selective FFR<sub>CT</sub>.

#### I.B. Significance of the Study

The goal of PRECISE is to define the optimal evaluation and management strategy of stable, symptomatic participants with suspected significant CAD. If the hypotheses of PRECISE are supported by the results of the trial, PRECISE will form the core of a compelling body of evidence supporting important changes in clinical practice guidelines and clinical care that will both improve outcomes for patients and reduce the use of unnecessary (low yield) testing and associated medical costs. Chest pain is one of the most common symptoms that bring patients into the health care system and one of the most difficult for providers to address confidently. The variability of current practice and the frequent overuse of testing derive from the lack of consensus among experts and among guidelines about how best to achieve a secure diagnosis and appropriate management plan. The results of PRECISE will have major implications for all health systems where stable chest pain is a common reason for participants to seek care.

#### III. BACKGROUND AND STUDY RATIONALE

#### **III.A.** Prior Literature and Studies

<u>Unmet need to develop novel approaches for the diagnostic evaluation in stable chest pain</u> patients

CAD is an extremely common diagnosis worldwide and results in significant morbidity and mortality <sup>1</sup>. Among the common presentations, stable symptoms of chest pain or exertional dyspnea can be diagnostically puzzling and often require diagnostic testing or angiography to be certain of the diagnosis and treatment. Current US, EU and UK guidelines recommend risk stratification using presentation characteristics and risk factors to determine which patients require noninvasive testing or should be referred directly to invasive catheterization<sup>3</sup>. However, in the current era, the results of using these recommended strategies are unsatisfactory. The population undergoing noninvasive testing has a low rate of obstructive CAD (10-20%) and very low annual event rates (~1-2%/year) <sup>4</sup>, <sup>5</sup>, <sup>59</sup>, while patients undergoing invasive angiography frequently don't have actionable CAD<sup>6</sup>. These patterns of care have resulted in high costs without accompanying clinical benefit<sup>7</sup>. A new approach to the risk stratification and subsequent diagnostic evaluation and management of patients with stable symptoms suggestive of CAD is urgently needed.

<u>Uncertainty Regarding the Optimal First Test for Detection and Exclusion of Coronary Artery</u> Disease: Evidence For cCTA

While a number of functional and anatomic non-invasive tests are available for the evaluation of stable chest pain patients, the optimal evaluation strategy for patients with stable chest pain is uncertain, and recommendations in current guidelines differ markedly. In a recent attempt to address these issues systematically, two large, multicenter, open-label, randomized controlled trials explored the diagnostic evaluation of patients with symptoms that may represent coronary artery disease. The SCOT-HEART (Scottish Computed Tomography of the HEART)<sup>4,59</sup> and PROMISE (PROspective Multicenter Imaging Study for Evaluation of chest pain)<sup>5</sup> trials sought to address evidence gaps in noninvasive testing in stable chest pain, an area in which few randomized trials had previously been conducted.

Key findings from SCOT-HEART and PROMISE: The overall results and important similarities and differences between the two trials have been recently described<sup>8</sup>. The SCOT-HEART study enrolled 4,146 patients with stable chest pain to cCTA in addition to usual care (which generally included electrocardiogram [ECG] stress testing) or to usual care alone. The trial used an upstream primary endpoint related to diagnostic thinking: managing clinician certainty of the diagnosis of angina secondary to CAD, which showed an increase in the cCTA group (RR: 1.79; 95% confidence interval [CI]: 1.62 to 1.96), as did the secondary endpoint of certainty of diagnosis of CAD (RR: 2.56; 95% CI: 2.33 to 2.79). The clinical outcomes-related secondary endpoint of the rate of cardiovascular death or nonfatal myocardial infarction (MI) appeared to be reduced in the cCTA group at 20 months (RR: 0.62, 95% CI: 0.38 to 1.01; p=0.0527), although the overall event rates were low in both arms, reflecting the inclusion of a large number of patients without

CAD. Of note, a landmark analysis excluding the 7 week delay to receiving a cCTA yielded a hazard ratio of 0.50 for CV death and MI<sup>9</sup>.

The larger PROMISE trial randomly assigned 10,003 symptomatic, stable outpatients requiring evaluation for suspected CAD to either initial cCTA or functional stress testing (exercise treadmill testing [ETT], nuclear stress testing, or stress echocardiography), with a median follow-up of 25 months. The event related composite primary endpoint (death, MI, hospitalization for unstable angina, or major cardiovascular procedural complication) occurred at similar rates in the cCTA and functional testing groups (3.3% and 3.0%), which was lower than previously established historical rates. More patients in the cCTA group underwent cardiac catheterization within 90 days after randomization (12.2% vs. 8.1%), but the secondary endpoint of the frequency of catheterization showing no obstructive CAD was significantly lower in the cCTA group (3.4% vs. 4.3%, p=0.02) as was the rate of death and MI at 12 months (HR 0.66; p=0.049). Furthermore, among patients randomized to an intended nuclear testing strategy, the mean cumulative radiation exposure was lower in the cCTA group compared with the functional testing group (12.0

- 8.4 mSv vs. 14.1 - 7.6 mSv). This encompassed all downstream radiation within 90 days, including that associated with cardiac catheterization, and is particularly intriguing because more cCTA patients received cardiac catheterization.

In addition to improving triage to the cardiac catheterization lab and potentially reducing radiation exposure, mounting evidence has demonstrated that use of cCTA, compared to functional testing, yields improved preventive medical treatment and better prognostic information<sup>4, 5, 10</sup>. Patients in the PROMISE trial who underwent cCTA experienced greater uses of indicated cardio-protective medications such as aspirin and statins<sup>10</sup>. This increase is prognostically important, as data from the CONFIRM registry (Coronary CT Angiography Evaluation for Clinical Outcomes International Multicenter) demonstrated that baseline statin therapy among patients with non-obstructive CAD<sup>11</sup> identified on cCTA was associated with a reduction in mortality compared to non-use<sup>12</sup>, while statin therapy among patients with obstructive CAD identified on cCTA was associated with a reduction in MACE<sup>13</sup>.

The identification of non-obstructive CAD with high risk plaque characteristics can only be accomplished non-invasively by cCTA and is an important prognostic indicator, with even mild abnormalities conferring nearly three times the risk of death, MI and unstable angina compared to patients with a normal study<sup>14, 15</sup>. Furthermore, cCTA leads to higher yield of positive results with actionable or obstructive CAD, among patients undergoing cardiac catheterization<sup>5</sup>. This is in line with data from the CONFIRM registry, where investigators demonstrated that cCTA could be used as an effective gatekeeper prior to invasive coronary angiography<sup>16</sup>.

Most importantly, a recent meta-analysis largely based on PROMISE and SCOT-HEART data showed a clear benefit in 'hard' cardiovascular outcomes to a cCTA first strategy, with a 29% reduction in MI<sup>17</sup>. This was potentially driven by the increase in medication utilization in the cCTA arm of the study as well as more catheterization and revascularization<sup>17</sup>.

To summarize, there are several practical and clinical implications of SCOT-HEART and PROMISE which inform the proposed design of PRECISE:

Contemporary patients with stable chest pain are at low risk of clinical events. Therefore, a
strategy to test only those with an elevated likelihood of having obstructive CAD or risk for
events, while instituting optimal medical care including deferring testing in those unlikely to
benefit (i.e. using the PROMISE Risk Score), may be feasible, clinical important and efficient.

- cCTA is a reasonable first test for routine assessment of patients with stable chest pain, and when compared to functional testing, is associated with an increase in preventive medication use and a reduction in myocardial infarction.
- Future trials investigating the optimal evaluation of patients with stable chest pain should include the evaluation of clinical outcomes and other measures of testing efficiency (i.e., cardiac catheterization without obstructive CAD).

#### The Case for the Use of cCTA with selective FFR<sub>CT</sub> as the Optimal First Test

The current noninvasive diagnostic testing strategies using functional testing have relatively poor accuracy given the low disease prevalence in this population, leading to high rates of false- positive results<sup>18</sup>. Specifically, current diagnostic strategies lead to high rates (~50%) of cardiac catheterization without significant obstructive disease or need for revascularization<sup>5,7</sup>. As described above, incorporating cCTA into testing strategies can reduce the frequency of cardiac catheterization without obstructive disease but tends to increase rates of invasive angiography <sup>4, 5</sup>

Non-invasive computationally-derived FFR<sub>CT</sub> has been developed using resting coronary CT images without the administration of adenosine or change in underlying cCTA protocols¹8-21. The methodology has been previously described elsewhere.²² In short, FFR<sub>CT</sub> uses the accurate anatomical model of the coronary arteries and myocardium obtained with conventional cCTA and applies the physical laws that govern flow, microcirculatory resistance, coronary branching, and simulated hyperemia. The Navier-Stokes equations that solve for velocity, resistance and pressure for all Newtonian fluids are applied to provide a 3-dimensional pressure map across the coronary tree. This use of computational fluid dynamics generates FFR values from 0 to 1, with ≤0.80 considered hemodynamically significant. The values are congruent with invasive FFR, as shown in several prospective validation studies¹8-20. Finally, the anatomical modeling has been improved by the use of advanced deep and machine learning techniques applied to the large data sets acquired via central analysis.

The addition of FFR<sub>CT</sub> may reduce a potential limitation of a cCTA-first approach, excess invasive angiography, by providing both functional and anatomic data. Specifically, FFR<sub>CT</sub> markedly reduces the false positive rate of cCTA alone vs. invasive FFR adjudicated ischemia with 68% of false positive CT interpretations in the NXT Trial reclassified as true negative. A retrospective analysis from the PROMISE trial in 181 patients with cCTA, cardiac catheterization and FFR<sub>CT</sub> revealed that FFR<sub>CT</sub> was a better predictor of revascularization and events than cCTA alone. Modelling of the incorporation of FFR<sub>CT</sub> into catheterization decision making suggested a reduction in catheterization rate with cCTA from 12.2% to 7.8% while reducing the rate of catheterization without obstructive CAD from 27% to 15% and increasing the yield of catheterization leading to revascularization from 49% to 61%<sup>23</sup>. Given that PCI of lesions with negative FFR is associated with worse outcomes<sup>24, 25</sup>, while treatment of FFR positive lesions with PCI vs. optimal medical therapy results in improved clinical outcomes, the potential clinical value of adding FFR<sub>CT</sub> to a cCTA based diagnostic strategy is evident.

The safety and utility of a CT/ FFR<sub>CT</sub> strategy were further tested in the PLATFORM Study (Prospective LongitudinAl Trial of FFR<sub>CT</sub>: Outcome and Resource Impacts) which evaluated rates of invasive catheterization without obstructive CAD in patients undergoing invasive evaluation. Patients in 2 sequential non-overlapping cohorts of patients referred for ICA were assigned to either undergo ICA or cCTA/ FFR<sub>CT</sub> with ICA use based on the results of the cCTA and FFR<sub>CT</sub>. The cCTA/FFR<sub>CT</sub> strategy resulted in a significant reduction in the rate of cath lab finding of no obstructive disease, from 73 to 12%<sup>7</sup>. Furthermore, ICA was deferred in 61% of cCTA/FFR<sub>CT</sub> strategy patients. A follow-up at one year demonstrated that cCTA with selective FFR<sub>CT</sub> strategy yielded similar clinical outcomes and quality of life, at a substantially reduced cost.

While much of the early focus has been on a reduction in referral for ICA in the absence of actionable CAD, more recently there has been growing interest in using FFR<sub>CT</sub> to enhance catheterization lab efficiency by increasing the proportion of catheterizations that include revascularization (PCI or CABG / ICA ratio) and providing guidance regarding revascularization strategies before the invasive angiogram. Importantly, in this case FFR<sub>CT</sub> is not being used only in a binary fashion but rather to provide a richer understanding of the pattern and degree of pressure loss across the epicardial coronary system and its connection to the extent of ischemia present.

The value of cCTA and FFR<sub>CT</sub> has been recognized by The National Institute for Health and Care Excellence (NICE) in their advisory for stable chest pain (Clinical Guidance 95) and technical evaluation of FFR<sub>CT</sub>, as well as by establishment of reimbursement standards by the Centers for Medicare and Medicaid Services (CMS) <sup>26, 27</sup>. The 2016 NICE guidance recognized the difficulties with risk stratification in an era of reduced obstructive CAD prevalence in the population undergoing evaluation and the importance of anatomical assessment of CAD<sup>26, 27</sup>. In response, it recommends coronary cCTA as the first-line investigation for patients presenting with new-onset chest pain felt to be due to CAD based on its superior clinical diagnostic utility and cost- effectiveness<sup>26, 27</sup>. Further, based on the results of the PLATFORM trial, the NHS recommends addition of FFR<sub>CT</sub> to cCTA as a cost savings measure<sup>26</sup>. In the United States, CMS approved a New Technology Ambulatory Payment Classification (APC) for HeartFlow FFR<sub>CT</sub> analysis on January 1, 2018<sup>28</sup>. The acknowledgement of FFR<sub>CT</sub> by CMS is a critical step toward increasing the availability of the technology to patients who may benefit. However, other organizations' standards documents have not yet been revised to incorporate the emerging evidence base supporting CCTA and FFR<sub>CT</sub>, indicating that there is still a need for additional evidence to support the routine use of FFR<sub>CT</sub> in clinical practice.

## Rationale and Evidence for Incorporation of a Strategy of Guideline-recommended Care without Planned Testing in Low Risk patients

Given the low prevalence of obstructive CAD (10-20%) and very low annual event rates (~1-2%/year) among stable chest pain patients undergoing non-invasive testing, combined with the high cost of testing<sup>4, 5</sup>, prospective evaluation of the safety and efficacy of an approach of guideline-recommended care without planned testing has become a necessity. Although there are no data regarding outcomes and costs of a guideline-recommended care without planned testing in symptomatic patients, it is possible to define in principle a cohort in whom deferred testing might be the optimal strategy. The argument for testing this is further strengthened by the equivalence of medical and invasive strategies in preventing cardiovascular events in stable CAD, as several trials have shown no benefit of revascularization over optimal medical treatment <sup>29, 30</sup>. It is reasonable to hypothesize that this may be especially true for those at lowest risk, in whom noninvasive testing is even less likely to lead to outcomes-improving revascularization, thereby removing the need for testing as a gateway to the catheterization laboratory.
The COURAGE trial (Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation) demonstrated no significant difference in a composite of death, myocardial infarction, and stroke between patients with objective evidence of myocardial ischemia and significant CAD on medical therapy vs. those undergoing PCI (19.5% vs. 20.0%, p=0.62)<sup>29</sup>. The more recent ORBITA trial (Percutaneous coronary intervention instable angina) randomized 200 patients with stable angina and a single-vessel stenosis to optimal medical therapy + PCI vs. optimal medical therapy plus a sham procedure, with a primary endpoint of difference in exercise time during a 6-week follow-up period<sup>30</sup>. The authors found no significant difference in improvement in exercise time (+28.4 seconds in PCI group vs. +11.8 seconds in sham group, p=0.2), nor any significant change in the secondary outcome of Seattle Angina Questionnaire (SAQ)-angina frequency from baseline (14.0 in PCI group vs. 9.6 in sham group, p=0.26)<sup>30</sup>. The ongoing improvements in medical management of CAD risk, angina and established coronary artery disease further emphasize the need for diagnostic strategies that minimize unnecessary invasive angiography and revascularization by emphasizing guideline-recommended care in patients at very low risk for obstructive disease.

These studies support the development of a patient-centric strategy to identify those who may derive minimal benefit from testing, a strategy which carries several desirable implications for patients, clinicians, and clinical practice in general. For patients, this process can mean a reduction in use of testing from which they would not benefit, thereby saving time, anxiety, and cost, as well as potential reductions in radiation exposure and false-positive test results that could lead to more invasive, unnecessary procedures. For clinicians, a tool identifying the lowest risk patients has the potential to help optimize office-based decision making. From a practice and societal perspective, in an era in which practitioners are increasingly held accountable for costs and quality, the ability to confidently identify patients highly unlikely to benefit from potentially expensive testing and who may therefore be managed conservatively has many potential economic and process-of-care advantages.

The PROMISE Risk Tool was expressly developed to identify low-risk patients with stable chest pain who are unlikely to benefit from non-invasive testing, and for whom guideline-recommended medical management alone may be safe. Current guidelines recommend using a version of the Diamond and Forrester risk score for pretest likelihood of obstructive CAD, but multiple investigators have found that this tool grossly over estimates actual presence of disease<sup>5, 31, 32</sup>. The consequence is an imprecise evaluation strategy for millions of patients, resulting in unhelpful testing of lower risk individuals. For a significant portion of these, a false positive functional testing leads them to have invasive cardiac catheterizations to rule out the disease they do not have. The Risk Tool developed using the PROMISE cohort employs 10 readily available clinical variables (such as tobacco usage, ethnicity/race, and age) and has been validated in the SCOT-HEART population<sup>33,</sup> <sup>34</sup>. This risk tool identifies patients with stable chest pain who have no coronary plague or calcification by cCTA and no cardiac events over 2 years, and who therefore would be predicted to derive minimal or no value from noninvasive testing<sup>33, 34</sup>. Testing whether this risk tool can be employed prospectively to safely and effectively risk stratify low risk patients into a strategy of guideline-recommended care with symptom and risk factor management and without diagnostic testing is one of the core secondary objectives of the PRECISE research program.

#### III.B. Rationale for the Current Study: A Precision Approach to Chest Pain Evaluation

Despite the high-burden of stable chest pain in the U.S., and the enormous research literature reporting on the comparative effectiveness of different options, no single diagnostic strategy has emerged with a broad consensus of support. Each testing community continues to favor its own technology and the clinicians who must select the testing approach to use for their patients are caught in the middle, unable to resolve the controversies that have characterized this area of cardiovascular medicine for decades. The situation is complicated by the heterogeneity of the current population's burden of disease. More than a quarter (27%) of the PROMISE cohort had no coronary plaque whatsoever, while high-risk CAD, defined as left main stenosis ( $\geq$ 50% stenosis) or either (a)  $\geq$ 50% stenosis '[50]' or (b)  $\geq$ 70% stenosis '[70]' of 3 vessels or 2-vessel CAD involving the proximal left anterior descending artery was identified in 6.6% [50] and 2.4%

[70] of patients. Thus, the first goal of any optimal management strategy for stable symptoms in patients with suspected CAD is determination of an individual patient's risk. Using the PROMISE Risk Tool to accurately assess patient risk<sup>33, 34</sup>, we will prospectively test the hypothesis that low risk patients can be correctly identified with only baseline clinical data and that emphasizing guideline-recommended care while deferring testing in these patients improves chest pain decision making by reducing unnecessary invasive angiography without leading to an increase in MACE, and by reducing cost.

Among patients in whom contemporary risk evaluation suggests an elevated risk for obstructive CAD, the observational data suggest that cCTA with selective FFR<sub>CT</sub> may improve appropriate triage to invasive angiography<sup>5, 23</sup>, while reducing cost<sup>9</sup>.

Thus, the case for an adequately powered randomized clinical trial with a pragmatic design, comparing clinical outcomes following testing strategies regularly used in current clinical practice to a precision evaluation strategy is compelling. PRECISE is designed to be that trial.

If the findings of PRECISE are positive as hypothesized, it is expected that the trial will lead to updates in appropriate use criteria, clinical practice guidelines, and payer policies such that cCTA with selective FFR<sub>CT</sub> receives a class IA recommendation for stable chest pain patients to improve outcomes and reduce costs. PRECISE will identify those chest pain patients for whom non- invasive testing may be safely deferred and simultaneously improve the efficiency of testing for elevated risk patients. The results of this study will shift the paradigm of clinical thinking in this area from the current approach of identifying a single best test for all, to incorporating a patient- centric risk-based evaluation and management strategy for stable chest pain patients.

#### IV. STUDY OVERVIEW AND OBJECTIVES

#### IV.A. Overview of PRECISE

PRECISE is a multicenter, randomized, trial that will enroll approximately 2100 participants in a comparison of a risk-based precision evaluation strategy of guideline-recommended medical management without planned testing (in minimal risk participants) and cCTA with selective FFR<sub>CT</sub> (in elevated risk participants) with usual care in stable symptomatic patients with suspected significant CAD.

#### Location

Participants will be enrolled at approximately 100 sites in the US and outside of the US. No center may enroll more than 315 (15%) participants in the trial.

#### Participant Population and Selection

Participants will be symptomatic patients with suspected significant CAD and a stable clinical course who are recommended by their managing clinician to have a non-invasive diagnostic test or ICA. Patients will be excluded if they have any history of documented CAD (including revascularization, myocardial infarction or any degree of CAD proven by imaging) or have had diagnostic cardiovascular testing for suspected CAD within the last year. Patients will also be excluded if their symptoms are not clearly stable or if their managing clinician feels testing is needed on an urgent or emergent basis.

Diagnostic testing for the assessment of CAD symptoms is ordered by physicians and other clinicians from many specialties and is performed in multiple settings, including physician offices, hospital outpatient departments, and diagnostic testing facilities. A trial, such as PRECISE, that seeks to improve the management of non-ACS chest pain must incorporate this diversity in order to be broadly relevant to the target population under study. PRECISE site selection will seek to encompass this diversity.

#### Study duration

The anticipated total duration of the PRECISE study will be approximately 36 months for start-up, enrollment, follow up, and close out. Participants will be followed for 12 months after enrollment.

#### Study design

The figure below represents a diagrammatic representation of the trial design.



#### **IV.B. Primary Objective and Endpoints**

The primary objective of the PRECISE study is to assess clinical outcomes, patient-reported outcomes, decision making regarding noninvasive testing and invasive angiography, and costs using a precision evaluation strategy as compared to a usual care strategy in participants with stable symptoms suggestive of significant coronary artery disease. The precision evaluation strategy will be based on a pre-test risk assessment which will be used to assign participants to either cCTA with selective FFR<sub>CT</sub> or guideline-recommended care with symptom and risk factor management and no immediately planned testing. In addition, patients with known mild coronary plaque without obstructive stenosis or extensive coronary calcium randomized to the precision evaluation arm are mandated to undergo cCTA +/- FFR<sub>CT</sub>, independent of their PROMISE risk score strata. We hypothesize that in stable patients with a clinical recommendation for testing to evaluate suspected significant CAD, the proposed precision evaluation strategy will improve outcomes and reduce costs compared to usual care evaluation.

The primary endpoint is a composite of: MACE (all cause death and non-fatal MI) or invasive cardiac catheterization without CAD (no coronary stenosis ≥50% according to QCA by core-lab adjudication or site interpretation if QCA is not available, or with FFR≤0.80, instantaneous wave free ratio (iFR) ≤0.89) or other validated NHPR. The primary study hypothesis will be tested at one

year using an intention to treat analysis.

#### IV.C. Secondary Endpoints

Endpoints will be assessed at 45 days, 6 months, and 1 year. Secondary endpoints include:

- 1. Hierarchical analysis (Finkelstein and Schoenfeld (FS) and Pocock's win ratio) of primary endpoint (gives priority to clinical importance of the components of the composite outcome rather than time to event)
- 2. Resource use patterns (all participants) and medical costs (US participants): resources to be assessed include index testing, follow up testing, diagnostic and other cardiac procedures and hospitalizations. Primary comparisons will be made at 12 months.
- 3. QoL: the Seattle Angina Questionnaire (SAQ) will be used to assess angina-specific Quality of Life; the EuroQoL 5D (EQ-5D-5L) survey will be used for a brief assessment of overall (generic) health status; patient satisfaction with diagnostic process will be assessed once at 45 days using a 4-item instrument created for this trial.
- 4. Death: All-cause, cardiovascular, non-cardiovascular
- 5. Myocardial infarction: All, procedural, spontaneous MI
- 6. Hospitalizations: All, cardiovascular, non-cardiovascular, and for progressive or unstable angina
- 7. Rates of preventive medication use (ASA, statins) in participants with clinical indication for use: hyperlipidemia, diabetes, documented CAD
- 8. Cumulative radiation exposure at 1 year
- 9. Proportion of invasive coronary angiogram patients who undergo revascularization (PCI or CABG) within 6 months of enrollment (catheterization efficiency)

#### IV.D. Rationale for the Selection of Outcome Measures

#### Rationale for Clinical Assessments

Major adverse cardiovascular events (MACE) are a primary concern for clinicians and patients presenting with stable chest pain. The primary composite endpoint of MACE at 12 months (all cause death, non-fatal MI), invasive cardiac catheterization without obstructive CAD (diameter stenosis ≥50% by QCA, FFR≤0.80 or iFR≤0.89) is clinically relevant and, the components taken together, represent a sound measure of an effective diagnostic chest pain evaluation<sup>4, 5, 35, 36</sup>. The selection of 12 months is based on the rationale that the longer the duration between the evaluation strategy and an eventual outcome, the less likely it is that the evaluation strategy is directly related to the outcome of interest. In PROMISE, there was a significant reduction in death and MI in the cCTA arm compared to the usual care arm at 12 months, which was no longer significant after a median 25 months of follow-up<sup>5</sup>. The use of this composite clinical endpoint will be critical to assessing the PRECISE hypothesis that a precision evaluation strategy with cCTA and selective FFR<sub>CT</sub> and guideline-recommended medical management without planned testing will yield superior outcomes at lower cost compared with a usual care testing strategy.

#### Rationale for Economic and Quality of Life (QoL) Assessments in PRECISE

Non-invasive diagnostic testing for the evaluation of stable chest pain represents a significant cost

to the U.S. and other healthcare systems. In the past when payers in the US have attempted to control costs by reducing the reimbursements provided for diagnostic testing, clinicians responded by increasing the number of tests obtained. An emphasis on generating evidence for cost-savings via a safer and more efficient approach is critical in enhancing value while reducing the financial burden on patients, providers, and the system alike. In addition, this precision-based approach to diagnostic evaluations in CAD participants may result in improvements in the quality of care of our participants. Further, since there has been no prospective trial of guideline- recommended care without planned testing, the ability of such an approach to provide equivalent symptom relief compared with usual care is of great importance and critical to the evaluation of this approach. For these reasons, the potential impact of a precision-based approach on resource use and QoL must be evaluated in PRECISE.

#### IV.E. Rationale for Selection of Testing in Each Arm

#### Usual Care Arm

Functional stress testing with stress nuclear, stress echocardiography, and exercise ECG for the diagnosis of CAD is well-established in clinical practice (ACC/AHA 2012 Stable Ischemic Heart Disease guidelines, class I, Level of Evidence (LOE) B³7. While stress CMR is less commonly used, it also receives a class IIa, LOE B recommendation in patients who are unable to exercise³7 and is used in some centers. In contrast, it is common for patients to be referred direct to diagnostic angiography without undergoing a functional test. This group represents up to 50% of elective catheterization populations and is thus an important usual care approach to suspected CAD³5, ³8, ³9. In order to accurately capture the wide variety of testing strategies available to and used by community clinicians and real-world practice patterns, a usual care strategy arm with site clinician decision-making should include all of the above options. This will improve the generalizability of the trial while accurately capturing the potential impact of the implementation of a precision approach. Participants with history of known obstructive CAD (prior myocardial infarction, CABG or PCI, stenosis ≥50%) are excluded from enrollment into the trial. In all participants in the usual care arm, cCTA is prohibited as a subsequent test for the first 45 days after randomization.

#### Precision Evaluation Arm

PRECISE will evaluate whether a precision evaluation strategy that combines contemporary risk stratification using the PROMISE Risk Tool with functional and anatomic non-invasive evaluation with cCTA with selective FFR<sub>CT</sub> can improve outcomes over usual care in stable chest pain patients while safely deferring further testing in low-risk patients and reducing cost overall. While current guidelines recommend the non-invasive and invasive initial testing approaches for patients with stable chest pain<sup>37</sup>, current practice is known to lead to high rates of ICA without obstructive CAD<sup>6, 40</sup>. Further, although guidelines also recommend no testing in the lowest risk groups (pre-test probability of obstructive CAD <10 or 15%), currently available risk tools result in many clinicians appearing to ignore this recommendation: current patterns of care using available risk stratification tools results in testing populations with a prevalence of obstructive CAD of only 10-20%, and a prevalence of no coronary plaque of >25%<sup>4, 5</sup>. The intervention in PRECISE will triage patients into two risk groups who will be assigned to receive either guideline-recommended medical management without planned testing or cCTA with selective FFR<sub>CT</sub>. The PROMISE Risk Tool can identify low-risk patients with stable chest pain that would be expected to derive minimal value from noninvasive testing and is superior to either Framingham Risk Score or Diamond and Forrester assessments<sup>33</sup>.

<sup>34</sup>. cCTA with selective FFR<sub>CT</sub> represents a combined functional and anatomic testing modality that can lower the frequency of finding no obstructive CAD at catheterization and thus reduce costs<sup>7,41</sup>.

#### IV.F. Randomization Method

Participants who meet all inclusion criteria and none of the exclusion criteria will be randomized in a ratio of 1:1 within a clinical center to either a precision evaluation strategy or usual care using an interactive web or voice-based system (IXRS). Randomization will be stratified by intended first test (if randomized to usual care) and by classification as low vs. elevated risk by the minimal risk model. Participants with known non-obstructive plaque will be included in the elevated risk strata regardless of risk score. The randomization scheme within a clinical center will be carried out by the method of random permuted block design with variable block size.

Enrollment in the randomization strata of intended first test being noninvasive (vs. direct to catheterization) will be capped at 90% of the sample size.

Risk will be classified by a risk tool using pre-test clinical characteristics (including tobacco usage, ethnicity, and age) derived in the PROMISE trial and validated in SCOT-HEART or by the presence of non-obstructive plaque/CAC < 100 AU. Participants randomized to follow a precision strategy group will be assigned to either guideline-recommended care with symptom and risk factor management and no immediately planned testing (low risk group) or cCTA with selective FFR<sub>CT</sub> (elevated risk of obstructive coronary disease and/or events). Participants randomized to precision evaluation and risk stratified into the low risk group and their providers will be provided informational materials explaining the rationale for this decision and the safety of this strategy based on outcomes of similar participants in the PROMISE trial.

Participants randomized to usual care will undergo either noninvasive stress testing or invasive testing (direct to diagnostic catheterization), as recommended by their managing clinician and agreed to by the participant. Acceptable noninvasive testing options will include exercise electrocardiogram, stress nuclear imaging (including PET), stress MR or stress echocardiogram. The use of cCTA is explicitly excluded as the initial diagnostic strategy in this arm and prohibited as a subsequent test for the first 45 days after randomization.

In both arms, all subsequent decisions regarding additional testing, medications, and/or procedures will be at the discretion of the responsible clinical care team. Each care team will be provided with informational materials summarizing current standards for test interpretation and preventive care. However, specific medical treatment will not be mandated by the study.

#### IV.G. Diagnostic Evaluations and Subsequent Care

#### Description of Evaluations to be performed

Participants will be assessed per the individual clinicians' routine approach to patients presenting with stable chest pain. Initial evaluation will include an appropriate medical history, physical examination, resting 12-lead ECG, and other routine blood work. A pregnancy test will be required for female participants of childbearing potential (those who have not been surgically sterilized or are not postmenopausal), and a creatinine blood test will be required for participants without a

recent normal value (most recent measurement taken within previous 90 days). At the time of randomization, the site clinician will specify the preferred first diagnostic strategy (noninvasive stress test vs. direct to catheterization) if randomized to the usual care arm and this choice will be used to stratify randomization. Also part of the randomization process, every participant will undergo risk stratification with the PROMISE risk calculator although sites will be blinded to results. Participants randomized to the precision evaluation arm will be assigned to either no planned testing vs cCTA/FFR<sub>CT</sub> based on risk score results and the presence of known non-obstructive coronary atherosclerosis.

Sites will be provided with informational materials outlining standards of care for all noninvasive test interpretation. Guideline recommendations for care and informational materials on symptom and risk factor management will also be provided. These are intended to be followed for all participants. Participant-friendly versions of these materials will be provided to sites and may be used as handouts.

Symptoms and Quality of Life (QoL) will be assessed by the EuroQoL 5D (EQ-5D-5L) survey to assess overall (generic) health status and the Seattle Angina Questionnaire (SAQ) to assess angina-specific Quality of Life.

#### Equipment, Protocols & Interpretation

All participating sites will use standard equipment and procedures for usual care testing, including diagnostic angiography, stress echocardiography, stress nuclear perfusion imaging, stress CMR, and exercise ECG as defined by current practice guidelines<sup>42-49</sup>. Sites must also use at least 64-slice multi-detector computed tomography (MDCT) for coronary cCTA<sup>49, 50</sup>. All testing protocols will be in accordance with current best-practice standards<sup>42-48, 50</sup>.

#### <u>Interpretation</u>

The interpretation of all diagnostic tests will be performed in a timely fashion and will capture the presence and extent of findings including diagnosing or excluding CAD (diagnostic angiography), fixed or inducible LV perfusion and wall motion abnormalities (stress echo, cMR and stress nuclear), and functional capacity (in the case of exercise ECG, exercise echo and exercise nuclear). The site interpretation and clinical report of all diagnostic tests, including noninvasive stress testing, cCTA and invasive angiography, will be uploaded through the EDC.

cCTA study interpretation will be carried out by site physicians with at least ACC COCATS (Core Cardiology Training Symposium) level 2 training, Society of Cardiovascular Computed Tomography level 2, recognized by the Certification Board of Computed Cardiovascular Tomography, or equivalent<sup>50</sup>. Certification by the Certification Board of Nuclear Cardiology or Board Certification in nuclear medicine or radiology will be considered satisfactory for interpretation of stress nuclear imaging studies. Stress echo and cMR readers also be at least COCATS level 2 trained or equivalent. Prior to being opened to participant enrollment, sites will be certified to ensure that quality cCTA images can be obtained.

#### Referral of precision evaluation cCTA participants for FFR<sub>CT</sub> determinations

Participants randomized to the precision evaluation arm who are either 1) determined to be at elevated risk or 2) have known non-obstructive coronary atherosclerosis will undergo cCTA as the initial diagnostic strategy according to current best practice standards. Image sets showing at least

one 30-90% stenosis in epicardial vessels of 2mm diameter or greater should be promptly sent to HeartFlow for analysis of FFR<sub>CT</sub>. Results will be returned to sites in < 24 hours to enable rapid incorporation into clinical decision making.

#### Subsequent Care

Subsequent care will be provided by the individual site clinicians at their own discretion, with encouragement to follow guideline-based approaches. Information will be provided to the individual sites on diagnostic test interpretation and subsequent management approaches for the various imaging modalities, including relevant guideline recommendations for primary and secondary prevention.

For patients in the Precision Evaluation Arm, ICA should not be performed unless at least one of the following criteria are met:

- Any stenosis ≥90% identified by cCTA
- Left Main stenosis ≥30% identified by cCTA
- Plaque rupture identified by cCTA
- Lesion-specific FFR<sub>CT</sub> ≤0.85 in vessels with reference vessel diameter of 2.0mm or greater

#### Need for testing in low risk participants randomized to the precision care arm

Participants randomized to the precision evaluation arm and determined to be at low risk will be treated for symptoms and risk factor management according to current guideline recommendations. While it is expected that this will resolve symptoms in nearly all cases it is recognized that chest pain will persist in some despite medical treatment. In some cases, additional non-cardiac diagnostic testing may be pursued. In other cases, the site clinician may decide that further cardiac testing is warranted, in which case a cCTA followed by selective FFR<sub>CT</sub> should be performed. Details regarding such decision making will be captured in the case report form.

#### V.STUDY PROCEDURES

#### V.A. Patient Screening for Eligibility

Patients will be screened by site personnel for eligibility and provided information about the study. Patients' not meeting inclusion and or having exclusion criteria will be documented as being excluded. Patients meeting inclusion and not meeting any exclusion criteria will be provided an informed consent form to review and sign prior to being randomized into the study.

#### **Inclusion Criteria**

- 1. Age ≥18 years
- 2. Stable typical or atypical symptoms suggesting possible significant coronary artery disease (CAD) with further non-emergent testing or elective catheterization recommended to evaluate the presence of suspected significant CAD. Stable chest pain (or equivalent) includes those who have fully been ruled out for Acute Coronary Syndrome (ACS) and for whom elective testing is recommended, regardless of the venue in which they are seen.
- 3. If prior CV testing has occurred, it must have been performed greater than one year prior to randomization, and the following must be met:
  - a) cCTA or invasive coronary angiography (ICA) with stenosis < 50%
  - b) Quantified coronary artery calcium (CAC) < 100 AG
- 4. Safe performance of cCTA:
  - a) Creatinine clearance ≥45 ml/min per most recent measurement within 90 days
  - b) For a female participant of childbearing potential (those who have not been surgically sterilized or are not postmenopausal), a pregnancy test must be performed with negative results known within 7 days prior to randomization
- 5. Willingness to comply with all aspects of the protocol, including adherence to the assigned strategy and follow-up visits regardless of actual testing performed
- 6. Ability to provide written informed consent

#### **Exclusion Criteria**

- 1. Acute chest pain (in patients who have not been ruled out for ACS)
- 2. Unstable clinical status
- 3. Noninvasive or invasive CV testing for CAD within 1 year. CV testing for CAD refers to any stress tests, invasive coronary angiography (ICA), and cCTA (including calcium scoring) only.
  - a) Resting ECG, resting echocardiogram and resting CMR (MRI) are not exclusionary regardless of when they were performed.
- 4. Lifetime history of known obstructive CAD (prior myocardial infarction, CABG or PCI, stenosis ≥50%), known EF≤40% or other moderate to severe valvular or congenital cardiac disease
- 5. Contraindications to cCTA including but not limited to creatinine clearance (GFR) <45 ml/min as per most recent measurement taken within 90 days
- 6. Exceeds the site's weight or size limit for cCTA or cardiac catheterization
- 7. Any condition leading to possible inability to comply with the protocol procedures and follow-up
- 8. Any condition that might interfere with the study procedures or follow-up
- 9. Enrolled in an investigational trial that involves a non-approved cardiac drug or device which has not reached its primary endpoint
- 10. Life expectancy less than 2 years due to non-cardiovascular comorbidities

#### Screening visit (in-person)

Participant will be randomized to either the usual care arm or the precision evaluation arm within 14 days of screening.

At the screening visit, patients will undergo the following:

- Review consent form and have all questions appropriately answered.
- Provide consent by signing the Informed Consent Form
- Review of medical history
- Review of concomitant medications
- Pregnancy test (for females of child-bearing potential those who have not been surgically sterilized or are not postmenopausal)
- Creatinine test (if not done in last 90 days)

Resting 12-lead ECG (optional, clinical care only) Assessment of CAD risk will be performed during screening to ensure eligibility. It will include:

- General medical history
- Cardiovascular risk factors and comorbidities as well as prior testing or events
- Physical exam
- Laboratory testing

The following major cardiac risk factors will be assessed:

- Age
- Sex
- BP/hypertension
- Diabetes
- Cholesterol (including low-density lipoprotein [LDL], high-density lipoprotein [HDL]), if available
- Smoking status
- Family history
- Sedentary life style
- Obesity (BMI, waist hip ratio)
- Cerebrovascular and peripheral arterial disease (PAD)
- Ankle brachial index (ABI)

#### V.B. Randomization and Enrollment

Once a participant has consented to participate in the trial, participant information will be entered into the database. If a patient is a screen failure, the data that has been collected up until this point for the patient for screening purposes will be entered into the case report forms (CRF) in the electronic data capture (EDC) system. No additional information will be collected after this point for such a patient.

For eligible participants, medical history data will be captured in the EDC. In addition, sites will need to specify the intended first test which would be performed if the participant is randomized to the usual care arm. The participant will then be randomized to either the usual care arm or the precision evaluation arm. Once randomization occurs, the participant is considered enrolled in the study. If randomized to the precision evaluation arm, participants will be further assigned to guideline-

recommended without planned testing or cCTA with selective FFR<sub>CT</sub>.

#### V.C. Participant Cohort Assignment

Participant will be randomized to either the usual care arm or the precision evaluation arm within 14 days of screening.

#### Usual Care Arm

Participants randomized to the usual care arm will undergo either noninvasive stress testing (exercise electrocardiogram, stress nuclear imaging including PET, stress MR, or stress echocardiogram), with the specific modality at the discretion of the participant's clinician, or invasive catheterization. In all participants in the usual care arm, cCTA is prohibited as a subsequent test for the first 45 days after randomization.

#### **Precision Evaluation Arm**

Participants randomized to the precision evaluation arm will be assigned a management approach based on their PROMISE Risk Score, a risk model based on pre-test clinical characteristics derived from the PROMISE trial and validated in SCOT-HEART<sup>34</sup> or the presence of known non- obstructive atherosclerosis. Participants will be assigned to either 1) guideline-recommended medical management without planned testing (low risk) or 2) cCTA with selective FFR<sub>CT</sub> (elevated risk or those with known plaque. independent of the PROMISE Risk Tool assessment). Participants assigned to the strategy of guideline-recommended medical management without planned testing will be treated with risk-appropriate preventive care and symptom control (including therapeutic trials of anti-anginal medications). Participants and their providers will be provided informational materials demonstrating the safety of this strategy based on pre-test probabilities and the PROMISE Risk Score. Participants with intractable symptoms despite maximal medical management whose clinicians opt for further testing (crossovers) will undergo cCTA with selective FFR<sub>CT</sub>.

Participants undergoing cCTA as the initial test (both assigned or crossover) should have  $FFR_{CT}$  analysis ordered if cCTA shows at least one 30-90% stenosis in epicardial vessels of 2mm diameter or greater. Image sets will be sent promptly to HeartFlow for analysis and results will be returned to sites in < 24 hours to enable rapid incorporation into clinical decision making.

#### V.D. Participant Follow-Up

Participants will be followed up at 45 (+/-14) days and at 6 and 12 months (+/- 30 days) after enrollment. For US participants, follow-up at 45 days and at 6 and 12 months will be done by phone interviews conducted by the DCRI Outcomes Call Center, unless not allowed by their enrolling site. For participants outside of the US, follow-up will be conducted by the site coordinators.

Activities to be conducted at each follow up contact are described below and in the Schedule of Events.

45 (+/-14) day follow-up visit (in-person, portions may be done by phone) At the 45-day follow-up visit, participants will be asked the following:

Assessment if any MACE has occurred since enrollment

- CV Update: Review and documentation of any cardiovascular diagnostic test, cardiovascular procedure, or hospitalizations/clinic visits due to cardiovascular symptoms and complications since enrollment
- Review and documentation of concomitant cardiovascular medication changes since enrollment
- Complete the following 3 questionnaires:
  - Seattle Angina Questionnaire
  - EQ-5D-5L Questionnaire
  - Participant Satisfaction Questionnaire
- Collection of the following:
  - o Any cardiovascular test both written report and test output
  - o Any cardiovascular imaging both written report and image file

#### 6 months (+/-30 days) follow-up contact

At the 6-month follow-up contact, participants will be asked the following:

- Assessment if any MACE has occurred since the 45-day visit
- CV Update: Review and documentation of any cardiovascular diagnostic test, cardiovascular procedure, or hospitalizations/clinic visits due to cardiovascular symptoms and complications since last visit
- Review and documentation of concomitant cardiovascular medication changes since enrollment
- Complete the following 2 questionnaires:
  - Seattle Angina Questionnaire
  - o EQ-5D-5L Questionnaire
- Collection of the following:
  - Any cardiovascular test both written report and test output
  - o Any cardiovascular imaging both written report and image file

#### 12 months (+/-30 days) follow-up contact

At the 12-month follow-up visit, participants will be asked the following:

- Assessment if any MACE has occurred since the 6-month visit/phone call
- CV Update: Review and documentation of any cardiovascular diagnostic test, cardiovascular procedure, or hospitalizations/clinic visits due to cardiovascular symptoms and complications since last visit
- Review and documentation of concomitant cardiovascular medication changes since enrollment
- Complete the following 2 questionnaires:
  - Seattle Angina Questionnaire
  - EQ-5D-5L Questionnaire
- Collection of the following:
  - Any cardiovascular test both written report and test output
  - Any cardiovascular imaging both written report and image file

## V.E. Testing in precision evaluation arm for participants assigned to no immediate testing

Precision evaluation participants determined to be at very low risk and assigned to the strategy of guideline-recommended medical management with no immediately planned testing are highly

unlikely (by definition) to have significant obstructive CAD. The managing clinician is encouraged to treat them with guideline-recommended preventive care, anti-anginal medications and other medical therapy as deemed appropriate to their clinical circumstances. This is expected to control or eliminate symptoms in most participants. In the unlikely event that symptoms are intractable or accelerating, despite reasonable medical treatment or if other compelling reasons for additional evaluation are present, testing may be warranted.

Unless there are urgent or emergent indications to proceed with invasive testing, all such participants requiring testing should have a cCTA followed by selective FFR<sub>CT</sub> rather than stress testing or elective invasive catheterization. cCTA with selective FFR<sub>CT</sub> should only be pursued if the participant is having:

- 1. Unstable/accelerating symptoms (i.e. no longer falls into stable angina cohort)
- 2. Continued stable symptoms despite risk factor modification including:
  - a) Optimized blood pressure control with goal <130/80 mmHg
  - b) Optimized lipid management with high-intensity statin in appropriate patients
  - c) Optimized diabetes management with blood glucose control in appropriate patients
  - d) Antiplatelet therapy in appropriate patients
  - e) Tobacco cessation in patients who smoke
  - f) Lifestyle counseling regarding diet exercise and stress reduction
  - g) Anti-anginal therapy including utilization of beta-blockers, calcium channel blockers, short and long-acting nitrates, and/or ranolazine

The assignment to no immediate testing is not time limited and is valid for the duration of the participant's enrollment in the trial. Testing in such participants should be infrequent and the reasons for this will be carefully documented and monitored.

#### V.F. Participant Withdrawal

In accordance with the Declaration of Helsinki, each participant is free to withdraw from the study at any time. Investigator(s) also have the right to withdraw participants from the study in the event of illness or other reasons concerning the health or wellbeing of the participant, or in the case of lack of cooperation. Should a participant decide to withdraw or should the investigator(s) decide to withdraw the participant, all efforts will be made to complete and report the observations up to the time of withdrawal as thoroughly as possible. If possible, a complete final evaluation at the time of the participant's withdrawal should be made. The reason for withdrawal must be noted in the eCRFs.

PRECISE Protocol CP-907-001-A Oct 11, 2019 v1.5

#### V.G. Schedule of Assessments

| | | Randomization | Day 45 | 6-mo. | 12-mo. |
|---|---|---|---|---|---|
| | Screening | Day 1 | ( +/-14 d) | (+/- 30d) | (+/- 30d) |
| Informed consent | X | | | | |
| Medical history | Х | | | | |
| Cardiovascular update 1 | | | Х | Х | Χ |
| Concomitant cardiovascular medications | Х | | Χ | Х | Χ |
| Cardiovascular risk factors (including PROMISE minimal risk score data entry for randomization) | Х | | | | |
| Pregnancy test <sup>2</sup> | Х | | | | |
| Creatinine | X | | | | |
| Resting 12-lead ECG | X | | | | |
| QoL evaluation: SAQ, EQ5D-5L | Х | | X | X | X |
| Participant Satisfaction Questionnaire | | | Х | | |
| Randomization | | Х | | | |
| Initial diagnostic invasive or noninvasive test performed (if assigned) | | Prior to 45 day<br>visit | | | |
| Cardiac imaging/testing clinical report and image collection | | | Х | Х | Х |
| Interval assessment for CV events and testing | | | Х | Х | Χ |
| Endpoint assessments | | | Х | Х | Χ |

During cardiovascular update, if participants have received an additional diagnostic test, a cardiovascular procedure or have been hospitalized since the last visit, additional data will be collected
 For a female participant of childbearing potential, a pregnancy test must be performed with negative results known within 7 days prior to randomization

<sup>3.</sup> Creatinine blood draw required only for participants without a recent normal value (most recent within previous 90 days)
4. Resting 12-lead ECG preferred in last 30 days (optional, clinical care only)

#### VI. ADDITIONAL ASSESSMENTS AND SUBSTUDIES

#### VI.A. Quality of Life Assessments

A short battery of instruments will be used to provide a relevant assessment of health-related quality of life that will capture the most likely health benefits to be associated with the precision strategy while not being burdensome to study participants. Quality of life (QoL) assessments will be conducted at baseline, 45 days, 6 months, and 12 months. Chest pain specific QOL will be assessed with the Seattle Angina Questionnaire (SAQ). While the full instrument has 19 items covering 5 dimensions of the impact of chest pain on QoL, we will use the scales for physical limitations, angina frequency, and disease perception/quality of life (14 items total)¹. These three scales will also allow calculation of the recently described 7-item short SAQ². The SAQ has been used as the primary disease-specific QoL outcome measure in a number of major clinical trials (including COURAGE, PROMISE, and ISCHEMIA) and is useful for this trial because it assesses chest pain and its impact on functioning and well-being regardless of whether the symptoms are due to coronary disease or are non-coronary. Since many participants in this study will be found not to have significant coronary disease and will be provided with that reassuring finding, the SAQ will allow us to assess the extent to which such information is associated with changes in the 3 dimensions noted above.

Overall health status will be assessed briefly using the EQ-5D-5L, a standardized generic measure that can also be used to link specific health states to general population-based utilities<sup>5</sup>. The EQ-5D-5L consists of two parts: (1) a descriptive assessment of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each of which can take one of five responses corresponding to the level of severity within each dimension, and (2) a self-rating 0- 100 "thermometer" of current health-related quality of life.

#### VI.B. Economic and Resource Utilization Assessments

The primary economic analyses in PRECISE will be performed from the perspective of the US health care system. Detailed information regarding the quantity and cost of health care services received by participants in each treatment group will be collected prospectively as part of the trial. Relevant health care resource consumption during initial testing through 1-year follow-up will be collected on the clinical trial electronic case report form (eCRF). (The cost of acute and non-acute hospital care will be derived from billing data collected from patients enrolled at US sites.) Physician and other outpatient care reported in the eCRF will be valued using secondary sources. Primary resource use and cost comparisons will be based on participants enrolled in the US. Secondary analyses will examine the consistency of treatment related differences in resource use in the US with the sites outside the US.

#### VI.C. Imaging and other Cardiac Assessments

For all participants in either arm in whom an invasive coronary angiogram is performed, procedural reports and angiographic images will be uploaded via the electronic data capture (EDC) system to create an angiographic image repository. In addition, the report, as well as imaging and / or graphic data from any procedures performed to assess stenosis significance or severity such as, FFR, IVUS, OCT should be uploaded. Similarly, for all participants receiving cCTA imaging, the cCTA images and reports will be uploaded via the EDC system to create an image repository. Invasive angiography will be evaluated by a core lab for QCA; other core lab(s) may be added to analyze

additional images.

### VII. ENDPOINT DETERMINATION, SAFETY, AND MONITORING

#### VII.A. Primary Endpoint Definitions

## Major Adverse Cardiovascular Events (all cause death, non-fatal myocardial infarction) All cause death

All cause death is defined as death resulting from any cause. In addition, the cause of death will be adjudicated, including cardiovascular death defined as death due to myocardial infarction, sudden cardiac death, heart failure, stroke, cardiovascular procedures, cardiovascular hemorrhage, or death due to other cardiovascular causes<sup>51</sup>.

#### Myocardial infarction

Acute myocardial infarction (MI) is defined as having evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia. Specifically, the Fourth Universal Definition<sup>51</sup> of type I MI is defined as:

Detection of a rise and/or fall of cTn values with at least 1 value above the 99th percentile URL and with at least 1 of the following:

- Symptoms of acute myocardial ischemia;
- New ischemic ECG changes;
- Development of pathological Q waves;
- Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality in a pattern consistent with an ischemic etiology;
- Identification of a coronary thrombus by angiography including intracoronary imaging or by autopsy.\*

cTn indicates cardiac troponin; ECG, electrocardiogram; URL, upper reference limit.

\*Postmortem demonstration of an atherothrombus in the artery supplying the infarcted myocardium, or a macroscopically large circumscribed area of necrosis with or without intramyocardial hemorrhage, meets the type 1 MI criteria regardless of cTn values.

A complete definition of the criteria for MI can be found in the Fourth Universal Definition of Myocardial Infarction (2018). This definition will be followed for spontaneous as well as periprocedural MIs, for which the elevation in cTn must be at least cTn values >5 times the 99th percentile URL for PCI and >10 times for CABG related infarctions<sup>51</sup>.

## Cardiac catheterization without obstructive coronary artery disease (diameter stenosis <50%, any FFR >0.80 or iFR >0.89)

Cardiac catheterization without obstructive coronary artery disease will be defined as the absence of any ≥50% stenosis or hemodynamic indication of significance in any major epicardial vessel including side branches ≥2 mm in diameter, as determined by core-lab adjudicated QCA. The Steering Committee may consider the use of other validated NHPRS as they become clinically available. Equivalent cut points for each approved test will be determined

at that time.

#### VII.B. Secondary Endpoint Definitions

#### Hierarchical analysis

Finkelstein and Schoenfeld (FS) and Pocock's win ratio analysis of primary endpoint is defined in section VII B Statistical Analysis Plan.

#### Resource use

Resource use is defined as counts and types of baseline testing, follow up testing, diagnostic and therapeutic procedures, and both inpatient and outpatient care. Costs from the US perspective will be estimated.

#### Quality of Life Metrics

Quality of Life assessments to be completed by the participants are the Seattle Angina Questionnaire and the EQ-5D-5L.

#### <u>Death</u>

Death will be categorized as all-cause, cardiovascular, non-cardiovascular.

#### Myocardial infarction

Myocardial infarction will be characterized according to the 4th Universal MI definition for both spontaneous and for periprocedural MI<sup>51</sup> MIs.

#### Hospitalizations

All, cardiovascular, non-cardiovascular, and for progressive or unstable angina. Urgent and unscheduled hospitalizations for other cardiovascular causes that do not meet the criteria for the specific events listed above will be classified as hospitalization for other cardiovascular causes (e.g., hospitalization for cardiac chest pain that does not meet the criteria for MI, hospitalization for arrhythmias, hospitalization for pulmonary embolism). Non-cardiovascular hospitalization are defined as any hospitalization whose primary cause is not thought to be CV in nature.

#### Preventive medication use

Information on preventive medication use will be acquired at study entry and 45 days. Participants with a clear clinical indication for use of ASA/antiplatelet agents and or, statins eg: hyperlipidemia, diabetes, documented CAD, will be characterized according to use/nonuse for each medication class.

#### Radiation safety endpoint – cumulative dose at 1 year

The cumulative radiation exposure over the 12 months following enrollment will be calculated based on the participant's exposure to radiation for cardiovascular care from one or more of the following modalities. For cCTA, the administered radiation dose (computed tomography dose index volume and dose length product for cCTA) will be recorded by the individual sites. For stress nuclear imaging, the radiotracer dose(s) will be collected and converted to equivalent radiation doses for comparison to cCTA. For ICA, the radiation dose from fluoroscopy administered will be recorded by sites and converted using standardized approaches to allow for comparison to radiation from cCTA. In instances in which the information required to assess actual dose is not available, a standard

dose based on accepted average exposures will be imputed for that form of testing. Cumulative radiation exposure from additional cardiac testing and procedures during the entire follow-up period will also be collected.

#### Catheterization efficiency

The proportion of invasive cardiac catheterization patients who undergo revascularization (PCI or CABG) within 6 months of enrollment will be determined.

#### **VII.C Testing Complications and Reporting**

The study intervention is the implementation of a precision evaluation strategy compared to usual care evaluation in non-acute chest pain participants with no history of CAD or recent testing whose clinicians recommend non-emergent non-invasive testing or ICA. Since all trial procedures represent standard of care for the eligible study population, there are no specific safety events associated with investigative procedures in this trial. However, there are known complications from these clinically recommended tests and procedures which are outlined below. These complications will be reported by site personnel.

#### For Precision Evaluation Strategy

#### For Guideline-recommended Medical Management

While participants assigned to the guideline-recommended care with no planned testing arm will have exceedingly low risk of events and are predicted to derive minimal or no value from noninvasive testing<sup>33, 34</sup>, there is a very small risk of missing left main or 3-vessel disease for which revascularization may be life-prolonging.

#### For cCTA with selective FFR<sub>CT</sub>:

Mild contrast reaction such as rash and hives.

- 1. Severe contrast reactions including anaphylaxis or death occurring within 24 hours of contrast administration.
- 2. Extravasation of contrast into the surrounding tissue of the extremity where contrast was administered intravenously.
- 3. Symptomatic bradycardia or hypotension in relation to beta blockade or nitrates administered for cCTA.
- 4. Acute bronchospasm following beta blockade administered for cCTA.

#### For Usual Care (noninvasive or invasive testing)

For exercise testing including during stress echo or stress nuclear (including PET):

- 1. Hypotension defined as systolic BP less than 80 mmHg or fall in systolic BP >20 mmHg
- 2. Stress-induced symptoms or ECG changes that do not resolve within 20 minutes
- 3. Rapid atrial fibrillation that does not slow or convert with standard interventions
- 4. Ventricular tachycardia
- 5. Hospital admission not otherwise captured by pre-specified study endpoints, due to one of the above

#### For stress nuclear (including PET):

1. Any adverse reactions potentially related to the use of vasodilators such as adenosine, regadenoson, or dipyridamole

#### For stress echo:

- 1. Any stress-induced wall motion abnormality that does not resolve within 20 minutes
- 2. Any adverse reaction to echo contrast
- 3. Any adverse reaction to dobutamine, including sustained ventricular tachycardia or other tachyarrhythmias

#### For stress cardiac MRI:

- 1. Any adverse reactions potentially related to the use of vasodilators such as adenosine, regadenoson, or dipyridamole
- 2. Any adverse reaction to MRI contrast agents, including gadolinium-based agents

#### For cardiac catheterization:

- 1. Any adverse reactions potentially related to the use of sedatives, local anesthetics, contrast agent or other medication's
- 2. Any adverse reactions potentially related to arterial puncture and wire/catheter introduction
- 3. Any adverse reaction to coronary catheterization including dissection, embolization, stroke, malignant arrhythmias and asystole, and death

#### VII.D. Independent Clinical Event Adjudication Committee

An independent clinical event committee (CEC) will be responsible for the blinded review and adjudication of the primary endpoint. The CEC will settle any disputes with committee review and discussion. Any uncertainty regarding the finding of cardiac catheterization without obstructive disease will prompt review of the original cardiac catheterization images for further independent adjudication. Collection of medical records and other documentation required for CEC reviews will be coordinated by the DCRI call center for US participants and by site coordinators for participants in all other regions.

#### VII.E. Data and Safety Monitoring Board

An independent Data and Safety Monitoring Board (DSMB) will be appointed to monitor participant safety and to review study performance. The DSMB will periodically review the study data and assess participant safety and adherence to the study protocol. The DSMB will define the operating guidelines and processes for study evaluation, interim analyses, event triggers for unscheduled review; these will be agreed upon at the initial meeting of the DSMB. Periodic reports will be prepared by HeartFlow (or its designee) for the DSMB on based on the operational plan outlined by the DSMB charter. The DSMB will make its recommendations to the study Steering Committee and the sponsor following their meeting.

#### **VIII. Statistical Methods**

Separate, complete Statistical Analysis Plan (SAP) documents will be prepared for the clinical outcome analyses and the economics and quality of life (EQOL) outcomes.

#### VIII.A. Sample Size Determination and Statistical Power

Sample size and power calculations for this study are based on the hypothesis that the precision evaluation arm is superior to the usual care arm on the time-to-first event of the composite MACE endpoint (defined as: all-cause death, non-fatal MI) or invasive cardiac catheterization without obstructive CAD (obstructive CAD defined as diameter -stenosis ≥50%, FFR≤0.80 or iFR ≤0.89). Time to event analysis will use the date of the event, including the date of catheterization which is used to determine the absence of obstructive CAD. Assuming 10% of usual care participants will receive angiography as a first test results in an 8% primary endpoint event rate at 1 year in the usual care group and 5% (absolute) event rate in the precision care group (i.e., 37.5% relative effect size) with an estimated ~20% assigned to guideline-recommended care with symptom management and no planned testing. Assumptions used in the primary endpoint event rate calculations (i.e. 8% vs. 5%) were: an overall ~10% will not receive randomized testing and within the precision evaluation arm, 30% of those assigned to guideline-recommended care will cross over to cCTA with selective FFR<sub>CT</sub>.

Enrolling 1050 patients per group (2100 total participants) would provide at least 90% power to detect a relative risk reduction of 37.5% in the precision evaluation arm. Sample size calculations are based on the log-rank test<sup>52</sup> with 12-month accrual period, a 12-month follow-up in all participants, 10% attrition rate (i.e., lost to follow- up, dropouts) and a two-sided type I error rate of 0.05.

| 1-yr event rate<br>in precision<br>evaluation arm | Power | Total<br>number of<br>participants<br>needed | Total number<br>of cath and<br>MACE<br>needed |
|---|---|---|---|
| 5% | 85% | 1792 | 173 |
| (37.5% effect | 90% | 2096 | 202 |
| size) | 95% | 2592 | 250 |

Table shows total number of participants needed for 85%, 90% and 95% power. Although, this is not an event-driven study, the table also provides total number of cath and MACE needed.

Power curves (Figure: Long-Rank for Two Survival Curves) provide total sample size needed for several relative effect size (i.e., 1-hazard ratio) scenarios.



Figure: Long-Rank for Two Survival Curves

#### VIII.B. Statistical Analysis Plan

#### Analysis of the Primary Endpoint

The primary endpoint of this study is based on time-to-first occurrence of any of the components, which is defined as a composite of MACE (all-cause death, non-fatal MI) or invasive cardiac catheterization without obstructive CAD (obstructive CAD defied as diameter stenosis ≥50%, FFR≤0.80, or iFR≤0.89) over 12-month follow-up. The time from randomization to the first event among the components of the primary endpoint will be measured (in days) for those who experienced an event and calculated as the date of the first event minus the date of randomization. For participants who do not experience any of the primary endpoint component events or who withdraw consent or drop out of the study before experiencing an event, time from randomization to the date of last contact will be used in the analysis, and those participants will be considered as censored observations in the time-to-event analysis.

The primary and secondary endpoint comparisons between the randomized groups in this study will be performed according to the principle of "intention-to-treat" (ITT); that is, participants will be analyzed according to the treatment arm to which they were randomized, regardless of subsequent crossover or post-randomization strategy.

The log-rank test<sup>53</sup> will be the primary analytic tool for statistically assessing outcome differences between the two randomized treatment strategies with respect to the primary composite endpoint. Cox proportional hazards model<sup>54</sup> will be used to estimate the hazard ratio (HR) and 95% confidence interval (CI) summarizing the difference in outcome between the two randomized arms, using treatment as the only predictor in the model. Proportionality assumption in the Cox model (i.e., constant hazard over time) will be checked and tested.

Cumulative event rates will be calculated according to the method of Kaplan and Meier<sup>55</sup> for each randomized arm as a function of time from randomization, and the estimated event probabilities

will be displayed graphically. Adjusted HR and its 95% CI will be estimated using Cox proportional hazards model by including pre-specified baseline risk factors as covariates in the model.

A sensitivity analysis for the primary composite MACE (all cause death and non-fatal MI) or invasive cardiac catheterization without CAD (no coronary stenosis  $\geq$ 50% according to QCA by core-lab adjudication or site interpretation if QCA is not available, or with FFR $\leq$ 0.80, or instantaneous wave free ratio (iFR)  $\leq$ 0.89) endpoint will be conducted using the method of "win-ratio" and Finkelstein and Schoenfeld rank-test method<sup>57</sup>. More details on primary, secondary and sensitivity analyses will be provided in the complete Statistical Analysis Plan (SAP).

#### Subgroup analyses

Subgroup analyses will be performed to assess whether the intervention effect is consistent across all participants, or whether it varies according to specific participant characteristics. In particular, these analyses will focus on whether the relative intervention effect compared to usual care differs according to the following baseline variables:

- Low risk vs. elevated risk by PROMISE Risk score or presence of known non-obstructive atherosclerosis
- Intended first test: functional vs. invasive
- Sex (male vs. female)
- Age (<65, 65 to 74, and >75 years)
- History of diabetes
- Presentation: primary symptom (chest pain vs. other), SAQ angina score (daily/weekly angina at baseline versus less frequent)
- Geographic region (US, Canada, Europe, Other Regions)

These analyses will utilize the Cox model and will be accomplished by testing for interactions between the randomized treatment strategy and the specific baseline variables listed above. In addition to the formal assessment of treatment by covariate interactions, the effect of the treatment strategy characterized by a hazard ratio and 95% confidence interval will be calculated and displayed using a forest plot for the subgroups of participants defined by the variables listed above. These descriptive hazard ratios will be carefully interpreted in conjunction with the formal interaction tests.

The effect of the treatment strategy may also be examined in other subgroups of clinical interest in addition to those listed above.

#### Analysis of the Secondary Endpoints

The secondary endpoints listed in section III.C. Secondary Endpoints that are measured as time-to-event will be analyzed using the same statistical methods used for the primary efficacy endpoint (Section VI.A. Primary Endpoint Definitions). Specifically, the log-rank test will be the primary analytic tool for statistically assessing mortality differences between the two randomized treatment strategies. A hazard ratio and 95% confidence interval summarizing the difference in outcome between the two randomized arms will be computed using the Cox model.

Participant deaths will be classified by the Clinical Events Committee (CEC) as to whether the mode of death was due to a cardiovascular (CV) cause. If insufficient source documents are obtained to allow CEC adjudication of the cause of death, and the CEC classifies the cause of

death as "unknown," then the site-reported cause of death (if available) will be used. If neither the site nor the CEC can provide a classification of the cause of death, the death will not be considered as a cardiovascular death. As supplemental analyses, however, this endpoint will also be examined using (a) only the deaths classified by the CEC as cardiovascular, and (b) using deaths classified by the CEC as cardiovascular category that are classified as unknown by the CEC.

Competing risks methodology of Fine and Gray<sup>58</sup>, where death due to a non-cardiovascular cause is considered as a competing risk. This methodology, rather than treating non-cardiovascular death as a censoring event, makes incidence use of the cumulative function, and is performed within the proportional hazards framework using the marginal failure sub-distribution associated with the event of interest (cardiovascular death). Similar analyses will be conducted for time-to- event endpoints in which death is not part of the endpoint of interest.

#### Analysis of Resource Use Endpoints

For the Economics outcomes, primary comparison will be at 12 months between treatment arms by intention-to-treat. All-cause hospitalizations, cardiovascular hospitalizations, ER visits not resulting in hospitalization, and major outpatient procedures will be enumerated. In addition, we will examine length of stay by intensity of care, numbers of CTAs, noninvasive stress tests (stress perfusion imaging, stress echocardiography, exercise electrocardiography, stress cardiac magnetic resonance imaging), invasive tests (invasive coronary angiography, invasive fractional flow reserve or equivalent, optical coherence tomography, intravascular ultrasound), coronary revascularization procedures (coronary artery bypass graft surgery (CABG), percutaneous coronary intervention (PCI), number of coronary stents), and cardiac medications (beta blockers, aspirin, statins, antiplatelet medications).

Confidence intervals for differences will be estimated using the bootstrap approach. Differences in resource use will be interpreted in the context of the trial clinical results, looking for both consistency and plausibility. Descriptive comparisons of intensity of care/resource consumption according to clinical variables defining subgroups of interest will be performed. The primary economic analyses will focus on the US enrollment and in secondary analyses, resource use patterns for all patients enrolled in the trial will be compared by intention-to-treat to develop an understanding of the degree to which treatment related differences in the trial are region dependent.

#### Analyses of Medical Costs

To compare medical costs between treatment arms, we must: 1) assign costs to all medical resources consumed during the study period; 2) compute mean costs by treatment group (defined by the principle of intention-to-treat); and 3) calculate the difference in mean costs between treatment arms and generate confidence intervals.

#### A) Derivation of Cost Estimates

The cost of US hospital-based care will be estimated by applying hospital-specific, revenue center level cost-to-charge ratios to empirical billing data collected during the study. This approach, which has been used successfully in numerous previous clinical trials including the PROMISE trial takes advantage of the objective, detailed account in hospital bills of services provided to patients and recalibrates hospital charges to more closely reflect costs. Based on experience in similar studies, we anticipate having complete billing data for 95% of patients treated in hospitals that generate bills. For patients without billing data (including patients outside US), we will impute costs using a generalized linear model developed using study data. In this model, the dependent variable will be

defined as total cost, and independent variables will include resource use elements available in the case report form, such as:

Number of hospitalized nights by intensity of care and number of relevant high cost procedures. Coefficients for model parameters will be estimated using study data of patients with complete costs and then used to predict costs for patients without billing information.

The cost of stays at non-acute care facilities will be estimated by multiplying the length of stay by the corresponding per-diem/reimbursement rate.

Costs for physician services will be estimated by mapping major inpatient and outpatient procedures and services recorded on the case report form to appropriate CPT codes in the Medicare Fee Schedule. We will also assign rounding fees for inpatient stays based on type of unit.

Costs for diagnostic testing procedures done in an outpatient or standalone facility will be derived from secondary sources available to the DCRI Outcomes Group at the time of study analysis.

The cost of medications of interest/relevance will be estimated on the basis of medication use recorded in the eCRF and unit costs by medication type and class, based on current estimates of acquisition cost.

#### B) Cost Comparisons

Primary statistical comparisons of costs between the two treatment groups will be performed using the intention-to-treat principle. A nonparametric partitioned estimator will be used to estimate diagnostic strategy-specific, 1-year medical costs with 4 partitions corresponding to follow-up intervals following randomization. Comparisons between the two testing strategies will be made using a normal approximation with standard errors estimated using the bootstrap approach. Bootstrapping will be performed using 10,000 repetitions, with percentile-based confidence intervals reported. The primary cost comparison will be made for cumulative costs at 12 months. The primary effect size will be the mean cost difference between the two arms with 95% confidence intervals. P values will be calculated for selective comparisons, with a "significant" p value equivalent to a 95% confidence interval that excludes 0. No adjustment in significance levels for multiple comparisons will be used.

Differences in cost will be interpreted in the context of the trial clinical results, looking for both consistency and plausibility. Costs will be presented both overall and by category (e.g., inpatient hospitalization, outpatient procedures, concomitant medications, non-acute institutional care). Hospitalizations will be classified as cardiovascular or non-cardiovascular by the Clinical Events Committee. For illustrative purposes, we will use bootstrap methods to plot the probability of a difference in total costs greater than arbitrary thresholds of interest (such as \$500, \$750, or \$1000).

#### C) Cost Sensitivity Analyses

In secondary sensitivity analyses, we will compare resource use and costs between treatment groups in the US. In this manner, the effect of overall patterns of resource use in the US cohort versus ex-US on cost differences by treatment group can be assessed. We will also perform a per protocol analysis of costs.

#### Analyses of Quality of Life Outcomes

For each of the QOL measures examined in this study, we will provide simple descriptive and comparative analyses by intention-to-treat. To address the multiple comparisons problem arising from testing each individual scale and time point separately, we propose two complementary approaches. First, we will pre-specify the angina frequency scale from the SAQ as the primary QOL comparison of interest and assign all other comparisons to a secondary (supportive) status.

Second, we will use a repeated-measures mixed model with the baseline score as a covariate, Day 45, Month 6, and Month 12 responses included as outcome variables, and time as a fixed variable. Restricted maximum likelihood estimation will be used to model all available data from each participant without imputing missing values. An unstructured covariance matrix will be used.

Point estimates for each diagnostic strategy arm and strategy arm mean differences (precision strategy – usual care) with 95% confidence intervals (CIs) will be generated for each time point. The primary assessment will be based on the strategy arm difference at Month 12.

Additionally the intervention effect at the other contact time points.

Additionally, the intervention effect will be averaged across all the follow-up time points. The estimated intervention difference and 95% CIs will be obtained using the ESTIMATE Statement in SAS PROC MIXED.

We expect to have analyzable data on ≥95% of survivors at each follow-up interview, and, with 90%+ data collection (945+ patients per treatment group), consistent with our past performance in trials of this size and complexity and using similar methods, even accounting for loss of data due to death or incapacity, we should have 90% or greater statistical power to detect clinically significant differences in our major QOL measures.

Major QOL subgroups to be examined will be those prespecified for the clinical analysis of this trial. In addition, we will use baseline angina frequency from the SAQ to create a subgroup of participants with daily or weekly chest pain versus those with less frequent symptoms.

#### IX. ETHICAL CONSIDERATIONS AND RISK ANALYSIS

#### IX.A. Ethical Considerations

PRECISE will be conducted in accordance with the recommendations for human research from the 18<sup>th</sup> World Medical Assembly, Helsinki 1964. All potential sites will obtain Institutional Review Board (IRB) or Ethics Committee (EC) approval of the protocol, the associated consent form and any participant facing recruitment tools. Written informed consent will be obtained from each patient before any study procedures are performed. Patients will have the option to consent for the study after receiving a full explanation of the risks, benefits, and available diagnostic options, with the right to refuse participation. Clinicians will have the option to pursue alternative diagnostic pathways if they deem it to be in the best interest of the patient, with the reason for study protocol deviation documented. Participants can withdraw from the study at any time.

#### IX.B. Study Risks and Benefits

#### Potential Risks

Participation in PRECISE does not present any extra risks other than the risks associated with the clinically indicated care recommended by the participant's treating physicians to evaluate and treat symptoms suggestive of CAD. As all approaches included in the trial are recognized as standard of care, the risk associated with the trial can be described in detail by the treating physician.

Noninvasive diagnostic imaging is generally considered a safe and effective diagnostic approach. FFR<sub>CT</sub> does not pose any additional risk to participants beyond the performance of cCTA itself. It

does offer the potential benefit to participants of the recognition of hemodynamically significant lesions (FFR  $\leq$ 0.80 or iFR  $\leq$ 0.89) that may not demonstrate anatomic significance (<50% diameter stenosis) and avoidance of unnecessary revascularization of  $\geq$ 50% lesions that are not hemodynamically significant (FFR>0.80 or iFR >0.89).

The risks of guideline-recommended care without planned testing in the lowest risk participants has not been extensively studied prospectively. However, validation of the PROMISE Risk Tool in SCOT-HEART indicate that participants in this risk category have a CV death/MI event rate <1%/year, similar to the event rate observed in an age and sex matched US population. While the risk of guideline-recommended care without planned testing in the precision evaluation arm has not been quantified prospectively it is not expected to differ from the excellent outcomes noted above in such patients who do undergo testing. Further, participants with continued symptoms not controlled by medications will be permitted to cross over to the precision strategy arm and receive, cCTA with selective FFR<sub>CT</sub>.

#### Potential Loss of Confidentiality

In any clinical trial, there is a possible risk of loss of confidentiality. To prevent this from occurring, HeartFlow has strict procedures in place to ensure that all study data are confidential and anonymized except as required for centralized follow-up data collection for the US, which will be performed by the DCRI Outcomes Call Center. For all data transferred from enrolling sites or from the Call Center, participants will be identified only by unique patient identifiers. Data transmitted will not contain any protected health information and participants will be identified only by unique patient identifiers. Data transmitted will not contain any protected health information. All applicable study data will be transferred in a secure manner and in accordance with applicable regulations.

#### Potential Benefits

The PRECISE results should improve the care of future patients recommended for additional evaluation for suspected significant CAD. In addition, the trial will deliver high-quality data on radiation exposure, incidental findings, and other clinically important "side effects" of the evaluation and management strategies that will be examined in a large real-world experience. All participants may benefit from increased contact with health care providers due to study-required visits.

## X. DATA HANDLING AND QUALITY ASSURANCE

#### X.A. Completing and Signing Case Report Forms

Electronic CRFs will be employed. Trained site personnel or the trained DCRI Outcomes Group will enter data into the eCRFs. Data changes and corrections should be done within the electronic system. The audit trail will record all changes made, the date and time of the correction, the person making the change and a reason for the change. The appropriate electronic signature will be provided by the investigator as indicated.

#### X.B. Clinical Data Management

The sponsor or its designees will be responsible for the handling, processing, and quality control of the data in compliance with all applicable regulatory guidelines.

The training of clinical site personnel and the DCRI Outcomes Group on eCRF completion will be the responsibility of the sponsor or its designees. To ensure uniform data collection, a Case Report Form Guide will be created to assist with eCRF completion. All clinical site research coordinators will undergo site initiation training to become thoroughly familiar with the protocol, case report forms, and with methods of data verification.

#### X.C. Archiving of Data

All study documentation at the investigator site and sponsor site will be archived in accordance with ICH GCP. It is HeartFlow's policy to retain the data collected in this clinical study for a minimum of 5 years after termination of the study. Clinical sites will be asked to retain the data for at least 2 years following completion of the study or longer as required by local laws.

### XI. STUDY MONITORING, AUDITING, AND INSPECTING

HeartFlow or its designees will monitor this clinical study to check the adequacy of clinical site staff and facilities, and to ensure adherence to the protocol, study procedures, and applicable regulations. In accordance with ICH E6 GCP guidelines, the clinical site monitor will also assess proper eCRF completion and source document retention. The investigator and clinical site staff are expected to provide adequate space for monitoring visits and to allocate sufficient time to permit adequate review of the study's progress. The investigator will permit study-related monitoring, audits, IRB review, and regulatory inspection(s), providing direct access to source data/documents and study-related facilities (e.g., pharmacy, diagnostic testing and laboratories).

#### XI.A. Study Monitoring

Study monitoring will be performed in accordance with ICH E6GCP, this protocol, and applicable local regulations. A Clinical Monitoring Plan will be written at the outset of the study to provide project-specific operational guidelines for the clinical monitoring process and procedures, define responsibilities of the Site Management/Monitoring Team, which will in turn ensure the quality and integrity of data collected.

#### XI.B. Auditing and Inspecting

HeartFlow quality assurance personnel and/or their designee(s) may conduct audits at the study site(s). Audits may include, but not be limited to: audit trail of data handling and processes, SOPs, presence of required documents, the informed consent process, and comparison of case report forms/database with source documents. The investigator agrees to accommodate and participate in audits conducted at a reasonable time in a reasonable manner, as needed.

#### XII. References

- Benjamin EJ, Virani SS, Callaway CW, Chamberlain AM, Chang AR, Cheng S, Chiuve SE, Cushman M, Delling FN, Deo R, de Ferranti SD, Ferguson JF, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Lutsey PL, Mackey JS, Matchar DB, Matsushita K, Mussolino ME, Nasir K, O'Flaherty M, Palaniappan LP, Pandey A, Pandey DK, Reeves MJ, Ritchey MD, Rodriguez CJ, Roth GA, Rosamond WD, Sampson UKA, Satou GM, Shah SH, Spartano NL, Tirschwell DL, Tsao CW, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS and Muntner P. Heart Disease and Stroke Statistics-2018 Update: A Report From the American Heart Association. Circulation. 2018;137:e67-e492.
- 2. World Health Organization. Cardiovascular diseases (CVDs).(Fact-sheet) 2017.
- 3. Fordyce CB and Douglas PS. Optimal non-invasive imaging test selection for the diagnosis of ischaemic heart disease. *Heart (British Cardiac Society)*. 2016;102:555-64.
- 4. Newby D, et al. CT coronary angiography in patients with suspected angina due to coronary heart disease (SCOT-HEART): an open-label, parallel-group, multicentre trial. *Lancet* (*London, England*). 2015;385:2383-91.
- 5. Douglas PS, Hoffmann U, Patel MR, Mark DB, Al-Khalidi HR, Cavanaugh B, Cole J, Dolor RJ, Fordyce CB, Huang M, Khan MA, Kosinski AS, Krucoff MW, Malhotra V, Picard MH, Udelson JE, Velazquez EJ, Yow E, Cooper LS and Lee KL. Outcomes of anatomical versus functional testing for coronary artery disease. *N Engl J Med*. 2015;372:1291-300.
- 6. Patel MR, Peterson ED, Dai D, Brennan JM, Redberg RF, Anderson HV, Brindis RG and Douglas PS. Low diagnostic yield of elective coronary angiography. *N Engl J Med*. 2010;362:886-95.
- 7. Douglas PS, De Bruyne B, Pontone G, Patel MR, Norgaard BL, Byrne RA, Curzen N, Purcell I, Gutberlet M, Rioufol G, Hink U, Schuchlenz HW, Feuchtner G, Gilard M, Andreini D, Jensen JM, Hadamitzky M, Chiswell K, Cyr D, Wilk A, Wang F, Rogers C and Hlatky MA. 1-Year Outcomes of FFR<sub>CT</sub>-Guided Care in Patients With Suspected Coronary Disease: The PLATFORM Study. *Journal of the American College of Cardiology*. 2016;68:435-445.
- 8. Fordyce CB, Newby DE and Douglas PS. Diagnostic Strategies for the Evaluation of Chest Pain: Clinical Implications From SCOT-HEART and PROMISE. *Journal of the American College of Cardiology*. 2016;67:843-52.
- 9. Williams MC, Moss A, Nicol E and Newby DE. Cardiac CT Improves Outcomes in Stable Coronary Heart Disease: Results of Recent Clinical Trials. *Curr Cardiovasc Imaging Rep.* 2017;10:14.
- Ladapo JA, Hoffmann U, Lee KL, Coles A, Huang M, Mark DB, Dolor RJ, Pelberg RA, Budoff M, Sigurdsson G, Severance HW and Douglas PS. Changes in Medical Therapy and Lifestyle After Anatomical or Functional Testing for Coronary Artery Disease. *Journal of the American Heart Association*. 2016;5.

- 11. Schulman-Marcus J, Lin FY, Gransar H, Berman D, Callister T, DeLago A, Hadamitzky M, Hausleiter J, Al-Mallah M, Budoff M, Kaufmann P, Achenbach S, Raff G, Chinnaiyan K, Cademartiri F, Maffei E, Villines T, Kim Y-J, Leipsic J, Feuchtner G, Rubinshtein R, Pontone G, Andreini D, Marques H, Chang H-J, Chow BJW, Cury RC, Dunning A, Shaw L and Min JK. Coronary revascularization vs. medical therapy following coronary-computed tomographic angiography in patients with low-, intermediate- and high-risk coronary artery disease: results from the CONFIRM long-term registry. *European heart journal cardiovascular Imaging*. 2017;18:841-848.
- 12. Chow BJ, Small G, Yam Y, Chen L, McPherson R, Achenbach S, Al-Mallah M, Berman DS, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Cheng VY, Chinnaiyan K, Cury R, Delago A, Dunning A, Feuchtner G, Hadamitzky M, Hausleiter J, Karlsberg RP, Kaufmann PA, Kim YJ, Leipsic J, LaBounty T, Lin F, Maffei E, Raff GL, Shaw LJ, Villines TC and Min JK. Prognostic and therapeutic implications of statin and aspirin therapy in individuals with nonobstructive coronary artery disease: results from the CONFIRM (COronary CT Angiography Evaluation For Clinical Outcomes: An InteRnational Multicenter registry) registry. Arteriosclerosis, thrombosis, and vascular biology. 2015;35:981-9.
- 13. Schulman-Marcus J, Hartaigh BO, Giambrone AE, Gransar H, Valenti V, Berman DS, Budoff MJ, Achenbach S, Al-Mallah M, Andreini D, Cademartiri F, Callister TQ, Chang HJ, Chinnaiyan K, Chow BJ, Cury R, Delago A, Hadamitzky M, Hausleiter J, Feuchtner G, Kim YJ, Kaufmann PA, Leipsic J, Lin FY, Maffei E, Pontone G, Raff G, Shaw LJ, Villines TC, Dunning A and Min JK. Effects of cardiac medications for patients with obstructive coronary artery disease by coronary computed tomographic angiography: results from the multicenter CONFIRM registry. Atherosclerosis. 2015;238:119-25.
- 14. Hoffmann U, Ferencik M, Udelson JE, Picard MH, Truong QA, Patel MR, Huang M, Pencina M, Mark DB, Heitner JF, Fordyce CB, Pellikka PA, Tardif JC, Budoff M, Nahhas G, Chow B, Kosinski AS, Lee KL and Douglas PS. Prognostic Value of Noninvasive Cardiovascular Testing in Patients With Stable Chest Pain: Insights From the PROMISE Trial (Prospective Multicenter Imaging Study for Evaluation of Chest Pain). Circulation. 2017;135:2320-2332.
- 15. Ferencik M, Mayrhofer T, Bittner DO, Emami H, Puchner SB, Lu MT, Meyersohn NM, Ivanov AV, Adami EC, Patel MR, Mark DB, Udelson JE, Lee KL, Douglas PS and Hoffmann U. Use of High-Risk Coronary Atherosclerotic Plaque Detection for Risk Stratification of Patients With Stable Chest Pain: A Secondary Analysis of the PROMISE Randomized Clinical Trial. *JAMA Cardiol.* 2018;3:144-152.
- 16. Shaw LJ, Hausleiter J, Achenbach S, Al-Mallah M, Berman DS, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Kim YJ, Cheng VY, Chow BJ, Cury RC, Delago AJ, Dunning AL, Feuchtner GM, Hadamitzky M, Karlsberg RP, Kaufmann PA, Leipsic J, Lin FY, Chinnaiyan KM, Maffei E, Raff GL, Villines TC, Labounty T, Gomez MJ and Min JK. Coronarycomputed tomographic angiography as a gatekeeper to invasive diagnostic and surgical procedures: results from the multicenter CONFIRM (Coronary CT Angiography Evaluation for Clinical Outcomes: an International Multicenter) registry. Journal of the American College of Cardiology. 2012;60:2103-14.
- 17. Foy AJ, Dhruva SS, Peterson B, Mandrola JM, Morgan DJ and Redberg RF. Coronary Computed Tomography Angiography vs Functional Stress Testing for Patients With Suspected Coronary Artery Disease: A Systematic Review and Meta-analysis. *JAMA internal medicine*. 2017;177:1623-1631.

- 18. Norgaard BL, Leipsic J, Gaur S, Seneviratne S, Ko BS, Ito H, Jensen JM, Mauri L, De Bruyne B, Bezerra H, Osawa K, Marwan M, Naber C, Erglis A, Park SJ, Christiansen EH, Kaltoft A, Lassen JF, Botker HE and Achenbach S. Diagnostic performance of noninvasive fractional flow reserve derived from coronary computed tomography angiography in suspected coronary artery disease: the NXT trial (Analysis of Coronary Blood Flow Using CT Angiography: Next Steps). *Journal of the American College of Cardiology*. 2014;63:1145-1155.
- 19. Koo BK, Erglis A, Doh JH, Daniels DV, Jegere S, Kim HS, Dunning A, DeFrance T, Lansky A, Leipsic J and Min JK. Diagnosis of ischemia-causing coronary stenoses by noninvasive fractional flow reserve computed from coronary computed tomographic angiograms. Results from the prospective multicenter DISCOVER-FLOW (Diagnosis of Ischemia-Causing Stenoses Obtained Via Noninvasive Fractional Flow Reserve) study. *Journal of the American College of Cardiology*. 2011;58:1989-97.
- 20. Min JK, Leipsic J, Pencina MJ, Berman DS, Koo BK, van Mieghem C, Erglis A, Lin FY, Dunning AM, Apruzzese P, Budoff MJ, Cole JH, Jaffer FA, Leon MB, Malpeso J, Mancini GB, Park SJ, Schwartz RS, Shaw LJ and Mauri L. Diagnostic accuracy of fractional flow reserve from anatomic CT angiography. *JAMA*: the journal of the American Medical Association. 2012;308:1237-45.
- 21. Min JK, Taylor CA, Achenbach S, Koo BK, Leipsic J, Norgaard BL, Pijls NJ and De Bruyne B. Noninvasive Fractional Flow Reserve Derived From Coronary CT Angiography: Clinical Data and Scientific Principles. *JACC Cardiovascular imaging*. 2015;8:1209-22.
- 22. Taylor CA, Fonte TA and Min JK. Computational fluid dynamics applied to cardiac computed tomography for noninvasive quantification of fractional flow reserve: scientific basis. *Journal of the American College of Cardiology*. 2013;61:2233-41.
- 23. Lu MT, Ferencik M, Roberts RS, Lee KL, Ivanov A, Adami E, Mark DB, Jaffer FA, Leipsic JA, Douglas PS and Hoffmann U. Noninvasive FFR Derived From Coronary CT Angiography: Management and Outcomes in the PROMISE Trial. *JACC Cardiovascular imaging*. 2017;10:1350-1358.
- 24. De Bruyne B, Fearon WF, Pijls NH, Barbato E, Tonino P, Piroth Z, Jagic N, Mobius-Winckler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd K, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Limacher A, Nuesch E and Juni P. Fractional flow reserve-guided PCI for stable coronary artery disease. *N Engl J Med*. 2014;371:1208-17.
- 25. De Bruyne B, Pijls NH, Kalesan B, Barbato E, Tonino PA, Piroth Z, Jagic N, Mobius-Winkler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd KG, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Juni P and Fearon WF. Fractional flow reserve-guided PCI versus medical therapy in stable coronary disease. *N Engl J Med*. 2012;367:991-1001.
- 26. National Clinical Guideline Centre for A and Chronic C. Chest Pain of Recent Onset: Assessment and Diagnosis of Recent Onset Chest Pain or Discomfort of Suspected Cardiac Origin: NICE (National Institute for Health and Care Excellence); 2010.

- 27. Moss AJ, Williams MC, Newby DE and Nicol ED. The Updated NICE Guidelines: Cardiac CT as the First-Line Test for Coronary Artery Disease. *Curr Cardiovasc Imaging Rep.* 2017;10:15.
- 28. Services DoHaH. Medicare program: Hospital Outpatient Prospective Payment and Ambulatory Surgical Center Payment Systems and Quality Reporting Programs. *42 CFR Parts 414, 416 and 419.* December 14, 2017;82:282.
- 29. Boden WE, O'Rourke RA, Teo KK, Hartigan PM, Maron DJ, Kostuk WJ, Knudtson M, Dada M, Casperson P, Harris CL, Chaitman BR, Shaw L, Gosselin G, Nawaz S, Title LM, Gau G, Blaustein AS, Booth DC, Bates ER, Spertus JA, Berman DS, Mancini GB and Weintraub WS. Optimal medical therapy with or without PCI for stable coronary disease. *N Engl J Med*. 2007;356:1503-16.
- 30. Al-Lamee R, Thompson D, Dehbi HM, Sen S, Tang K, Davies J, Keeble T, Mielewczik M, Kaprielian R, Malik IS, Nijjer SS, Petraco R, Cook C, Ahmad Y, Howard J, Baker C, Sharp A, Gerber R, Talwar S, Assomull R, Mayet J, Wensel R, Collier D, Shun-Shin M, Thom SA, Davies JE and Francis DP. Percutaneous coronary intervention in stable angina (ORBITA): a double-blind, randomised controlled trial. *Lancet (London, England)*. 2018;391:31-40.
- 31. Genders TS, Steyerberg EW, Alkadhi H, Leschka S, Desbiolles L, Nieman K, Galema TW, Meijboom WB, Mollet NR, de Feyter PJ, Cademartiri F, Maffei E, Dewey M, Zimmermann E, Laule M, Pugliese F, Barbagallo R, Sinitsyn V, Bogaert J, Goetschalckx K, Schoepf UJ, Rowe GW, Schuijf JD, Bax JJ, de Graaf FR, Knuuti J, Kajander S, van Mieghem CA, Meijs MF, Cramer MJ, Gopalan D, Feuchtner G, Friedrich G, Krestin GP and Hunink MG. A clinical prediction rule for the diagnosis of coronary artery disease: validation, updating, and extension. *Eur Heart J*. 2011;32:1316-30.
- 32. Hadamitzky M, Achenbach S, Al-Mallah M, Berman D, Budoff M, Cademartiri F, Callister T, Chang HJ, Cheng V, Chinnaiyan K, Chow BJ, Cury R, Delago A, Dunning A, Feuchtner G, Gomez M, Kaufmann P, Kim YJ, Leipsic J, Lin FY, Maffei E, Min JK, Raff G, Shaw LJ, Villines TC and Hausleiter J. Optimized prognostic score for coronary computed tomographic angiography: results from the CONFIRM registry (COronary CT Angiography Evaluation For Clinical Outcomes: An InteRnational Multicenter Registry). Journal of the American College of Cardiology. 2013;62:468-76.
- 33. Adamson PD, Fordyce CB, McAllister DA, Udelson JE, Douglas PS and Newby DE. Identification of patients with stable chest pain deriving minimal value from coronary computed tomography angiography: An external validation of the PROMISE minimal-risk tool. *International journal of cardiology*. 2018;252:31-34.
- 34. Fordyce CB, Douglas PS, Roberts RS, Hoffmann U, Al-Khalidi HR, Patel MR, Granger CB, Kostis J, Mark DB, Lee KL and Udelson JE. Identification of Patients With Stable Chest Pain Deriving Minimal Value From Noninvasive Testing: The PROMISE Minimal-Risk Tool, A Secondary Analysis of a Randomized Clinical Trial. *JAMA Cardiol*. 2017;2:400-408.
- 35. Douglas PS, Pontone G, Hlatky MA, Patel MR, Norgaard BL, Byrne RA, Curzen N, Purcell I, Gutberlet M, Rioufol G, Hink U, Schuchlenz HW, Feuchtner G, Gilard M, Andreini D, Jensen JM, Hadamitzky M, Chiswell K, Cyr D, Wilk A, Wang F, Rogers C and De Bruyne B. Clinical outcomes of fractional flow reserve by computed tomographic angiography-guided diagnostic strategies vs. usual care in patients with suspected coronary artery disease: the

- prospective longitudinal trial of FFR(CT): outcome and resource impacts study. *Eur Heart J*. 2015;36:3359-67.
- 36. Fordyce CB and Douglas PS. Outcomes-Based CV Imaging Research Endpoints and Trial Design: From Pixels to Patient Satisfaction. *JACC Cardiovascular imaging*. 2017;10:253-263.
- 37. Fihn SD, Gardin JM, Abrams J, Berra K, Blankenship JC, Dallas AP, Douglas PS, Foody JM, Gerber TC, Hinderliter AL, King SB, 3rd, Kligfield PD, Krumholz HM, Kwong RY, Lim MJ, Linderbaum JA, Mack MJ, Munger MA, Prager RL, Sabik JF, Shaw LJ, Sikkema JD, Smith CR. Jr., Smith SC. Jr., Spertus JA and Williams SV. ACCF/AHA/ACP/AATS/PCNA/SCAI/STS Guideline for the diagnosis and management of patients with stable ischemic heart disease: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines, and the American College of Physicians, American Association for Thoracic Surgery, Preventive Cardiovascular Nurses Association, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. Journal of the American College of Cardiology. 2012;60:e44-e164.
- 38. Bradley SM, Spertus JA, Kennedy KF, Nallamothu BK, Chan PS, Patel MR, Bryson CL, Malenka DJ and Rumsfeld JS. Patient selection for diagnostic coronary angiography and hospital-level percutaneous coronary intervention appropriateness: insights from the National Cardiovascular Data Registry. *JAMA internal medicine*. 2014;174:1630-9.
- 39. Lin GA, Dudley RA, Lucas FL, Malenka DJ, Vittinghoff E and Redberg RF. Frequency of stress testing to document ischemia prior to elective percutaneous coronary intervention. *JAMA : the journal of the American Medical Association*. 2008;300:1765-73.
- 40. Patel MR, Dai D, Hernandez AF, Douglas PS, Messenger J, Garratt KN, Maddox TM, Peterson ED and Roe MT. Prevalence and predictors of nonobstructive coronary artery disease identified with coronary angiography in contemporary clinical practice. *American heart journal*. 2014;167:846-52.e2.
- 41. Colleran R, Douglas PS, Hadamitzky M, Gutberlet M, Lehmkuhl L, Foldyna B, Woinke M, Hink U, Nadjiri J, Wilk A, Wang F, Pontone G, Hlatky MA, Rogers C and Byrne RA. An FFRCT diagnostic strategy versus usual care in patients with suspected coronary artery disease planned for invasive coronary angiography at German sites: one-year results of a subgroup analysis of the PLATFORM (Prospective Longitudinal Trial of FFR<sub>CT</sub>: Outcome and Resource Impacts) study. *Open heart*. 2017;4:e000526.
- 42. Gibbons RJ, Balady GJ, Bricker JT, Chaitman BR, Fletcher GF, Froelicher VF, Mark DB, McCallister BD, Mooss AN, O'Reilly MG, Winters WL, Gibbons RJ, Antman EM, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Hiratzka LF, Jacobs AK, Russell RO and Smith SC. ACC/AHA 2002 guideline update for exercise testing: summary article. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Update the 1997 Exercise Testing Guidelines). Journal of the American College of Cardiology. 2002;40:1531-40.
- 43. Pellikka PA, Nagueh SF, Elhendy AA, Kuehl CA and Sawada SG. American Society of Echocardiography Recommendations for Performance, Interpretation, and Application of

- Stress Echocardiography. *Journal of the American Society of Echocardiography*. 2007;20:1021-1041.
- 44. Tilkemeier PL, Bourque J, Doukky R, Sanghani R and Weinberg RL. ASNC imaging guidelines for nuclear cardiology procedures. *Journal of Nuclear Cardiology*. 2017;24:2064-2128.
- 45. Henzlova MJ, Duvall WL, Einstein AJ, Travin MI and Verberne HJ. ASNC imaging guidelines for SPECT nuclear cardiology procedures: Stress, protocols, and tracers. *Journal of nuclear cardiology : official publication of the American Society of Nuclear Cardiology*. 2016;23:606-39.
- 46. Henzlova MJ, Duvall WL, Einstein AJ, Travin MI and Verberne HJ. Erratum to: ASNC imaging guidelines for SPECT nuclear cardiology procedures: Stress, protocols, and tracers. *Journal of nuclear cardiology: official publication of the American Society of Nuclear Cardiology.* 2016;23:640-642.
- 47. Dilsizian V, Bacharach SL, Beanlands RS, Bergmann SR, Delbeke D, Dorbala S, Gropler RJ, Knuuti J, Schelbert HR and Travin MI. ASNC imaging guidelines/SNMMI procedure standard for positron emission tomography (PET) nuclear cardiology procedures. *Journal of nuclear cardiology : official publication of the American Society of Nuclear Cardiology*. 2016;23:1187-1226.
- 48. Hundley WG, Bluemke DA, Finn JP, Flamm SD, Fogel MA, Friedrich MG, Ho VB, Jerosch-Herold M, Kramer CM, Manning WJ, Patel M, Pohost GM, Stillman AE, White RD and Woodard PK. ACCF/ACR/AHA/NASCI/SCMR 2010 expert consensus document on cardiovascular magnetic resonance: a report of the American College of Cardiology Foundation Task Force on Expert Consensus Documents. *Circulation*. 2010;121:2462-508.
- 49. Leipsic J, Abbara S, Achenbach S, Cury R, Earls JP, Mancini GJ, Nieman K, Pontone G and Raff GL. SCCT guidelines for the interpretation and reporting of coronary CT angiography: a report of the Society of Cardiovascular Computed Tomography Guidelines Committee. *Journal of cardiovascular computed tomography*. 2014;8:342-58.
- 50. Abbara S, Blanke P, Maroules CD, Cheezum M, Choi AD, Han BK, Marwan M, Naoum C, Norgaard BL, Rubinshtein R, Schoenhagen P, Villines T and Leipsic J. SCCT guidelines for the performance and acquisition of coronary computed tomographic angiography: A report of the society of Cardiovascular Computed Tomography Guidelines Committee: Endorsed by the North American Society for Cardiovascular Imaging (NASCI). *Journal of cardiovascular computed tomography*. 2016;10:435-449.
- 51. Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). J Am Coll Cardiol. 2018 Oct 30;72(18):2231-2264. doi: 10.1016/j.jacc.2018.08.1038. Epub 2018 Aug 25.
- 52. Collet D. Modeling survival data in medical research (2nd edition). London: Chapman & Hall; 2003.

- 53. Kalbfleisch JD, Prentice RL. The Statistical Analysis of Failure Time Data. 2nd edition. 2002, John Wiley & Sons, Inc. Hoboken, New Jersey.
- 54. Cox DR. Regression Models and Life-Tables. *Journal of the Royal Statistical Society Series B (Methodological)*. 1972;34:187-220.
- 55. Kaplan EL and Meier P. Nonparametric Estimation from Incomplete Observations. *Journal of the American Statistical Association*. 1958;53:457-481.
- 56. Pocock SJ, Ariti CA, Collier TJ and Wang D. The win ratio: a new approach to the analysis of composite endpoints in clinical trials based on clinical priorities. *Eur Heart J.* 2012;33:176-82.
- 57. Finkelstein DM and Schoenfeld, DA. Combining mortality and longitudinal measures in clinical trials. *Statistics in Medicine*. 1999;18:1341-1354.
- 58. Fine JP and Gray RJ. A Proportional Hazards Model for the Subdistribution of a Competing Risk. *Journal of the American Statistical Association*. 1999;94:496-509.
- 59. Newby, D. E.; Adamson, P. D.; Berry, C.; Boon, N. A.; Dweck, M. R.; Flather, M.; Forbes, J.; Hunter, A.; Lewis, S.; MacLean, S.; Mills, N. L.; Norrie, J.; Roditi, G.; Shah, A. S. V.; Timmis, A. D.; van Beek, E. J. R.; Williams, M. C., Coronary CT Angiography and 5-Year Risk of Myocardial Infarction. *N Engl J Med* **2018**, 379 (10), 924-933.

## **Summary of Protocol Amendments**

## Amendment from version 1.0 dated June 29, 2018 to version 1.1 dated July 31, 2018

| Section | Version 1.0 | Version 1.1 |
|---|---|---|
| Table of Contents | Sections listed | Sections listing updated based on the changes |
| I. Study Synopsis Secondary Effectiveness Endpoints | #2. Resource use patterns (all patients) and medical costs (US patients) to 12 months | #2. Resource use patterns and medical costs |
| V. STUDY PROCEDURES V.A. Patient Screening for Eligibility (Exclusion Criteria) | #3. Noninvasive CV testing within 1 year (for suspected CAD) | #3. Noninvasive CV testing within 1 year (for suspected CAD), including coronary artery calcium score |
| V. STUDY PROCEDURES V.D. Participant Follow-Up (D45) | 45 (+/-14) day follow-up visit (in-<br>person) | 45 (+/-14) day follow-up visit<br>(in-person, portions may be<br>done by phone) |
| V. STUDY<br>PROCEDURES | Review and documentation of concomitant medication changes since enrollment | Review and documentation of concomitant cardiovascular medication changes since |
| V.D. Participant<br>Follow-Up (D45, 6M<br>and 12M) | | enrollment |
| V. STUDY<br>PROCEDURES | NA | Collection of the following: |
| V.D. Participant<br>Follow-Up (24M) | | test output Any cardiovascular imaging – both written report and image file |
| V.I. ADDITIONAL<br>ASSESSMENTS AND<br>SUBSTUDIES | Quality of life (QoL) assessments will be conducted at baseline, 45 days, 6 months and 12 months. | Quality of life (QoL) assessments will be conducted at baseline, 45 days, 6 months, 12 months, and 24 months. |
| V.I.A. Quality of Life<br>Assessments | | |
| VIII.B. Statistical Analysis Plan C) Cost Sensitivity Analyses | In secondary sensitivity analyses, we will apply US unit costs to all resource use of all patients and compare costs between treatment groups across all patients enrolled in the trial. | In secondary sensitivity analyses, we will compare resource use and costs between treatment groups in the US. |
| XII. REFERENCES | References listed | References updated via<br>EndNote |

## Amendment from version 1.1 dated July 31, 2018 to version 1.2 dated September 10, 2018

| Section | Version 1.1 | Version 1.2 |
|---|---|---|
| Table of Contents | V.E. Cross Over Participants | V.E. Testing in precision evaluation arm for participants assigned to no immediate testing |
| I. Study<br>Synopsis –<br>Study Design<br>and Methods | All subsequent decisions in the usual care arm regarding additional testing, medications, and/or procedures will be at the discretion of the responsible clinical care team; the use of cCTA as the initial diagnostic strategy is not allowed in the usual care arm. | All subsequent decisions in the usual care arm regarding additional testing, medications, and/or procedures will be at the discretion of the responsible clinical care team; the use of cCTA as the initial diagnostic strategy is not allowed in the usual care arm and prohibited as a subsequent test for the first 45 days after randomization. |
| | Usual Care: For participants randomized to usual care, the participant's care team will select the specific noninvasive stress test (exercise electrocardiogram, stress nuclear imaging [including PET], stress MR, or stress echocardiogram); OR invasive test: (direct to diagnostic catheterization). The use of cCTA as the initial diagnostic strategy is explicitly excluded in this arm. | Usual Care: For participants randomized to usual care, the participant's care team will select the specific noninvasive stress test (exercise electrocardiogram, stress nuclear imaging [including PET], stress MR, or stress echocardiogram); OR invasive test: (direct to diagnostic catheterization). The use of cCTA as the initial diagnostic strategy is explicitly excluded in this arm and prohibited as a subsequent test for the first 45 days after randomization. |
| I. Study Synopsis -<br>Sample Size<br>Considerations | Assumed rates are based on 30% assigned to guideline- recommended care with symptom management and no planned testing (within which 30% will cross over to cCTA with selective FFR <sub>CT</sub> ); and overall 10% will not receive assigned testing; enrolling 1050 participants per group (2100 total participants) would provide at least 90% power to demonstrate superiority accounting for 10% attrition rate. | Assumed rates are based on 20% assigned to guideline-recommended care with symptom management and no planned testing (within which 30% will cross over to cCTA with selective FFR <sub>CT</sub> ); and overall 10% will not receive assigned testing; enrolling 1050 participants per group (2100 total participants) would provide at least 90% power to demonstrate superiority accounting for 10% attrition rate. |

| III.A. Prior Literature and Studies – Rationale and Evidence for Incorporation of a Strategy of Guideline- Recommended Care without Planned Testing in Low Risk patients | The Risk Tool developed using the PROMISE cohort employs 10 readily available clinical variables and has been validated in the SCOT-HEART population <sup>33, 34</sup> | The Risk Tool developed using the PROMISE cohort employs 10 readily available clinical variables (such as tobacco usage, ethnicity/race, and age) and has been validated in the SCOT-HEART population <sup>33, 34</sup> |
|---|---|---|
| IV.E. Rationale<br>for Selection of<br>Testing in Each<br>Arm – Usual<br>Care Arm | The use of cCTA is explicitly excluded as the initial diagnostic strategy in this arm. | The use of cCTA is explicitly excluded as the initial diagnostic strategy in this arm and prohibited as a subsequent test for the first 45 days after randomization. |
| IV.F.<br>Randomization<br>Method | Risk will be classified by a risk tool using pre-test clinical characteristics derived in the PROMISE trial and validated in SCOT-HEART. | Risk will be classified by a risk tool using pre-test clinical characteristics (including tobacco usage, ethnicity/race, and age) derived in the PROMISE trial and validated in SCOT-HEART. |
| IV.F.<br>Randomization<br>Method | The use of cCTA is explicitly excluded as the initial diagnostic strategy in this arm. | The use of cCTA is explicitly excluded as the initial diagnostic strategy in this arm and prohibited as a subsequent test for the first 45 days after randomization. |
| V.C. Participant<br>Cohort<br>Assignment –<br>Usual Care Arm | Performance of cCTA as the initial test is excluded in this arm. | Performance of cCTA as the initial test is excluded in this arm and prohibited as a subsequent test for the first 45 days after randomization. |
| V.E Cross over in precision evaluation arm participants | Section title: Cross over in precision evaluation arm participants Previous text deleted and replaced | Section title: Testing in precision evaluation arm for participants assigned to no immediate testing New text |

| VIII.A. Sample | Assuming 10% of usual care | Assuming 10% of usual care |
|---|---|---|
| Size | participants will receive angiography | participants will receive |
| Determination | as a first test results in an 8% | angiography as a first test results in |
| and Statistical | primary endpoint event rate at 1 year | an 8% primary endpoint event rate |
| Power | in the usual care group and 5% | at 1 year in the usual care group |
| | (absolute) event rate in the precision | and 5% (absolute) event rate in the |
| | care group (i.e., 37.5% relative effect | precision care group (i.e., 37.5% |
| | size) with 30% assigned to guideline- | relative effect size) with 20% |
| | recommended care with symptom | assigned to guideline- |
| | management and no planned testing. | recommended care with symptom |
| | | management and no planned |
| | | testing. |

# Amendment from version 1.2 dated September 10, 2018 to version 1.3 dated November 21, 2018

| Section | Version 1.2 | Version 1.3 |
|---|---|---|
| Throughout | Non hyperemic pressure ratio (NHPR) | Instantaneous wave free ratio (iFR) |
| protocol | | |
| | NHPR NHPR <0.90 | iFR iFR ≤0.89 |
| | Time to a composite of: MACE (all | Time to a composite of: MACE (all |
| <ul><li>Primary</li></ul> | cause death, non-fatal MI) or invasive | cause death, non-fatal MI) or invasive |
| Endpoint | cardiac catheterization without | cardiac catheterization without |
| | obstructive CAD (obstructive CAD | obstructive CAD (obstructive CAD |
| | defined as diameter stenosis ≥50% | defined as diameter stenosis ≥50% |
| | according to clinical site interpretation, | |
| | FFR≤0.80, or NHPR<0.90) at one year | quantitative coronary analysis (QCA), |
| | (intention to treat) | FFR≤0.80, or iFR≤0.89) at one year |
| | | (intention to treat) |
| , , , , | Stable typical or atypical symptoms | Stable typical or atypical symptoms |
| | suspicious for coronary artery disease | suggesting possible coronary artery |
| | with further non-emergent testing or | disease (CAD) with further non- |
| | elective catheterization recommended | emergent testing or elective |
| | to evaluate the presence of suspected | catheterization recommended to |
| | coronary artery disease | evaluate the presence of suspected |
| | Safe performance of cCTA: | CAD. Stable chest pain includes those |
| | Creatinine clearance ≥45 ml/min | who have fully been ruled out for Acute |
| | For a female participant of | Coronary Syndrome (ACS) and for |
| | childbearing potential, a pregnancy | whom elective testing is |
| | test must be performed with negative | recommended, regardless of the |
| | results known within 7 days prior to | venue in which they are seen. |
| | randomization | Safe performance of cCTA: |
| | | Creatinine clearance ≥45 ml/min per |
| | | most recent measurement within 90 |
| | | days |
| | | For a female participant of |
| | | childbearing potential (those who have |
| | | not been surgically sterilized or are not |
| | | postmenopausal), a pregnancy test |

| | | must be performed with negative results known within 7 days prior to randomization |
|---|---|---|
| I. Study<br>Synopsis –<br>Exclusion<br>Criteria | <ol> <li>Noninvasive or invasive CV testing for CAD within 1 year</li> <li>Lifetime history of any obstructive CAD (no prior CABG or PCI, stenosis ≥505) or known EF ≤40% or moderate to severe valvular or congenital cardiac</li> <li>Contraindications to cCTA including but not limited to estimated creatinine clearance (GFR) &lt;45 m/min measured within 90 days.</li> <li>Exceeds local weight or size limit for cCTA or cardiac catheterization</li> </ol> | <ol> <li>Noninvasive or invasive CV testing within 1 year (for suspected CAD). CV testing for CAD refers to any stress tests, ICA and cCTA (including calcium scoring) only. Resting ECG and resting echocardiogram are not exclusionary.</li> <li>Lifetime history of known obstructive CAD (prior myocardial infarction, CABG or PCI, stenosis ≥50%), known EF ≤40% or other moderate to severe valvular or congenital cardiac disease.</li> <li>Contraindications to cCTA including but not limited to creatinine clearance (GFR) &lt;45 ml/min as per most recent measurement taken within 90 days.</li> <li>Exceeds the site's weight or size limit for cCTA or cardiac catheterization</li> </ol> |
| IV.B.<br>Primary<br>Objective<br>and<br>Endpoints | The primary endpoint is a composite of: MACE (all cause death and nonfatal MI) or invasive cardiac catheterization without CAD (no coronary stenosis ≥50%, or with FFR≤0.80, or nonhyperemic pressure ratio (NHPR) <0.90). The primary study hypothesis will be tested at one year using an intention to treat analysis | The primary endpoint is a composite of: MACE (all cause death and nonfatal MI) or invasive cardiac catheterization without CAD (no coronary stenosis ≥50% according to QCA by core-lab adjudication, or with FFR≤0.80, or instantaneous wave free ratio (iFR) ≤0.89). The primary study hypothesis will be tested at one year using an intention to treat analysis |
| IV.G. Diagnostic Evaluations and Subsequent Care – Description of Evaluations to be performed | A pregnancy test will be required for female participants of childbearing potential, and a creatinine blood test will be required for participants without a recent normal value (within previous 90 days). | A pregnancy test will be required for female participants of childbearing potential (those who have not been surgically sterilized or are not postmenopausal), and a creatinine blood test will be required for participants without a recent normal value (most recent measurement taken within previous 90 days). |

| IV.G. Diagnostic | | Added text: |
|---|---|---|
| Evaluations and<br>Subsequent<br>Care –<br>Subsequent<br>Care | | For patients in the Precision Evaluation Arm, ICA cannot be performed unless one of the following criteria are met: • Any stenosis ≥90% identified by cCTA • Left Main stenosis ≥30% identified by cCTA • Plaque rupture identified by cCTA • Lesion-specific FFR <sub>CT</sub> ≤0.85 in vessels with reference vessel size 2.0mm or greater in diameter |
| V.A. Patient | At the screening visit, patients will | At the screening visit, patients will |
| | <u>undergo the following:</u> | undergo the following: |
| Eligibility – Screening visit (in- | <br>Pregnancy test (for females of child- | Pregnancy test (for females of child- |
| , | bearing potential) | bearing potential – those who have |
| | , | not |
| | <u></u> | been surgically sterilized or are not postmenopausal) |
| | | · ′ |
| V.A. Patient<br>Screening for<br>Eligibility –<br>Inclusion<br>Criteria | 2. Stable typical or atypical symptoms suggesting possible coronary artery disease (CAD) with further non-emergent testing or elective catheterization recommended to evaluate the presence of suspected CAD. | 2. Stable typical or atypical symptoms suggesting possible coronary artery disease (CAD) with further non-emergent testing or elective catheterization recommended to evaluate the presence of suspected CAD. Stable chest pain includes those who have |
| | <ul><li>3. Safe performance of cCTA:</li><li>a. Creatinine clearance ≥45 ml/min</li></ul> | fully been ruled out for Acute Coronary Syndrome (ACS) and for whom elective testing is recommended, regardless of the venue in which they are seen. |
| | b. For a female participant of childbearing potential, a pregnancy test must be performed with negative results known within 7 days prior to randomization | 3. Safe performance of cCTA: a. Creatinine clearance ≥45 ml/min per most recent measurement within 90 days |

#### b. For a female participant of childbearing potential (those who have not been surgically sterilized or are not postmenopausal), a pregnancy test must be performed with negative results known within 7 days prior to randomization V.A. Patient 1. Acute chest pain 1. Acute chest pain Screening for 2. Unstable clinical status 2. Unstable clinical status Eligibility – 3. Noninvasive CV testing within 1 3. Noninvasive or invasive CV Exclusion vear (for suspected CAD). testing within 1 year for Criteria including coronary artery suspected CAD, CV testing calcium score refers to stress tests, ICA, and 4. History of known obstructive cCTA (including coronary artery CAD (prior myocardial calcium score) only. Resting infarction, CABG or PCI, ECG and resting stenosis ≥50%), known EF≤40% echocardiogram are not or other moderate to severe exclusionary. valvular or congenital disease 4. Lifetime history of known 5. Contraindications to cCTA obstructive CAD (prior myocardial infarction, CABG or including but not limited to PCI, coronary artery stenosis estimated creatinine clearance ≥50%), known EF≤40% or other (GFR) <45 ml/min moderate to severe valvular or 6. Any condition leading to congenital cardiac disease possible inability to comply with the protocol 5. Contraindications to cCTA 7. Exceeds the weight or size limit including but not limited to creatinine clearance (GFR) <45 for cCTA or cardiac catheterization at the site ml/min as per most recent measurement taken within 90 8. Life expectancy less than 2 days years due to non-cardiovascular 6. Exceeds the site's weight or comorbidities size limit for cCTA or cardiac 9. Enrolled in an investigational trial that involves a noncatheterization 7. Any condition leading to approved cardiac drug or device possible inability to comply which has not reached its with the protocol procedures primary endpoint and follow-up 10. Any condition that might 8. Any condition that might interfere with the study interfere with the study procedures or follow-up procedures or follow-up 9. Enrolled in an investigational trial that involves a nonapproved cardiac drug or device which has not reached its primary endpoint 10. Life expectancy less than 2 years due to non-cardiovascular

| | | comorbidities |
|---|---|---|
| VII.A. Primary Endpoint Definitions – Cardiac catheterization without obstructive coronary artery disease (diameter stenosis <50%, any FFR >0.80 or NHPR ≥0.90) | Cardiac catheterization without obstructive coronary artery disease will be defined as the absence of any ≥50% stenosis or hemodynamic indication of significance in any major epicardial vessel including side branches ≥2 mm in diameter, as determined by the clinical site interpretation. | Cardiac catheterization without obstructive coronary artery disease will be defined as the absence of any ≥50% stenosis or hemodynamic indication of significance in any major epicardial vessel, including side branches, ≥2 mm in diameter, as determined by core-lab adjudicated QCA or invasive FFR or iFR. |
| • | Myocardial infarction Myocardial infarction will be | Myocardial infarction Myocardial infarction will be |
| 1 - | characterized according to Universal | characterized according to the 4 <sup>th</sup> |
| | MI definition subtypes as Type 1, 2, 3, | Universal MI definition for |
| | 4a, | Spontaneous MI and the |
| | 4b, 4c, and 5. | SCAI definition for periprocedural Mls. |

## Amendment from version 1.3 dated November 21, 2018 to version 1.4 dated February 1, 2019

| Section | Version 1.3 | Version 1.4 |
|---|---|---|
| VII.A. Primary<br>Endpoint<br>Definitions –<br>Myocardial<br>infarction | Acute myocardial infarction (MI) is defined as having evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia 51. Specifically, MI is defined as having: | Acute myocardial infarction (MI) is defined as having evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia. Specifically, the Fourth Universal Definition <sup>51</sup> of type I MI is defined as: |
| | 1) Typical rise and/or gradual fall in cardiac biomarker level (cardiac troponin preferred) with values exceeding the 99 <sup>th</sup> percentile of the institutional upper limit of normal (ULN) (generally 2x the ULN) AND either: 2) Clinical presentation defined as typical cardiac ischemic type pain/discomfort or dyspnea felt to be due to ischemia and consistent with the diagnosis of myocardial ischemia and infarction | Detection of a rise and/or fall of cTn values with at least 1 value above the 99th percentile URL and with at least 1 of the following: - Symptoms of acute myocardial ischemia; - New ischemic ECG changes; - Development of pathological Q waves; - Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality in a pattern consistent with an ischemic etiology; - Identification of a coronary thrombus by angiography |

| | | including intracoronary |
|---|---|---|
| | Or | imaging or by autopsy* |
| | 3) ECG manifestations of acute myocardial ischemia (in absence of left ventricular hypertrophy and left bundle branch block) including evolving ST elevation, ST depression, T-wave changes, new pathological Q-waves (R waves in V1-2) in at least two consecutive leads or new left bundle branch block. A complete definition of the criteria for MI can be found in the 2017 Cardiovascular and Stroke Endpoint Definitions for Clinical Trials <sup>51</sup> . Peri-procedural infarctions are defined as greater than 3x ULN for serum CK-MB for PCI and greater than 5x ULN for CABG. | cTn indicates cardiac troponin; ECG, electrocardiogram; URL, upper reference limit. *Postmortem demonstration of an atherothrombus in the artery supplying the infarcted myocardium, or a macroscopically large circumscribed area of necrosis with or without intramyocardial hemorrhage, meets the type 1 MI criteria regardless of cTn values. A complete definition of the criteria for MI can be found in the Fourth Universal Definition <sup>51</sup> of Myocardial Infarction (2018). The exception will be for periprocedural myocardial infarctions, which are defined as biomarker elevation ≥10 times the upper reference limit (URL) for creatine kinase MB |
| | | (CKMB) and/or ≥70 URL for troponin as outlined in the most recent SCAI (Society for Cardiovascular Angiography and |
| | | Interventions) definition <sup>60</sup> . |
| Table of Abbreviations | I. | CAC: Coronary Artery Calcium added |
| Table of<br>Abbreviations | Not applicable | SCAI: Society for Cardiovascular<br>Angiography and Interventions |
| Exclusi | Not applicable | New exclusion criteria #11 added: |
| on<br>criteria | | 11. Known CAD by coronary calcium presence, either by prior CAC scoring or definite coronary calcium reported on a non-cardiac chest CT scan. |
| Secondary<br>Effectiveness<br>Endpoints | Proportion of invasive cardiac catheterization patients who undergo revascularization (PCI or CABG) within 6 months of enrollment | "Invasive cardiac catheterization" has been updated to invasive coronary angiogram. |
| | | Proportion of invasive coronary angiogram patients who undergo revascularization (PCI or CABG) within 6 months of enrollment |

| V.D.<br>Participa<br>nt<br>Follow-<br>Up | For North American participants, follow-<br>up after 45 days will be done by phone<br>interviews conducted by the DCRI<br>Outcomes Call Center. | Visit 45 day has been added along with further clarification on site participation: For North American participants, follow-up at 45 days and at 6, 12, and 24 months visits will be done by phone interviews conducted by the DCRI Outcomes Call Center, unless not allowed by their enrolling site. |
|---|---|---|
| IV.A<br>Overview of<br>PRECISE-<br>Diagram | Specify usual care preferred 1st test Data entered for PROMISE risk calculator | Randomization stratified by preferred first test if usual care and PROMISE risk score. |
| | Diagram from version 1.3. | Diagram updated to provide clarification on the pre-randomization step. |
| Referral of precisio n evaluati on cCTA participants for FFR <sub>CT</sub> determination s | Image sets showing at least one 30-90% stenosis in epicardial vessels of 2mm diameter or greater will be | Language updated to "should" from "will": Image sets showing at least one 30-90% stenosis in epicardial vessels of 2mm diameter or greater should be |
| IV.G.<br>Diagnostic<br>Evaluations<br>and | For patients in the Precision Evaluation Arm, ICA cannot be performed unless at least one of the following criteria are met: | With this amendment, the language has been softened from "cannot" to "should not": |
| Subsequent<br>Care | | For patients in the Precision Evaluation Arm, ICA should not be performed unless at least one of the following criteria are met: |
| Rationale for<br>Selection of<br>Testing in | Use of cCTA as the initial diagnostic strategy is specifically excluded in the usual care strategy arm and prohibited as a subsequent test for the first 45 | With this amendment, "or a calcium score" has been added to the protocol. Use of cCTA or a calcium score as the |
| Each Arm | days after randomization | initial diagnostic strategy is specifically excluded in the usual care strategy arm and prohibited as a subsequent test for the first 45 days after randomization |

| Selection of<br>Testing in<br>Each Arm | assigned to receive either guideline-<br>recommended medical management<br>without planned testing or cCTA with<br>selective FFR <sub>CT</sub> | "Including no CAC" language has been added with this amendment: The intervention in PRECISE will triage patients into two risk groups who will be assigned to receive either guideline- recommended medical management without planned testing (including no CAC) or cCTA with selective FFR <sub>CT</sub> |
|---|---|---|
| V.C<br>Participant<br>Cohort<br>Assignment | | score" has been added to the protocol. |
| V.C<br>Participant<br>Cohort<br>Assignment | (elevated risk). | "Including no CAC score" has been added: Participants will be assigned to either guideline-recommended medical management without planned testing (low risk) including no CAC score or cCTA with selective FFR <sub>CT</sub> (elevated risk). |
| References-<br>51 and 60 | 51. Hicks KA, Mahaffey KW, et al. | Reference 51 is updated and reference<br>60 is added with the new amendment<br>v1.4:<br>51.Thygesen K, Alpert JS, et al<br>60. Moussa ID, Klein LW, et al |

## Amendment from version 1.4 dated February 1, 2019 to version 1.5 dated October 15, 2019

|---|---|---|
| Investigator | NA | Included separate line for PI signature |
| Protocol | | |
| Signature Page | | |
| Table of | NA | AG: Agatston units |
| Abbreviations | <u>_</u> | |
| Table of | DECISION: Decisive Evaluation | Removed |
| Abbreviations | of <u>C</u> ardiac Ischemia, <u>S</u> ymptoms | |
| | and | |
| | Revascularizat <u>ion</u> | |
| Table of | HU: Hounsfield units | Removed |
| Abbreviations | | |

| IV. Study Overview<br>and Objectives -<br>Study duration | The anticipated total duration of the PRECISE study will be approximately 48 months for start-up, enrollment, follow up, and close out. Participants will be followed for 24 months after enrollment. | Overall study duration reduced to 36 month and patient follow up to 12 month after enrollment. "The anticipated total duration of the PRECISE study will be approximately 36 months for start-up, enrollment, follow up, and close out. Participants will be followed for 12 months after enrollment." |
|---|---|---|
| IV.A. Overview of PRECISE – figure of the trial design | Precision evaluation Strategy assigned by PROMISE risk strata Guideline rec medical management wo planned testing CCTA +/- FFR <sub>CT</sub> | Figure updated to remove 24 month and coprimary endpoints of DECISION. Arrows leading to GRMT or cCTA annotated "low risk" and "elevated risk" respectively. Patients with known nonobstructive coronary plaque or extensive coronary calcium randomized to the precision arm are mandated to undergo cCTA +/- FFRcT, independent from PROMISE risk score strata. |
| IV.B. Primary<br>Objective and<br>Endpoints | Per the exclusion criteria, any previous noninvasive or invasive CV diagnostic testing for suspected CAD must have been >1 year prior to enrollment. Patients with known obstructive CAD (prior myocardial infarction, CABG or PCI, any stenosis ≥50%) are ineligible for PRECISE. | Replaced with: "Patients with known nonobstructive coronary plaque or extensive coronary calcium randomized to the precision arm are mandated to undergo cCTA +/- FFR <sub>CT</sub> , independent from their PROMISE risk score strata." |
| IV.C. Secondary<br>Endpoints | Endpoints will be assessed at 45 days, 6 months, 1 year and 2 years. | Removed secondary endpoint assessment at 2 years: "Endpoints will be assessed at 45 days, 6 months and 1 year." |
| IV.C. Secondary<br>Endpoints | PRECISE primary endpoint at 24 month | Removed PRECISE primary endpoint at 24 month |